# **Cover Page for Statistical Analysis Plan**

| Sponsor name: | Novo Nordisk A/S |
|---|---|
| NCT number | NCT03061214 |
| Sponsor trial ID: | NN9535-4114 |
| Official title of study: | SUSTAIN <sup>TM</sup> CHINA - Efficacy and safety of semaglutide once-weekly versus sitagliptin once-daily as add-on to metformin in subjects with type 2 diabetes |
| Document date: | 22 August 2019 |

Semaglutide s.c (Ozempic®)
Trial ID: NN9535-4114
Clinical Trial Report
Appendix 16.1.9

Date: 22 August 2019
Version: 1.0
Status: Final

### 16.1.9 Documentation of statistical methods

# List of contents

| Statistical analysis plan | Link |
|---------------------------|------|
| Statistical documentation | Link |

Redacted statistical analysis plan Includes redaction of personal identifiable information only.

Statistical Analysis Plan Trial ID: NN9535-4114 UTN:U1111-1149-0432 EudraCT No.:NA


Date: Version: Status: Page: 28 May 2019 1.0 Final 1 of 30

Novo Nordisk

# Statistical Analysis Plan

Trial ID: NN9535-4114

Efficacy and safety of semaglutide once-weekly versus sitagliptin once-daily as add-on to metformin in subjects with type 2 diabetes

Author

Biostatistics Semaglutide s.c.

This confidential document is the property of Novo Nordisk. No unpublished information contained herein may be disclosed without prior written approval from Novo Nordisk. Access to this document must be restricted to relevant parties.


Date: Version: Status: Page:

28 May 2019 | Novo Nordisk 1.0 Final 2 of 30

# **Table of contents**

| | | | | | Page |
|---|---|---|---|---|---|
| Ta | ble of c | ontents | ••••• | | 2 |
| Lis | t of ab | breviation | s | | 3 |
| 1 | Intro | duction | ••••• | | 4 |
| | 1.1 | Trial inf | formation | | 4 |
| | 1.2 | Scope o | f the statistica | ıl analysis plan | 4 |
| 2 | Statis | tical consi | derations | | 5 |
| | 2.1 | | | 1S | |
| | 2.2 | Sample | size calculation | on | 6 |
| | 2.3 | Definition | on of analysis | sets | 7 |
| | 2.4 | Primary | endpoint | | 10 |
| | 2.5 | Seconda | ry endpoints | | 16 |
| | | 2.5.1 | Confirmat | ory secondary endpoints | 16 |
| | | 2.5.2 | Supportive | e secondary endpoints | 18 |
| | | | 2.5.2.1 | Efficacy endpoints | 18 |
| | | | 2.5.2.2 | Safety endpoints | 20 |
| | 2.6 | Health e | economics and | d/or patient reported outcomes | 25 |
| | 2.7 | China co | ohort | | 25 |
| 3 | Chan | ges to the | statistical an | alyses planned in the protocol | 27 |
| 4 | Refer | ences | | | 30 |

Statistical Analysis Plan
Trial ID: NN9535-4114
UTN:U1111-1149-0432
EudraCT No.:NA

Date:
28 May 2019
Version:
1.0
Status:
Final
Page:

### List of abbreviations

AACE American Association of Clinical Endocrinologists

ADA American Diabetes Association

AE adverse event

ANCOVA analysis of covariance

BG blood glucose
BMI body mass index
CTR clinical trial report

DTSQ Diabetes Treatment Satisfaction Questionnaire status

EAC event adjudication committee

ECG electrocardiogram FAS full analysis set

GLP-1 glucagon-like peptide-1 HDL high density lipoprotein

hsCRP highly sensitive C-reactive protein

ITT intention to treat

IWRS interactive voice/web response system

LLOQ lower limit of quantification LOCF last observation carried forward

MAR missing at random

MCAR missing completely at random MCMC markow chain Monte Carlo

MedDRA Medical Dictionary for Regulatory Activities

NDA new drug application

PP per protocol

PRO patient reported outcome

PT preferred term

REML restricted maximum likelihood

SAP statistical analysis plan SAS safety analysis set s.c. subcutanous

SD standard deviation SE standard error

TEAE treatment emergent adverse event

| Statistical Analysis Plan | Date: | 28 May 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.:NA | Page: | 4 of 30 | |

### 1 Introduction

#### 1.1 Trial information

This is a 30-week randomised, double-blind, double-dummy, active-controlled, multi-centre, multinational trial, four-armed, parallel-group trial comparing semaglutide 0.5 mg and 1.0 mg once weekly against sitagliptin 100 mg once-daily.

### **Primary objective**

To compare the effect of once-weekly dosing of two dose levels of semaglutide versus sitagliptin 100 mg once-daily on glycaemic control after 30 weeks of treatment.

To further detail the primary objective an estimand is defined which is an efficacy estimand. The scientific question is:

- What is the treatment difference between semaglutide and sitagliptin at week 30 for all randomised subjects if all subjects completed treatment and did not initiate rescue medication
- The population is defined by the inclusion/exclusion criteria of the trial
- The primary endpoint is change from baseline in HbA<sub>1c</sub> after 30 weeks of treatment
- Only data collected before the occurrence of the intercurrent events *initiation of rescue medication* and *discontinuation of trial product* are used in the analysis.

#### **Secondary objectives**

To compare the effects of once-weekly dosing of two dose levels of semaglutide versus sitagliptin 100 mg once-daily after 30 weeks of treatment on:

- Inducing and maintaining weight loss
- Other parameters of efficacy, safety and tolerability

An estimand similar to the one for the primary objective is defined for the secondary objective as addressed by weight loss, however with 'change from baseline in  $HbA_{1c}$  after 30 weeks' replaced by 'change from baseline in body weight after 30 weeks of treatment'.

#### 1.2 Scope of the statistical analysis plan

This SAP is based on the protocol "Efficacy and safety of semaglutide once-weekly versus sitagliptin once-daily as add-on to metformin in subjects with type 2 diabetes", version 3.0, and amendment 3. The SAP is relevant both for the analysis of data for the entire trial population and for the analysis of the China cohort by it self. See Section 2.7.

Statistical Analysis Plan
Trial ID: NN9535-4114
UTN:U1111-1149-0432
EudraCT No.:NA

Date: 28 May 2019 Version: 1.0
Status: Final
Page: 5 of 30

### 2 Statistical considerations

#### 2.1 General considerations

Results from the statistical analysis will generally be presented by two-sided confidence intervals with a confidence level of 95% and associated p-value. Superiority will be formulated and tested as one-sided hypotheses at a 2.5% significance level. Non-inferiority between two treatments will be evaluated by comparing the upper limit of the associated two-sided 95% confidence interval for the difference with the pre-defined non-inferiority margin.

The two sitagliptin/semaglutide placebo groups will be pooled in all outputs if not otherwise specified.

When grouping or analysing data by country, subjects from Hong Kong and Taiwan will be grouped with Chinese subjects if not otherwise specified. The same is done when grouping or analysing by region China/Other where subjects from South Africa, Korea, Brazil and Ukraine will be analysed together in the group referred to as "Other".

#### **Data transformations**

A number of the continuous parameters will be log-transformed prior to statistical analysis. The output tables and figures will show the results of the analysis back-transformed to the original scale, implying that log-treatment-differences are reported as treatment ratios. Confidence intervals for the treatment ratios will be calculated as exponentiated upper and lower limits for log-treatment difference confidence intervals. The standard errors (SE) of the back-transformed mean and ratio to baseline estimates are also provided; these SEs are calculated using the delta-method (first order Taylor approximation), whereby the SE on the original scale is calculated as the product of the SE on log-scale and the exponentiated estimate of the mean (geometric mean).

#### Handling of missing data

In the case of missing data no general imputation will be performed for the analyses, unless otherwise specified. If an assessment has been made both at screening and randomisation, the value from the randomisation visit will be used as the baseline value. If the value measured at the randomisation visit is missing and the assessment also has been made at screening, then the screening value will be used as the baseline value.

Laboratory values below the lower limit of quantification (LLOQ) will be set to ½ LLOQ.

The primary analysis model will be the mixed model for repeated measurements (MMRM), see Section 2.4 for further details. One of the assumptions behind MMRM is that the missing data mechanism is missing at random (MAR). This means that given the observed data, the mechanism

| Statistical Analysis Plan | Date: | 28 May 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.:NA | Page: | 6 of 30 | |

generating missing values is independent of the unobserved data, that is the missing data. The MMRM rely on the MAR assumption for generating unbiased estimates of treatment differences.

Based on previous semaglutide trials in subjects with type 2 diabetes, the treatment discontinuation rate from randomised treatment and trial withdrawal is expected to be about 20%. The treatments in this trial should be effective, given the historical documentation, and this should minimise treatment discontinuation due to ineffective therapy. The main reasons for treatment discontinuation are expected to be AEs, ineffective therapy and non-eligibility (subjects randomised although not fulfilling inclusion/exclusion criteria). Treatment discontinuation due to non-eligibility can be regarded as missing completely at random (MCAR), i.e. it does not depend on the observed or missing data values. This category of missing data is not expected to introduce bias in the estimated treatment differences. Treatment discontinuation due to lack of efficacy is expected to be reflected in the observed data obtained prior to the discontinuation from randomised treatment, and the corresponding missing data can therefore be assumed as MAR to some extent. Missing data due to AEs is expected to be similar between groups except for, potentially, a slightly higher incidence in the semaglutide treatment group due to gastrointestinal side effects. Together with potential withdrawals from trial due to the own will of the subject, the MAR assumption may be less adequate for this category of drop-outs.

Several different sensitivity analyses described in subsequent sections will be used to investigate whether the results from the MMRM approach are robust towards deviations from the assumption of MAR.

### 2.2 Sample size calculation

The primary objective is to compare the effect of two dose levels of semaglutide once-weekly treatment (0.5 mg or 1.0 mg) with sitagliptin 100 mg on the primary endpoint, change from baseline in  $HbA_{1c}$  after 30 weeks of treatment. In the power calculations below it is presumed that in the analysis the two sitagliptin/semaglutide placebo groups will be pooled assuming no correlation between endpoints and placebo volume.

At the time of finalising the first version of the protocol, the regulatory guidance in China was to have 300 subjects in region China treated with semaglutide. To ensure an adequate and robust evaluation of safety and efficacy in the subjects from China 300 subjects completing treatment with semaglutide is used. In the following, subjects from Hong Kong and Taiwan will be grouped with the Chinese subjects and referred to as region China. Assuming a treatment discontinuation rate of 25% in this region and considering the 2:2:1:1 randomisation, this means that 600 subjects need to be randomised in region China. Trial NN9535-4114 is a multi-regional clinical trial, and 258 subjects are planned to be randomised outside region China as has already been approved by local authorities for these countries. For some countries the allocated subject number is required to

| Statistical Analysis Plan | Date: | 28 May 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.:NA | Page: | 7 of 30 | |

support local NDA submissions. In total, 858 subjects are planned to be randomised in a 2:2:1:1 manner. Assuming that 20% of all randomised subjects discontinue randomised treatment, and further taking the assumption that these subjects are excluded from the per protocol (PP) analysis set, 228 subjects in each group are expected to be included in the PP analysis set.

In total six confirmatory hypotheses are to be tested (see Section <u>2.4</u>). The six hypothesis tests are assumed to be independent and for each of the hypotheses the power calculation is based on a t-statistic under the assumption of a one-sided test of size 2.5%.

Using a non-inferiority margin of 0.3%-point, a standard deviation (SD) of 1.1%-point and a total of 228 subjects per group in the PP analysis set will give 90% marginal power to conclude HbA<sub>1c</sub> non-inferiority for the comparison of a semaglutide dose vs. sitagliptin 100 mg if the true HbA<sub>1c</sub> treatment difference (semaglutide minus sitagliptin) is as low as -0.03 %-point. Thereby, the overall power to demonstrate HbA<sub>1c</sub> non-inferiority for the two dose levels of semaglutide vs. sitagliptin will be at least 80%, even if the true treatment difference for the low dose comparison is as low as -0.03 %-point. With 286 subjects per group in the full analysis set (FAS), a marginal power of at least 90% for demonstrating HbA<sub>1c</sub> superiority, for any dose of the two dose level comparisons, is obtained if the true treatment difference is as low as -0.30%-point.

For change in body weight, using a SD of 4 kg and 286 subjects per group, a marginal power of at least 90% for demonstrating superiority for the comparison of a semaglutide dose vs. sitagliptin 100 mg is obtained if the true treatment difference is as low as -1.09 kg body weight.

In SUSTAIN 2, the mother trial of NN9535-4114, semaglutide showed marked and significant reductions in HbA<sub>1c</sub> and body weight vs sitagliptin at week 56. The change over time in HbA<sub>1c</sub> and body weight in SUSTAIN 2 showed marked reductions in both endpoints already at week 30 which supports the above mentioned true treatment differences for trial NN9535-4114.

#### 2.3 Definition of analysis sets

The following analysis sets are defined in accordance with the ICH-E9 guideline<sup>58</sup>.

Full Analysis Set (FAS): includes all randomised subjects. Subjects in the FAS will contribute to the evaluation "as randomised".

Per Protocol (PP) Analysis Set:

Includes all subjects in the FAS who fulfil the following criteria:

| Statistical Analysis Plan | Date: | 28 May 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.:NA | Page: | 8 of 30 | |

- have not violated any inclusion criteria
- have not fulfilled any exclusion criteria
- have a non-missing HbA<sub>1c</sub> measurement at screening and /or randomisation
- have at least 23 weeks actual treatment weeks of exposure
- have at least one non-missing HbA<sub>1c</sub> measurement after 23 actual weeks of exposure

Subjects in the PP Analysis Set will contribute to the analysis "as treated".

Safety Analysis Set (SAS): includes all subjects exposed to at least one dose of trial product. Subjects in the SAS will contribute to the evaluation based on the trial product received for the majority of the period they were on treatment. This will be referred to as contributing to the evaluation "as treated".

Before data are locked for statistical analysis, a review of all data will take place. Any decision to exclude a subject or single observations from the statistical analysis is the joint responsibility of the members of the internal study group. Exclusion of data from analyses will be used restrictively and normally no data should be excluded from the FAS. The subjects or observations to be excluded, and the reasons for their exclusion must be documented and signed by those responsible before database lock. The subjects and observations excluded from analysis sets, and the reason for this, will be described in the CTR.

#### Data selections and observation periods

Subjects and data to be used in an analysis will be selected in a two-step manner.

- Firstly, subjects will be selected based on the specified analysis set
- Secondly, data points on the selected subjects from first step will be selected based on the specified observation period

Definition of the observation periods:

**In-trial:** This observation period represents the time period where subjects are considered to be in the trial after randomisation, regardless of discontinuation of trial product or initiation of rescue medication. The in-trial observation period starts at randomisation (as registered in IWRS) and ends at the date of:

- The last direct subject-site contact, which is scheduled to take place 5 weeks after planned last dose of trial product at a follow-up visit
- Withdrawal for subjects who withdraw their informed consent

| Statistical Analysis Plan | Date: | 28 May 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.:NA | Page: | 9 of 30 | |

- The last subject-investigator contact as defined by the investigator for subjects who are lost to follow-up
- Death for subjects who dies before any of the above

For subjects not randomised but exposed to trial product the in-trial periods starts at the date of first dose of trial product

**On-treatment:** This observation period represents the time period where subjects are considered treated with trial product. The observation period is a sub-set of the in-trial observation period. It starts at the date of first dose of trial product. Two slightly different end dates will be needed to cover all assessments appropriately according to the flow chart. For adjudicated events, ECG's and AEs including hypoglycaemic episodes, the observation period ends at the first date of any of the following:

- the follow-up visit (V10)
- the follow-up prematurely discontinuation visit (V10A)
- the last date on trial product + 42 days
- the end-date for the in-trial observation period

The follow-up visit is scheduled to take place 5 weeks after the last date on trial product corresponding to approximately five half-lives of subcutaneous semaglutide. The visit window for the follow-up visit is + 7 days, which is the reason for the 42 days specified in the bullet above. Hence, for those assessments this period reflects the period in which subjects are exposed.

For efficacy and other safety assessments (laboratory assessments, physical examination and vital signs) the observation period ends at the last date on trial product + 7 days in accordance with trial flow chart and assessment times. This ascertainment window corresponds to the dosing interval and will be used to avoid attenuation of a potential treatment effect on endpoints for which the effect is reversible shortly after treatment discontinuation. Hence, for those assessments this period reflects the period in which subjects are treated.

**On-treatment without rescue medication:** This observation period is a sub-set of the on-treatment observation period, where subjects are considered treated with trial product, but have not initiated any rescue medications. Specifically it starts at date of first dose of trial product and the observation period ends at the first date of any of the following:

- the last dose of trial product +7 days
- initiation of rescue medication

| Statistical Analysis Plan | Date: | 28 May 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.:NA | Page: | 10 of 30 | |

The 'on-treatment without rescue medication' observation period will be the primary observation period for efficacy evaluations. The in-trial observation period will be considered supportive for efficacy evaluation. Safety will be evaluated based on the in-trial and the on-treatment observation periods unless otherwise specified.

For subjects who have no post-baseline scheduled assessments available in the on-treatment without rescue period, the baseline value will be carried forward to the first scheduled visit for the associated endpoint to ensure that all randomised subjects will contribute to the statistical analysis. This will not be done for the PRO assessments which are only taken at baseline and the week 30 visit.

Data points collected outside an observation period will be treated as missing in the analysis. Baseline data will always be included in an observation period. For adjudicated events, the onset date will be the EAC adjudicated onset date.

### 2.4 Primary endpoint

The primary endpoint is change from baseline in HbA1c after 30 weeks of treatment. In the analysis the two sitagliptin/semaglutide placebo groups will be pooled assuming no correlation between HbA<sub>1c</sub> change after 30 weeks and placebo volume.

The primary endpoint will be based on FAS using data from the 'on-treatment without rescue medication' observation period in a Mixed Model for Repeated Measures (MMRM). A restricted maximum likelihood (REML) will be used. The model will include all post baseline HbA<sub>1c</sub> measurements collected at scheduled visits up to and including week 30 data as dependent variables. The independent effects included in the model will be treatment and region China/Other as fixed effects and baseline response as covariate, all nested within visit. An unstructured covariance matrix will be employed for measurements within the same subjects, assuming that measurements across subjects are independent. Regarding missing data this analysis approach relies on the assumption that data are missing at random (MAR). From this model, the two dose level estimated treatment differences between s.c. semaglutide versus sitagliptin at week 30 will be presented together with associated two-sided 95% confidence intervals and unadjusted two sided pvalues (nominal alpha=0.05) for testing non-inferiority and superiority. In order to preserve the overall type 1 error the conclusion of non-inferiority and superiority with treatment of each semaglutide dose versus sitagliptin after 30 weeks will be evaluated hierarchically according to the sequence below, and starting with the first. In this testing sequence it is necessary to fulfil the test criteria, which is to reject the corresponding null hypothesis in order to go to the next step. If the corresponding null hypothesis is not rejected, the testing will stop and no further conclusions will be drawn.

The following ordering in the statistical test sequence will be used:

1. Non-inferiority in change in  $HbA_{1c}$  for semaglutide 1.0 mg vs. sitagliptin

| Statistical Analysis Plan | Date: | 28 May 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.:NA | Page: | 11 of 30 | |

- 2. Non-inferiority in change in HbA<sub>1c</sub> for semaglutide 0.5 mg vs. sitagliptin
- 3. Superiority in change in HbA<sub>1c</sub> for semaglutide 1.0 mg vs. sitagliptin
- 4. Superiority in change in body weight for semaglutide 1.0 mg vs. sitagliptin
- 5. Superiority in change in body weight for semaglutide 0.5 mg vs. sitagliptin
- 6. Superiority in change in HbA<sub>1c</sub> for semaglutide 0.5 mg vs. sitagliptin

Non-inferiority will be concluded if the upper limit of the two-sided 95% confidence interval for the estimated difference in  $HbA_{1c}$  between semaglutide and situagliptin is less than 0.3%. Superiority for either change in  $HbA_{1c}$  or change in body weight will be claimed if the upper limit of the two-sided 95% confidence interval for the estimated difference is below 0% or 0 kg respectively.

When establishing non-inferiority the analysis will be based on the full analysis set (FAS) and supplemented by an analysis with the per protocol population using the data from the 'on treatment without rescue medication' observation period as supportive evidence. The FAS population will be used in the analysis when concluding superiority.

### Sensitivity analysis

To investigate the sensitivity of the main results, complimentary and separate analyses for primary endpoint and the confirmatory secondary endpoint will be performed, using the FAS only, except for  $HbA_{1c}$ , where the PP analysis set will be used in a sensitivity analysis regarding the non-inferiority evaluation. These analyses will investigate the sensitivity of the results due to the impact of missing values.

The primary analysis regarding non-inferiority of the primary endpoint change in  $HbA_{1c}$  after 30 weeks will also be performed separately based on the data in the PP analysis set only.

The primary endpoint and the secondary confirmatory endpoint will be evaluated in the following sensitivity analyses:

- An analysis of covariance (ANCOVA) model will be analysed with imputation of missing values according to the last observation carried forward (LOCF) method based on the FAS and using the data from the 'on-treatment without rescue medication' observation period. The model will include terms for treatment, region China/Other, and the corresponding baseline value as a covariate. The response variable will be the last available value obtained within the 30 weeks period of the trial
- The MMRM will be analysed based on all data from the 'in-trial' observation period A MMRM model will be analysed based on data only from subjects that completed treatment without receiving rescue treatment and who has a valid HbA1c assessment at visit 9 (week 30). The model will include terms for treatment, region China/Other, and the corresponding baseline value as a covariate.

| Statistical Analysis Plan | Date: | 28 May 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.:NA | Page: | 12 of 30 | |

A pattern mixture model based on the FAS using the 'on-treatment without rescue medication' observation period approach mimicking an ITT scenario where withdrawn subjects are assumed to be switched to a treatment inferior to the control treatment after treatment discontinuation will be performed for evaluation of non-inferiority for the primary endpoint change in  $HbA_{1c}$  at 30 weeks.

- In the first step intermittent missing values are imputed using a Markov Chain Monte Carlo (MCMC) method, in order to obtain a monotone missing data pattern. This imputation is done for each treatment group separately and 500 copies of the dataset will be generated.
- In the second step, for each of the 500 copies of the dataset, an analysis of variance model with the same factors as the primary model, and baseline HbA<sub>1c</sub> and HbA<sub>1c</sub> at 4 weeks (Visit 3) as covariate is fitted to the change in HbA<sub>1c</sub> from baseline to 8 weeks (Visit 5) for the sitagliptin group only. The estimated parameters, and their variance, from this model are used to impute missing value at 8 weeks for subjects in all treatment groups, based on region China/Other and HbA<sub>1c</sub> at baseline and 4 weeks.
- In the third step, for each of the 500 copies of the dataset, missing HbA1c values at 12 weeks (Visit 6) are imputed in the same way as for 8 weeks. Now the imputations are based on an analysis of variance model with the same factors and the HbA1c values at baseline, 4 weeks and 8 weeks as covariates, fitted to the control group.
- This stepwise procedure is then repeated sequentially over the available planned visits, adding one visit in each step until the last planned visit at 30 weeks (Visit 9).
- For each subject with imputed values in the investigational treatment groups, a value of 0.3% (the non-inferiority limit) is added to the change in HbA<sub>1c</sub> at 30 weeks.
- For each of the complete data sets, the change from baseline to week 30 is analysed using an analysis of variance model with the same set of factors and the baseline HbA<sub>1c</sub> value as a covariate.
- The estimates and standard deviations for the 500 data sets are pooled to one estimate and associated standard deviation using Rubin's rule (page 255-257)<sup>59</sup> From these pooled estimates the confidence interval for the treatment differences and the associated p-value are calculated. The upper limit of the two sided 95% confidence interval will be compared to the non-inferiority limit of 0.3%.

A pattern mixture model approach mimicking an ITT scenario where subjects after initiation of rescue medication or premature treatment discontinuation are assumed to be switched to the control treatment after treatment discontinuation will be performed separately for the evaluation of superiority in the primary endpoint change in  $HbA_{1c}$  and change in body weight at 30 weeks. The same types of approach as used for the non-inferiority assessment in change in  $HbA_{1c}$  will be employed, see above. However, the step where 0.3%, the non-inferiority limit, is added to the change in  $HbA_{1c}$  at 30 weeks will not be performed in this sensitivity analysis.

Furthermore to align with recent phase 3b trials evaluating safety and efficacy of semaglutide s.c., the following sensitivity analyses have been added:

| Statistical Analysis Plan | Date: | 28 May 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.:NA | Page: | 13 of 30 | |

- Tipping-point analysis (pattern mixture model like) based on the FAS using the 'ontreatment without rescue medication' observation period. In this analysis, subjects from the semaglutide group under investigation with missing observations will be given a penalty, i.e., it is assumed that subjects with missing observations who are randomised to semaglutide will receive a treatment that is worse than subjects with observed values who are randomised to semaglutide. The idea is to gradually increase the penalty to evaluate at which level the superiority/non-inferiority conclusion of the analyses in terms of statistical significance is changed for each of the two semaglutide dose levels separately. The tipping point is the penalty level, at which the magnitude of efficacy reduction in subjects with missing data creates a shift in the treatment effect of semaglutide from being statistically significantly better than sitagliptin to being non-statistically significantly better for the superiority test and similarly for the non-inferiority test. Technically, this analysis will be implemented in the following way:
  - Intermittent missing values are imputed using a Markov Chain Monte Carlo (MCMC) method, in order to obtain a monotone missing data pattern. This imputation is done for each of the treatment groups separately and 500 copies of the dataset will be generated.
  - A sequential regression approach for imputing monotone missing values at planned visits will be implemented starting with the first visit after baseline and sequentially continuing to the last planned visit at week 30. A model used to impute missing values at each planned visit will be fitted for each of the treatment groups using observed data. The model will include stratification factor region China/Other as a categorical effect and baseline and post-baseline HbA<sub>1c</sub> values observed or imputed prior to the visit in question as covariates. This step is similar to the detailed description given for the pattern mixture model approach described above.
  - O Subsequently, increasing penalty values will be added at week 30 to imputed observations in the semaglutide group under investigation. Specifically, when evaluating treatment differences involving the 0.5 mg semaglutide group, only subjects in this group are given a penalty, and vice versa for treatment differences involving the 1.0 mg semaglutide group. For each penalty and each of the 500 complete data set, HbA<sub>1c</sub> at week 30 will be analysed using an ANCOVA with treatment, and the stratification factor (region China/other) as categorical effects and baseline HbA<sub>1c</sub> as a covariate. Rubin's rules will be used to combine the analysis results in order to draw inference.
- Retrieved drop-out analysis based on the FAS using post-baseline measurements up to and including week 30 from the in-trial observation period. Missing data will be imputed using the same approach as described for the tipping point analysis above. However, the imputation will be done within the same group defined not only by the randomised treatment (semaglutide (0.5mg or 1.0 mg) /sitagliptin) but also by the status of treatment completion (still on randomised treatment at week 30 yes/no). It is hereby assumed that the likely values of what the missing data would have been if available are best described by information

| Statistical Analysis Plan | 1 | Date: | 28 May 2019 | Novo Nordisk |
|---|---|---|---|---|
| EudraCT No.:NA | | Page: | 14 of 30 | |

from subjects who at week 30 are similar in terms of randomised treatment and treatment completion status. The analysis model for the retrieved drop-out analysis is the same as for the tipping point analysis. This analysis could be considered addressing a treatment policy estimand. The retrieved drop-out is carried out for the superiority testing only.

In <u>Table 1</u> below a schematic overview of the different sensitivity analyses is provided.

Table 1 Summary of statistical analyses of the primary endpoint (HbA<sub>1c</sub>)

| Population | Period | Statistical model | Imputation <sup>1)</sup> | Hypothesis to be tested |
|---|---|---|---|---|
| | Primar | y non-inferiority | y analysis | |
| FAS | On-treatment without rescue medication | MMRM <sup>2)</sup> | Baseline values will be carried forward to week 4 for subjects with missing week 4 values. | Non-<br>inferiority |
| | Prima | ary superiority a | analysis | |
| FAS | On-treatment without rescue medication | MMRM <sup>2)</sup> | Baseline values will be carried forward to week 4 for subjects with missing week 4 values. | Superiority |
| | S | Sensitivity analy | ses | |
| PP | On-treatment without rescue medication | MMRM | Baseline values will be carried forward to week 4 for subjects with missing week 4 values. | Non-<br>inferiority |

Statistical Analysis Plan Trial ID: NN9535-4114 UTN:U1111-1149-0432 EudraCT No.:NA


Date: Version: Status: Page: 28 May 2019 1.0 Final 15 of 30

| Novo | Nordisk |
|------|---------|
| NOVO | NOTUISK |

| Complete cases | On-treatment without rescue medication | MMRM | Not applicable | Superiority |
|---|---|---|---|---|
| FAS | On-treatment without rescue medication | ANCOVA <sup>4)</sup> | Last<br>observation<br>carried forward<br>for subjects<br>with missing<br>value at week<br>30 | Superiority |
| FAS | In-trial | MMRM | Baseline values<br>will be carried<br>forward to<br>week 4 for<br>subjects with<br>missing week 4<br>values | Superiority |
| FAS | On-treatment without rescue medication | Pattern<br>mixture model<br>using an<br>ANCOVA <sup>4)</sup> | Multiple imputation | Non-<br>inferiority |
| FAS | On-treatment without rescue medication | Pattern<br>mixture model<br>using an<br>ANCOVA <sup>4)</sup> | Multiple imputation | Superiority |
| FAS | On-treatment without rescue medication | Tipping point<br>analysis using<br>an<br>ANCOVA <sup>4)5)</sup><br>model | Multiple<br>imputation | Non-<br>inferiority |
| FAS | On-treatment without rescue medication | Tipping point<br>analysis using<br>an ANCOVA<br>model <sup>4)</sup> | Multiple<br>imputation | Superiority |
| FAS | In-trial | Retrieved<br>dropout<br>analysis, using<br>an ANCOVA | Multiple imputation | Superiority |

| Statistical Analysis Plan | CONFIDENTIAL | Date: | 28 May 2019 |
|---------------------------|-----------------------|----------|-------------|
| Trial ID: NN9535-4114 | | Version: | 1.0 |
| UTN:U1111-1149-0432 | | Status: | Final |
| EudraCT No.:NA | | Page: | 16 of 30 |
| | model <sup>3)4)</sup> | | |

- 1) If a subject is missing baseline assessment the screening assessment will be used as the baseline assessment. If no measurement(s) have been obtained, at or prior to randomisation, the baseline value will be left missing.
- 2) MMRM model will be used to estimate the efficacy estimand
- 3) Retrieved dropout analysis, using an ANCOVA model, will be used to estimate the treatment policy estimand
- 4) Baseline and week 30 measurements will be used in the analysis
- 5) The non-inferiority margin of 0.3 is added as a penalty to imputed values in the semaglutide treatment groups

### 2.5 Secondary endpoints

The planned secondary endpoints used to support the primary and secondary objectives will be analysed as outlined in this section.

### 2.5.1 Confirmatory secondary endpoints

#### Weight loss

A confirmatory secondary variable is change in body weight after 30 weeks of treatment. This variable will be analysed in the same type of model as the primary endpoint although with baseline body weight as covariate and with similar sensitivity analyses.

In <u>Table 2</u> an overview of the sensitivity analyses for the confirmatory secondary endpoint is provided.


28 May 2019 | Novo Nordisk 1.0 Final 17 of 30

# Table 2 Summary of statistical analyses of confirmatory secondary endpoint (Body weight)

| Population | Period | Statistical model | Imputation <sup>1)</sup> | Hypothesis to be tested |
|---|---|---|---|---|
| | Co | onfirmatory ana | lysis | |
| FAS | On-treatment without rescue medication MMRM <sup>2)</sup> Baseline values will be carried forward to week 4 for subjects with missing week 4 values. | | Superiority | |
| | S | Sensitivity analy | ses | |
| Complete cases | On-treatment without rescue medication | MMRM | Not applicable | Superiority |
| FAS | On-treatment without rescue medication | ANCOVA <sup>4)</sup> | Last<br>observation<br>carried forward<br>for subjects<br>with missing<br>value at week<br>30 | Superiority |
| FAS | In-trial | MMRM | Baseline values will be carried forward to week 4 for subjects with missing week 4 values | Superiority |
| FAS | On-treatment without rescue medication | Pattern<br>mixture model<br>using an<br>ANCOVA<br>model <sup>4)</sup> | Multiple<br>imputation | Superiority |
| FAS | On-treatment without rescue | Tipping point<br>analysis using<br>an ANCOVA | Multiple imputation | Superiority |

| | _ | | |
|---|---|---|---|
| Statistical Analysis Plan | Date: | 28 May 2019 | Novo Nordisk |
| EudraCT No.:NA | Page: | 18 of 30 | |

| | medication | model <sup>4)</sup> | | |
|---|---|---|---|---|
| FAS | In-trial | Retrieved | Multiple | Superiority |
| | | dropout | imputation | |
| | | analysis, using | | |
| | | an ANCOVA | | |
| | | model <sup>3) 4)</sup> | | |
| | | an ANCOVA model <sup>3) 4)</sup> | | |

- 1) If a subject is missing baseline assessment the screening assessment will be used as the baseline assessment. If no measurement(s) have been obtained, at or prior to randomisation, the baseline value will be left missing.
- 2) MMRM model will be used to estimate the efficacy estimand
- 3) Retrieved dropout analysis, using an ANCOVA model, will be used to estimate the treatment policy estimand
- 4) Baseline and week 30 measurements will be used in the analysis

### 2.5.2 Supportive secondary endpoints

### 2.5.2.1 Efficacy endpoints

All efficacy endpoints in this section will be summarised and evaluated using the FAS.

### **Continuous variables**

Change from baseline to week 30 in:

- FPG
- Insulin
- C-peptide
- glucagon
- pro-insulin
- pro-insulin/insulin ratio
- HOMA-B
- HOMA-IR
- fasting blood lipids (total cholesterol, LDL-cholesterol, VLDL-cholesterol, HDL-cholesterol, triglycerides and free fatty acids)
- BMI
- waist circumference
- systolic and diastolic blood pressure

| Statistical Analysis Plan | Date: | 28 May 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.:NA | Page: | 19 of 30 | |

#### hsCRP

will all be analysed based on the same observation period and type of model as the primary endpoint, but with the associated baseline value as a covariate.

Except for FPG, BMI, waist circumference, and blood pressure the values of the variables will be log transformed subject to analysis.

#### **Beta-cell function**

Beta-cell function (fasting HOMA-B and fasting HOMA-IR) will be calculated based on fasting insulin and FPG. The calculation will be done at the same time points as for fasting insulin and FPG samples.

The calculation of the fasting HOMA endpoints will be done as follows: Fasting HOMA-B (%) = 20 x fasting insulin  $[\mu U/ml]/(FPG[mmol/l]-3.5)$  Fasting HOMA-IR (%) = fasting insulin  $[\mu U/ml]$  x FPG [mmol/l]/22.5

#### **PRO** outcomes

The PRO outcome endpoints:

- PRO questionnaire outcome DTSQs (individual items and treatment satisfaction score (6 of the 8 items summed)), and
- PRO questionnaire outcome SF-36v2<sup>TM</sup> short Form health survey: Total scores (physical component and mental component) and scores from the 8 domains will be analysed separately using the ANCOVA model based on the data from the on-treatment without rescue medication observation period. Factors in the model will be treatment and region China/Other. The baseline value of the corresponding endpoint will be used as covariate in the analysis model.

#### 7-point profile

Subjects will be asked to perform SMPG measurements as described in the protocol Section 8.5.1.5.

The endpoints from the 7-point profiles that will be analysed at week 30 are:

- Mean of the 7-point profile, defined as the area under the profile, calculated using the trapezoidal method, divided by the measurement time
- Mean increment over all meals

The mean of the 7-point profile and the mean of the post prandial increments at week 30 will be analysed separately with the same data and type of methods as primary endpoint but with the corresponding baseline assessment as a covariate.

| Statistical Analysis Plan | Date: | 28 May 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.:NA | Page: | 20 of 30 | |

### Response in HbA<sub>1c</sub> and/or weight loss after 30 weeks

The secondary variables related to fixed response in HbA<sub>1c</sub> and/or weight loss at 30 weeks will be:

- Responder in HbA<sub>1c</sub> after 30 weeks of treatment (yes/no) defined as HbA<sub>1c</sub><7.0% (<53 mmol/mol) ADA target</li>
- Responder in HbA<sub>1c</sub> after 30 weeks of treatment (yes/no) defined as HbA<sub>1c</sub> ≤6.5% (48 mmol/mol) AACE target
- Weight loss  $\geq 5\%$
- Weight loss  $\geq 10\%$
- HbA<sub>1c</sub> <7.0% (53 mmol/mol) without severe or confirmed symptomatic hypoglycaemia (plasma glucose  $\le$ 3.1 mmol/L) and no weight gain

All these variables will be analysed based on the 'on-treatment without rescue medication' observation period separately in the same type of logistic regression model. The model will include factors for treatment and region China/Other. For the two responder in  $HbA_{1c}$  endpoints, baseline  $HbA_{1c}$  will be included in the model as a covariate, whereas for the weight responder endpoint ( $\geq$ 5% and  $\geq$ 10% weight loss), baseline weight will be included instead. For the composite endpoint (cf. last bullet), both baseline  $HbA_{1c}$  and baseline weight will be included.

Missing response data at 30 weeks will be imputed from respectively the MMRM used for the primary analysis of HbA<sub>1c</sub> and the confirmatory secondary endpoint change in body weight at 30 weeks. The results will be described by the odds ratio and the associated 95% confidence interval for the odds ratio.

#### 2.5.2.2 Safety endpoints

The safety endpoints will be evaluated based on SAS using both the on-treatment observation period and the in-trial observation period unless otherwise stated.

The following secondary endpoints are used to support the safety objectives:

- Number of treatment emergent AEs during 30 weeks of treatment
- Number of treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes during 30 weeks of treatment
- Treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes during 30 weeks of treatment (yes/no)

Change in safety endpoints assessed from baseline to 30 weeks of treatment and/or follow up:

- Haematology
- Biochemistry
- Calcitonin
- Urinalysis
- UACR
- Pulse

| Statistical Analysis Plan | Date: | 28 May 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.:NA | Page: | 21 of 30 | |

- ECG evaluation
- Physical examination evaluation
- Eye examination

Occurrence of semaglutide antibodies during 35 weeks of study duration (yes/no):

- Anti-semaglutide antibodies
  - o Anti-semaglutide antibodies with in vitro neutralising effect
  - o Anti-semaglutide antibodies cross reacting with endogenous GLP-1
    - Cross reacting antibodies with in vitro neutralising effect to endogenous GLP-1

Anti-semaglutide antibody level during and after 30 weeks of treatment

All safety endpoints will be summarised and evaluated by descriptive statistics using the SAS.

| Statistical Analysis Plan | Date: | 28 May 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.:NA | Page: | 22 of 30 | |

#### **Adverse events**

The following endpoint related to adverse events is used to support the safety objective;

• Number of treatment emergent adverse events (TEAEs)

A treatment-emergent AE is an event that has onset date (or increase in severity) during the ontreatment observation period. These will therefore be referred to as 'on-treatment AEs' hereafter. On-treatment adverse events are summarised descriptively in terms of the number of subjects with at least one event (N), the percentage of subjects with at least one event (%), the number of events (E) and the event rate per 100 years (R). These summaries are replicated by outputs including all 'in-trial' adverse events (i.e., adverse events with onset date [or increase in severity] during the 'in-trial' observation period). Adverse events with onset after the end of the 'in-trial' observation period will be reported in a listing. The development over time in gastrointestinal AEs will be presented graphically.

The most frequent adverse events will be defined as preferred terms (PTs) that are experienced by at least 5% of the subjects in any of the treatment arms.

All AEs will be coded using the most recent version of the Medical Dictionary for Regulatory Activities (MedDRA) coding.

#### **Pulse**

Pulse will be analysed separately using an analysis similar to the primary analysis of the primary endpoint. However, this analysis will be based on SAS using the data from the on-treatment observation period but with the pulse value at baseline as a covariate.

#### Laboratory assessments

Amylase and lipase will be analysed separately with the same type of methods as for pulse with the corresponding baseline assessment as a covariate. The values will be log transformed in the analysis.

#### Calcitonin

In addition to the descriptive statistics and categorical summary showing number of values in the categories normal, high, >20 ng/L, 50 ng/L and >100 ng/L, all subjects with any post-baseline value of calcitonin above 20 ng/L will be assessed.

#### Classification of Hypoglycaemia

| Statistical Analysis Plan | 1 | Date: | 28 May 2019 | Novo Nordisk |
|---|---|---|---|---|
| EudraCT No.:NA | | Page: | 23 of 30 | |

<u>Treatment emergent</u>: hypoglycaemic episodes will be defined as treatment emergent if the onset of the episode occurs within the on-treatment observation period (see definition of observation periods in Section 2.3.

Nocturnal hypoglycaemic episodes: are episodes with time of onset between 00:01 and 05:59 both inclusive.

Hypoglycaemic episodes are classified according to the Novo Nordisk classification of hypoglycaemia and the ADA classification of hypoglycaemia (see <u>Figure 2–2</u>).

### Novo Nordisk classification of hypoglycaemia

In normal physiology, symptoms of hypoglycaemia occur below a plasma glucose level of 3.1 mmol/L  $(56 \text{ mg/dL})^{\frac{1}{2}}$ . Therefore, Novo Nordisk has included hypoglycaemia with plasma glucose levels below this cut-off point of hypoglycaemia.

In this trial Novo Nordisk use the following classification in addition to the ADA classification (see **Figure 2–1**):

• Severe or BG confirmed symptomatic hypoglycaemia: An episode that is severe according to the ADA classification<sup>2</sup> or BG confirmed by a plasma glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.



Note: Glucose measurements are performed with capillary blood calibrated to plasma equivalent glucose values

BG: blood glucose PG: plasma glucose SMPG: Self-measured plasma glucose

Figure 2-1 Novo Nordisk classification of hypoglycaemia

| Statistical Analysis Plan Trial ID: NN9535-4114 UTN:U1111-1149-0432 EudraCT No.:NA | Date:<br>Version<br>Status:<br>Page: | 28 May 2019<br>n: 1.0<br>Final<br>24 of 30 | Novo Nordisk |
|---|---|---|---|
|---|---|---|---|

## ADA classification of hypoglycaemia<sup>2</sup>

- Severe hypoglycaemia: An episode requiring assistance of another person to actively
  administer carbohydrate, glucagon, or take of other corrective actions. Plasma glucose
  concentration may not be available during an event, but neurological recovery following the
  return of plasma glucose to normal is considered sufficient evidence that the event was
  induced by a low plasma glucose concentration.
- Asymptomatic hypoglycaemia: An episode not accompanied by typical symptoms of hypoglycaemia, but with a measured plasma glucose concentration ≤ 3.9 mmol/L (70 mg/dL).
- Documented symptomatic hypoglycaemia: An episode during which typical symptoms of hypoglycaemia are accompanied by a measured plasma glucose concentration ≤ 3.9 mmol/L (70 mg/dL).
- Pseudo-hypoglycaemia: An episode during which the person with diabetes reports any of the typical symptoms of hypoglycaemia with a measured plasma glucose concentration > 3.9 mmol/L (70 mg/dL) but approaching that level.
- Probable symptomatic hypoglycaemia: An episode during which symptoms of hypoglycaemia are not accompanied by a plasma glucose determination but that was presumably caused by a plasma glucose concentration ≤ 3.9 mmol/L (70 mg/dL).



Note: Glucose measurements are performed with capillary blood calibrated to plasma equivalent glucose values PG: plasma glucose SMPG: Self-measured plasma glucose

| Statistical Analysis Plan | Date: | 28 May 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.:NA | Page: | 25 of 30 | |

Figure 2–2 ADA classification of hypoglycaemia

#### Number of severe or BG confirmed symptomatic hypoglycaemic episodes

Data on treatment emergent hypoglycaemic episodes are presented in terms of the number of subjects with at least one episode, the percentage of subjects with at least one episode (%), the total number of episodes and the episodes rate per 100 years of exposure. Summaries of treatment emergent hypoglycaemic episodes will be presented as an overview including all episodes and episodes by severity.

The summary will include the number of severe or BG confirmed symptomatic hypoglycaemic episodes

### Number of nocturnal hypoglycaemic episodes

The number of nocturnal (00:01-05:59 am) treatment emergent episodes will be displayed as described above for hypoglycaemic episodes.

### Treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes (yes/no)

The number of subjects with treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes (yes/no) including nocturnal severe or BG confirmed symptomatic hypoglycaemic episodes (yes/no) can be assessed from the above described tables.

#### 2.6 Health economics and/or patient reported outcomes

The PRO questionnaires, SF- $36v2^{TM}$  and DTSQs, will be used to evaluate the objective regarding Quality of Life, see Section <u>2.5.2.1</u> for the details of the corresponding statistical analysis.

#### 2.7 China cohort

In order to assess the effect of semaglutide in the Chinese population all analyses will be done in the same way as described for the entire trial, but only including subjects from region China. For the sensitivity analyses using multiple imputations the imputations for each subject based on the entire population will be used.

| Statistical Analysis Plan | Date: | 28 May 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.:NA | Page: | 26 of 30 | |

| Statistical Analysis Plan |
|---------------------------|
| Trial ID: NN9535-4114 |
| UTN:U1111-1149-0432 |
| EudraCT No.:NA |


28 May 2019 | Novo Nordisk 1.0 Final 27 of 30

#### Changes to the statistical analyses planned in the protocol 3

The changes to the statistical analyses planned in the protocol are described in the table below.

| Change to planned statistical analysis | Rationale for change |
|---|---|
| A description of the estimand pertaining to the | Updated for clarification and to be in line with |
| primary objective and primary endpoint has | the use of estimands. |
| been added. | |
| Similarly is done for the secondary objective | |
| and confirmatory secondary endpoint. See | |
| Section 1.1 | |
| It is clarified that the SAP is relevant both for | A separate report describing the results for the |
| the analysis of data for the entire trial | Chinese cohort will be made. To clarify that the |
| population and for the analysis of the China | SAP is relevant for both the report for |
| cohort by it self. See Section 2.1 | NN9535-4114 as well as the report for the |
| | Chinese cohort, this statement was added |
| A statement regarding which subjects belong in | Stratification was not done by country as |
| region China and which subjects belong in | specified in the protocol but by region |
| region Other was added. See Section 2.1 | China/Other. Therefore, this specification is |
| | needed. |
| "country" replaced by "region China/Other" in | Due to the change in stratification this change |
| all statistical analyses throughout the document | is necessary to comply with ICH E9. |
| A section describing data transformations has | Updated for clarification |
| been added. See Section 2.1 | |
| The second decrease 1 and 1 and 1 and 1 | II. 1 4 1 C - 1 - 'C - 4' |
| The completer analysis has been separated | Updated for clarification. |
| from the "in-trial" analysis. Furthermore, a | |
| detailed description of the completer definition | |
| has been added. See Section 2.4 | II. 1-4-1 f1:f:4: |
| In the description of the pattern mixture model | Updated for clarification. |
| sensitivity analysis it has been clarified that subjects should have initiated rescue | |
| medication or discontinued treatment | |
| prematurely to be assumed switched to control | |
| treatment. See Section 2.4 | |
| In the description of the pattern mixture model | Updated for clarification. |
| sensitivity analysis it has been clarified in | Opanion for charmention. |
| bullet 5 that it is subjects with an imputed value | |
| at visit 9 (week 30) who will have a penalty | |
| added. See Section 2.4 | |
| Two extra sensitivity analyses – a tipping point | The extra sensitivity analyses have been added |
| analysis and a retrieved dropout analysis – have | to be in line with the sensitivity analyses used |
| anarysis and a retrieved dropout anarysis – nave | to be in time with the sensitivity analyses used |

| Statistical Analysis Plan | CONFIDENTIAL | Date: | 28 May 2019 Novo Nordisk |
|---|---|---|---|
| Trial ID: NN9535-4114 | | Version: | 1.0 |
| UTN:U1111-1149-0432 | | Status: | Final |
| EudraCT No.:NA | | Page: | 28 of 30 |

| 1 11.17.71 2 12 27.27 | : |
|---|---|
| been added to the section regarding sensitivity | in recent phase 3b trials investigating the effect |
| analyses. See Section <u>2.4</u> | of semaglutide s.c. |
| A table has been added to get a schematic | Updated for clarification. |
| overview of all the sensitivity analyses for the | |
| primary endpoint. See Section <u>2.4</u> | |
| The statistical subgroup analysis of the | Since the stratification has been changed to be |
| interaction effect between treatment and | by region China/Other the planned subgroup |
| country has been removed as well as the | analysis and safety assessment for China and |
| evaluation of safety for China and Korea. See | Korea were less relevant. Furthermore for the |
| Section 2.4 | Chinese cohort, a separate report including all |
| | analyses planned for the entire trial population |
| | will be made. |
| A table has been added to get a schematic | Updated for clarification. |
| overview of all the sensitivity analyses for the | |
| primary endpoint. See Section 2.5.1 | |
| "data" has been changed to "observation | Updated for clarification |
| period" in the description on how to analyse | ^ |
| supportive secondary efficacy endpoints. See | |
| Section <u>2.5.1</u> | |
| Treatment emergent has been added to the | Updated for clarification |
| definition of "Treatment emergent severe or | |
| BG confirmed symptomatic hypoglycaemic | |
| episodes during 30 weeks of treatment | |
| (yes/no)" and to the definition of nocturnal | |
| hypoglycaemic episodes. See Section 2.5.2.2 | |
| It has been clarified that analysis of pulse is | Pulse is a safety measure. |
| based on SAS instead of FAS. See Section | T disc is a surety incasure. |
| 2.5.2.2 | |
| The description of how calcitonin will be | The update is to be in line with how calcitonin |
| reported has been updated. See Section | was reported in SUSTAIN 2 (trial NN9535- |
| 2.5.2.2 | 3626) which is the mother trial for NN9535- |
| 2.3.2.2 | 4114 |
| The analyses of number of severe or BG | The number of severe or BG confirmed |
| confirmed hypoglycaemic episodes, number of | episodes is so low that a statistical analysis is |
| nocturnal severe or BG confirmed | not meaningful. |
| hypoglycaemic episodes, number of subjects | |
| with severe or BG confirmed hypoglycaemic | |
| episodes and number of subjects with nocturnal | |
| severe or BG confirmed hypoglycaemic | |
| episodes have been removed. See Section 2.1 | |
| and Section 2.5.2.2 | XX 1 . 10 1 . C |
| A paragraph describing the analyses that will | Updated for clarification. |
| be done for the Chinese cohort has been added. | |
| See Section 2.7 | |

| Statistical Analysis Plan | Date: | 28 May 2019 | Novo Nordisk |
|---|---|---|---|
| EudraCT No.:NA | Page: | 29 of 30 | |

| A number of typos and a updates to wordings | To ease readability and understanding |
|---|---|
| have been added throughout the document. | |

| Statistical Analysis Plan | 1 | Date: | 28 May 2019 | Novo Nordisk |
|---|---|---|---|---|
| EudraCT No.:NA | | Page: | 30 of 30 | |

#### 4 References

<sup>1</sup> Schwartz NS, Clutter WE, Shah SD, Cryer PE. Glycemic thresholds for activation of glucose counterregulatory

systems are higher than the threshold for symptoms. J Clin Invest.1987;79(3):777-81

<sup>2</sup> Seaquist ER, Anderson J, Childs B, Cryer P, Dagogo-Jack S, Fish L, et al. Hypoglycemia and diabetes: a report of a workgroup of the American Diabetes Association and the Endocrine Society. Diabetes Care. 2013;36(5):1384-95.

| NN9535 | | Date: | 03 July 2019 | Novo Nordisk |
|---|---|---|---|---|
| NN9535-4114 | CONFIDENTIAL | Version: | 1.0 | |
| Clinical Trial Report | CONFIDENTIAL | Status: | Final | |
| Section 16.1.9 | | Page: | 1 of 152 | |

# **Table of contents**

| | Page |
|--------------------------------------------------------------|------|
| 16.1.9.1 Pre-defined MedDRA search - list of preferred terms | 3 |

| NN9535 | | Date: | 03 July 2019 | Novo Nordisk |
|---|---|---|---|---|
| NN9535-4114 | CONFIDENTIAL | Version: | 1.0 | |
| Clinical Trial Report | | Status: | Final | |
| Section 16.1.9 | | Page: | 2 of 152 | |

# 16.1.9 Documentation of statistical methods

 NN9535
 Date:
 03 July 2019
 Novo Nordisk

 NN9535-4114
 Version:
 1.0

Clinical Trial Report Status: Final 

### 16.1.9.1 Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Acute gallstone disease AIDS cholangiopathy Ampulla of Vater stenosis Bile culture positive Bile duct necrosis Bile duct obstruction Bile duct pressure increased Bile duct stenosis Bile duct stenosis traumatic Bile duct stent insertion Bile duct stent removal Bile duct stone Bile output abnormal Bile output decreased Bile output increased Biliary abscess Biliary anastomosis
Biliary anastomosis complication Biliary ascites Biliary cast syndrome Biliary cirrhosis Biliary colic Biliary dilatation Biliary dyskinesia Biliary fibrosis Biliary fistula Biliary fistula repair Biliary ischaemia Biliary sepsis Biliary sphincterotomy Biliary tract dilation procedure Biliary tract disorder Biliary tract infection Biliary tract operation Biliary-bronchial fistula Biliary-vascular fistula Bilirubin conjugated abnormal Bilirubin conjugated increased Bilirubin excretion disorder Biloma Biloma rupture Biopsy bile duct abnormal Biopsy gallbladder abnormal Blood bilirubin abnormal Blood bilirubin increased Cholangiectasis acquired Cholangiogram abnormal Cholangiolitis Cholangiostomy Cholangitis Cholangitis acute Cholangitis chronic Cholangitis infective Cholangitis sclerosing Cholecystectomy Cholecystitis Cholecystitis acute Cholecystitis chronic Cholecystitis infective Cholecystocholangitis Cholecystoenterostomy Cholecystogram intravenous abnormal

Cholecystogram oral abnormal

NN9535 NN9535-4114 Clinical Trial Report Section 16.1.9


03 July 2019 Date: Version: Status:

Page:

Novo Nordisk

1.0

Final


Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Acute gallstone disease Cholecystostomy Choledochectomy Choledochoenterostomy Choledocholithotomy Choledochostomy Choledochotomy Cholelithiasis Cholelithiasis migration Cholelithiasis obstructive Cholelithotomy Cholelithotripsy Cholestasis Cholestasis of pregnancy Dilatation intrahepatic duct acquired Emphysematous cholecystitis Endoscopic retrograde cholangiopancreatography abnormal Endoscopy biliary tract abnormal Gallbladder abscess
Gallbladder cholesterolosis Gallbladder disorder Gallbladder empyema Gallbladder enlargement Gallbladder fibrosis Gallbladder fistula Gallbladder fistula repair Gallbladder hyperfunction Gallbladder hypofunction Gallbladder injury Gallbladder mucocoele Gallbladder necrosis Gallbladder obstruction Gallbladder oedema Gallbladder operation Gallbladder palpable Gallbladder rupture Gallbladder varices Gallbladder volvulus Gallstone ileus Gallstone lieus
Haemobilia
Hepatitis cholestatic
Hepatobiliary disease
Hepatobiliary infection Hepatolithectomy Hydrocholecystis Hyperbilirubinaemia Hyperplastic cholecystopathy Jaundice Jaundice cholestatic Jaundice extrahepatic obstructive Lemmel's syndrome Limy bile syndrome
Malignant biliary obstruction
Pancreatobiliary sphincterotomy
Parenteral nutrition associated liver disease Perforation bile duct Porcelain gallbladder Post cholecystectomy syndrome Post procedural bile leak Primary biliary cholangitis Pseudocholelithiasis Reynold's syndrome Sphincter of Oddi dysfunction

Ultrasound biliary tract abnormal

Date: 03 July 2019 | Novo Nordisk Version: Status: 5 of 152Page:

1.0

Final

Pre-defined MedDRA search - list of preferred terms

| Pre-defined MedDRA search | Preferred term |
|---|---|
| Acute gallstone disease | Vanishing bile duct syndrome<br>X-ray hepatobiliary abnormal |
| Acute renal failure | Acute kidney injury Acute phosphate nephropathy Albuminuria Anuria |
| | Azotaemia<br>Blood creatinine abnormal<br>Blood creatinine increased<br>Blood urea abnormal |
| | Blood urea increased Blood urea nitrogen creatinine ratio increased |
| | Continuous haemodiafiltration Creatinine renal clearance abnormal Creatinine renal clearance decreased |
| | Creatinine urine abnormal Creatinine urine decreased Crystal nephropathy |
| | Dialysis Foetal renal impairment Fractional excretion of sodium |
| | Glomerular filtration rate abnormal Glomerular filtration rate decreased |
| | Haemodialysis<br>Haemofiltration<br>Hypercreatininaemia |
| | Hyponatriuria<br>Intradialytic parenteral nutrition<br>Kidney injury molecule-1<br>Neonatal anuria |
| | Nephritis Nephropathy toxic Oedema due to renal disease |
| | Oliguria Peritoneal dialysis Prerenal failure |
| | Protein urine present Proteinuria Renal failure |
| | Renal failure neonatal<br>Renal function test abnormal<br>Renal impairment |
| | Renal impairment neonatal<br>Renal transplant<br>Renal tubular disorder |
| | Renal tubular dysfunction Renal tubular injury Renal tubular necrosis |
| | Tubulointerstitial nephritis Urea renal clearance decreased Urine output decreased |
| Allergic reactions | Acquired C1 inhibitor deficiency Acute generalised exanthematous pustulosis |
| | Administration related reaction Administration site dermatitis Administration site eczema |
| | Administration site hypersensitivity<br>Administration site rash<br>Administration site recall reaction |
| | Administration site urticaria |


Date: Version: Status: Page: 03 July 2019 1.0

Final 6 of 152

Novo Nordisk

 ${\tt Pre-defined} \ {\tt MedDRA} \ {\tt search} \ {\tt -list} \ {\tt of} \ {\tt preferred} \ {\tt terms}$ 

Pre-defined MedDRA search Preferred term Allergic reactions Administration site vasculitis Allergic bronchitis Allergic colitis Allergic cough Allergic cystitis Allergic eosinophilia Allergic gastroenteritis Allergic hepatitis Allergic keratitis Allergic oedema Allergic otitis externa Allergic otitis media Allergic pharyngitis
Allergic reaction to excipient Allergic respiratory disease Allergic respiratory symptom Allergic sinusitis Allergic stomatitis
Allergic transfusion reaction Allergy alert test positive Allergy test positive
Allergy to immunoglobulin therapy Allergy to surgical sutures Allergy to vaccine Alveolitis allergic Anaphylactic reaction Anaphylactic shock Anaphylactic transfusion reaction Anaphylactoid reaction Anaphylactoid shock Anaphylaxis treatment Angioedema Anti-neutrophil cytoplasmic antibody positive vasculitis Antiallergic therapy Antiendomysial antibody positive Application site dermatitis Application site eczema Application site hypersensitivity Application site rash Application site recall reaction Application site urticaria Application site vasculitis Arthritis allergic Aspirin-exacerbated respiratory disease Atopic cough Atopy Blepharitis allergic Blood immunoglobulin E abnormal Blood immunoglobulin E increased Bromoderma Bronchospasm Catheter site dermatitis Catheter site eczema Catheter site hypersensitivity Catheter site rash Catheter site urticaria Catheter site vasculitis Chronic eosinophilic rhinosinusitis
Chronic hyperplastic eosinophilic sinusitis
Circulatory collapse
Circumoral oedema
Circumoral swelling

Conjunctival oedema


Date: Version: Status: Page: 03 July 2019 1.0 Final


Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Idiopathic angioedema

Allergic reactions

Conjunctivitis allergic Contact stomatitis Contrast media allergy Contrast media reaction Corneal oedema Cutaneous vasculitis Dennie-Morgan fold Dermatitis Dermatitis acneiform Dermatitis allergic Dermatitis atopic Dermatitis bullous Dermatitis contact Dermatitis exfoliative Dermatitis exfoliative generalised Dermatitis herpetiformis Dermatitis infected Dermatitis psoriasiform Device allergy Dialysis membrane reaction Distributive shock Documented hypersensitivity to administered product Drug eruption Drug hypersensitivity Drug provocation test Drug reaction with eosinophilia and systemic symptoms Eczema Eczema infantile Eczema nummular Eczema vaccinatum Eczema vesicular Eczema weeping Encephalitis allergic Encephalopathy allergic Eosinophilic granulomatosis with polyangiitis Epidermal necrosis Epidermolysis Epidermolysis bullosa Epiglottic oedema Erythema multiforme Erythema nodosum Exfoliative rash Eye allergy Eye oedema Eye swelling Eyelid oedema Face oedema Fixed eruption Giant papillary conjunctivitis Gingival oedema Gingival swelling Gleich's syndrome Haemorrhagic urticaria Hand dermatitis Henoch-Schonlein purpura Henoch-Schonlein purpura nephritis Heparin-induced thrombocytopenia Hereditary angioedema
Hereditary angioedema with C1 esterase inhibitor deficiency
Hypersensitivity Hypersensitivity myocarditis Hypersensitivity vasculitis


2019 Novo Nordisk 1.0 Final

Pre-defined MedDRA search - list of preferred terms

 ${\tt Pre-defined \ MedDRA \ search}$ 

Preferred term

Idiopathic urticaria

Allergic reactions

Immediate post-injection reaction Immune thrombocytopenic purpura Immune tolerance induction
Immune-mediated adverse reaction Implant site dermatitis
Implant site hypersensitivity Implant site rash Implant site urticaria Incision site dermatitis Incision site rash Infusion related reaction Infusion site dermatitis Infusion site eczema Infusion site hypersensitivity Infusion site rash Infusion site recall reaction Infusion site urticaria Infusion site vasculitis Injection related reaction Injection site dermatitis Injection site eczema Injection site hypersensitivity Injection site rash Injection site recall reaction Injection site urticaria Injection site vasculitis Instillation site hypersensitivity Instillation site rash Instillation site urticaria Interstitial granulomatous dermatitis Intestinal angioedema Iodine allergy Kaposi's varicelliform eruption Kounis syndrome Laryngeal oedema Laryngitis allergic Laryngospasm Laryngotracheal oedema Limbal swelling Lip oedema Lip swelling Mast cell degranulation present Medical device site dermatitis Medical device site eczema Medical device site hypersensitivity Medical device site rash Medical device site recall reaction Medical device site urticaria Mouth swelling Mucocutaneous rash Multiple allergies Nephritis allergic Nikolsky's sign Nodular rash Oculomucocutaneous syndrome Oculorespiratory syndrome Oedema mouth
Oral allergy syndrome
Oropharyngeal blistering
Oropharyngeal oedema Oropharyngeal spasm Oropharyngeal swelling


 Date:
 03 July 2019

 Version:
 1.0

 Status:
 Final

 Page:

Novo Nordisk

 ${\tt Pre-defined} \ {\tt MedDRA} \ {\tt search} \ {\tt -list} \ {\tt of} \ {\tt preferred} \ {\tt terms}$ 

Pre-defined MedDRA search Preferred term Allergic reactions Palatal oedema Palatal swelling Palisaded neutrophilic granulomatous dermatitis Palpable purpura Pathergy reaction Perioral dermatitis Periorbital oedema Periorbital swelling Pharyngeal oedema Procedural shock Pruritus allergic Radioallergosorbent test positive Rash Rash erythematous Rash follicular Rash generalised Rash macular Rash maculo-papular Rash maculovesicular Rash morbilliform Rash neonatal Rash papulosquamous Rash pruritic Rash pustular Rash rubelliform Rash scarlatiniform Rash vesicular Reaction to azo-dyes Reaction to colouring Reaction to excipient Reaction to preservatives Red man syndrome Rhinitis allergic Scleral oedema Scleritis allergic Scrotal oedema Serum sickness Serum sickness-like reaction Shock Shock symptom Skin necrosis Skin reaction Skin test positive Solar urticaria Solvent sensitivity Stevens-Johnson syndrome Stoma site hypersensitivity Stoma site rash Swelling face Swelling of eyelid Swollen tongue
Symmetrical drug-related intertriginous and flexural exanthema Therapeutic product cross-reactivity Tongue oedema Toxic epidermal necrolysis Toxic skin eruption Tracheal oedema Type II hypersensitivity
Type III hypersensitivity
Type III immune complex mediated reaction
Type IV hypersensitivity reaction

Urticaria


Date: Version: Status: Page: 03 July 2019 | Novo Nordisk

1.0 Final 10 of 152

Pre-defined MedDRA search - list of preferred terms

| Preferred term |
|---|
| Urticaria cholinergic |
| Urticaria chronic |
| Urticaria contact |
| Urticaria papular |
| Urticaria physical |
| Urticaria pigmentosa |
| Urticaria vesiculosa |
| Urticarial vasculitis |
| Vaccination site dermatitis |
| Vaccination site eczema |
| Vaccination site exfoliation |
| Vaccination site hypersensitivity |
| Vaccination site rash |
| Vaccination site recall reaction |
| Vaccination site urticaria |
| Vaccination site vasculitis Vaccination site vesicles |
| Vaginal exfoliation |
| Vaginal ulceration Vasculitic rash |
| Vernal keratoconjunctivitis |
| Vessel puncture site rash |
| Vessel puncture site rash Vessel puncture site vesicles |
| Vulval ulceration |
| Vulvovaginal rash |
| Vulvovaginal ulceration |
| Vulvovaginitis allergic |
| varvovagimiero arreigie |
| Antibody test |
| Antibody test abnormal |
| Antibody test positive |
| Autoantibody positive |
| Autoantibody test |
| Drug specific antibody |
| Drug specific antibody present |
| Inhibiting antibodies |
| Neutralising antibodies |
| Neutralising antibodies positive |
| Non-neutralising antibodies positive |
| Through a second of more ment |
| Abnormal precordial movement |
| Accelerated idioventricular rhythm Accessory cardiac pathway |
| Acquired cardiac septal defect |
| Acute aortic syndrome |
| Acute cardiac event |
| Acute coronary syndrome |
| Acute haemorrhagic oedema of infancy |
| Acute kidney injury |
| Acute left ventricular failure |
| Acute myocardial infarction |
| Acute pulmonary oedema |
| Acute respiratory failure |
| Acute right ventricular failure |
| Adams-Stokes syndrome |
| Administration site thrombosis |
| Administration site vasculitis |
| Administration site vasculitis<br>Adrenal thrombosis |
| Administration site vasculitis<br>Adrenal thrombosis<br>Agnosia |
| Administration site vasculitis<br>Adrenal thrombosis<br>Agnosia<br>Agonal rhythm |
| Administration site vasculitis<br>Adrenal thrombosis<br>Agnosia |


 Date:
 03 July 2019

 Version:
 1.0

 Status:
 Final

 Page:

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Cardiovascular disorders Amyloid related imaging abnormalities Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits Amyloid related imaging abnormality-oedema effusion Anaphylactic reaction Anaphylactic shock Anaphylactic transfusion reaction Anaphylactoid reaction Anaphylactoid shock Angina pectoris Angina unstable Anginal equivalent Angiogram abnormal Angiogram cerebral abnormal Angiogram peripheral abnormal Angioplasty Anomalous atrioventricular excitation Anti-neutrophil cytoplasmic antibody positive vasculitis Antibody test abnormal Antibody test positive
Antineutrophil cytoplasmic antibody increased
Antineutrophil cytoplasmic antibody positive Anuria Aortic bypass Aortic embolus Aortic surgery Aortic thrombosis Aortitis Aortogram abnormal Aphasia Application site thrombosis Application site vasculitis Arrhythmia Arrhythmia neonatal Arrhythmia supraventricular Arrhythmogenic right ventricular dysplasia Arterectomy
Arterectomy with graft replacement Arterial angioplasty Arterial bypass occlusion Arterial bypass operation Arterial bypass thrombosis Arterial graft Arterial occlusive disease Arterial stent insertion Arterial therapeutic procedure Arterial thrombosis Arteriogram abnormal Arteriogram carotid abnormal Arteriogram coronary abnormal Arteriosclerosis coronary artery Arteriospasm coronary Arteriotomy Arteriovenous fistula occlusion Arteriovenous fistula thrombosis Arteriovenous graft thrombosis Arteritis Arteritis coronary Artificial blood vessel occlusion Artificial heart implant

Ascites Atherectomy


 Date:
 03 July 2019

 Version:
 1.0

 Status:
 Final

 Page:

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Cardiovascular disorders Atherosclerotic plaque rupture Atrial appendage closure Atrial appendage resection Atrial conduction time prolongation Atrial enlargement Atrial fibrillation Atrial flutter Atrial hypertrophy Atrial natriuretic peptide abnormal Atrial natriuretic peptide increased Atrial parasystole Atrial pressure increased Atrial septal defect acquired Atrial tachycardia Atrial thrombosis Atrioventricular block Atrioventricular block complete Atrioventricular block first degree Atrioventricular block second degree Atrioventricular conduction time shortened Atrioventricular dissociation Atrioventricular node dispersion Autoimmune myocarditis Axillary vein thrombosis Balint's syndrome Basal ganglia haematoma Basal ganglia haemorrhage Basal ganglia infarction Basal ganglia stroke Baseline foetal heart rate variability disorder Basilar artery aneurysm Basilar artery occlusion Basilar artery perforation Basilar artery stenosis Basilar artery thrombosis Behcet's syndrome Bendopnoea Bezold-Jarisch reflex Bifascicular block Biopsy heart abnormal Blindness transient Blood brain barrier defect Blood creatine phosphokinase MB abnormal Blood creatine phosphokinase MB increased Blood creatine phosphokinase abnormal Blood creatine phosphokinase increased Blood pressure diastolic abnormal Blood pressure diastolic decreased Blood pressure diastolic increased Blood pressure fluctuation Blood pressure immeasurable Blood pressure inadequately controlled Blood pressure systolic abnormal Blood pressure systolic decreased Blood pressure systolic increased Blood viscosity increased Bone infarction Brachiocephalic arteriosclerosis Brachiocephalic artery occlusion Brachiocephalic artery stenosis Brachiocephalic vein occlusion

Brachiocephalic vein thrombosis

Bradyarrhythmia


03 July 2019 Novo Nordisk

1.0 Final 13 of 152

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term

Cardiovascular disorders

Bradycardia Bradycardia foetal Bradycardia neonatal Brain hypoxia Brain injury Brain natriuretic peptide abnormal Brain natriuretic peptide increased Brain stem embolism Brain stem haematoma

Brain stem haemorrhage Brain stem infarction Brain stem ischaemia Brain stem microhaemorrhage

Brain stem stroke Brain stem thrombosis Brain stent insertion

Brugada syndrome Budd-Chiari syndrome Bundle branch block Bundle branch block bilateral

Bundle branch block left Bundle branch block right CADASIL

CARASIL syndrome

CSF bilirubin positive CSF red blood cell count positive

CT hypotension complex

Capillaritis

Capsular warning syndrome Cardiac amyloidosis Cardiac aneurysm Cardiac arrest

Cardiac arrest neonatal

Cardiac asthma

Cardiac cirrhosis

Cardiac contractility modulation therapy

Cardiac death

Cardiac dysfunction

Cardiac electrophysiologic study abnormal

Cardiac failure Cardiac failure acute Cardiac failure chronic

Cardiac failure congestive Cardiac failure high output

Cardiac fibrillation Cardiac flutter

Cardiac function test abnormal

Cardiac hypertrophy

Cardiac imaging procedure abnormal

Cardiac index abnormal Cardiac index decreased

Cardiac index increased Cardiac iron overload Cardiac monitoring abnormal

Cardiac operation

Cardiac output decreased Cardiac pseudoaneurysm

Cardiac resynchronisation therapy

Cardiac sarcoidosis

Cardiac septal hypertrophy Cardiac stress test abnormal Cardiac telemetry abnormal

Cardiac ventricular scarring


Final 14 of 152

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Cardiac ventricular thrombosis

Cardiovascular disorders

Cardiac ventriculogram abnormal Cardiac ventriculogram left abnormal Cardiac ventriculogram right abnormal Cardio-respiratory arrest Cardio-respiratory arrest neonatal Cardio-respiratory distress Cardiogenic shock Cardiomegaly Cardiomyopathy Cardiomyopathy acute Cardiomyopathy alcoholic Cardiomyopathy neonatal Cardiopulmonary exercise test abnormal Cardiopulmonary failure Cardiorenal syndrome Cardiothoracic ratio increased Cardiotoxicity Cardiovascular disorder Cardiovascular event prophylaxis Cardiovascular function test abnormal Cardiovascular insufficiency Carotid aneurysm rupture Carotid angioplasty Carotid arterial embolus Carotid arteriosclerosis Carotid artery aneurysm Carotid artery bypass Carotid artery disease Carotid artery dissection Carotid artery dolichoectasia Carotid artery insufficiency Carotid artery occlusion Carotid artery perforation Carotid artery restenosis Carotid artery stenosis Carotid artery stent insertion Carotid artery stent removal Carotid artery thrombosis Carotid endarterectomy Carotid revascularisation Catheter site thrombosis Catheterisation venous Cavernous sinus thrombosis Central bradycardia Central nervous system haemorrhage Central nervous system vasculitis Central pain syndrome Central venous catheterisation Central venous pressure increased Cerebellar artery occlusion Cerebellar artery thrombosis Cerebellar embolism Cerebellar haematoma Cerebellar haemorrhage Cerebellar infarction Cerebellar ischaemia Cerebellar microhaemorrhage Cerebellar stroke Cerebral amyloid angiopathy Cerebral aneurysm perforation Cerebral aneurysm ruptured syphilitic

Cerebral arteriosclerosis


Page:

1.0 Final 15 of 152

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Cardiovascular disorders Cerebral arteriovenous malformation haemorrhagic Cerebral arteritis Cerebral artery embolism Cerebral artery occlusion Cerebral artery perforation Cerebral artery restenosis Cerebral artery stenosis Cerebral artery thrombosis Cerebral capillary telangiectasia Cerebral circulatory failure Cerebral congestion Cerebral endovascular aneurysm repair Cerebral gas embolism Cerebral haematoma Cerebral haemorrhage Cerebral haemorrhage foetal Cerebral haemorrhage neonatal Cerebral haemosiderin deposition Cerebral hypoperfusion Cerebral infarction Cerebral infarction foetal Cerebral ischaemia Cerebral microangiopathy Cerebral microembolism Cerebral microhaemorrhage Cerebral reperfusion injury Cerebral revascularisation Cerebral septic infarct Cerebral small vessel ischaemic disease Cerebral thrombosis Cerebral vascular occlusion Cerebral vasoconstriction Cerebral venous thrombosis Cerebral ventricular rupture Cerebrospinal thrombotic tamponade Cerebrovascular accident Cerebrovascular accident prophylaxis Cerebrovascular arteriovenous malformation Cerebrovascular disorder Cerebrovascular insufficiency Cerebrovascular operation Cerebrovascular stenosis Chagas' cardiomyopathy Charcot-Bouchard microaneurysms Chest X-ray abnormal Chest pain Choroidal infarction Chronic left ventricular failure Chronic right ventricular failure
Chronic right ventricular failure
Chronotropic incompetence
Circulatory collapse
Coeliac artery occlusion Cogan's syndrome Collateral circulation Compression garment application Computerised tomogram coronary artery abnormal Computerised tomogram thorax abnormal Conduction disorder Congenital cerebrovascular anomaly Congenital hemiparesis Congestive cardiomyopathy Cor pulmonale


Date: Version: Status: Page: 03 July 2019


2019 Novo Nordisk 1.0 Final

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Cor pulmonale acute

Echocardiogram abnormal

Cardiovascular disorders

Cor pulmonale chronic Cor pulmonale chronic
Coronary angioplasty
Coronary arterial stent insertion
Coronary artery bypass
Coronary artery compression
Coronary artery disease
Coronary artery dissection
Coronary artery embolism Coronary artery embolism
Coronary artery insufficiency
Coronary artery occlusion
Coronary artery reocclusion
Coronary artery restenosis Coronary artery restenosis
Coronary artery stenosis
Coronary artery surgery
Coronary artery thrombosis
Coronary brachytherapy
Coronary bypass stenosis
Coronary bypass thrombosis
Coronary endarterectomy Coronary no-reflow phenomenon Coronary ostial stenosis Coronary revascularisation Coronary vascular graft occlusion Coronary vascular graft stenosis Coxsackie carditis Coxsackie myocarditis Cryoglobulinaemia Cryoglobulins present Cutaneous vasculitis Cytomegalovirus myocarditis Cytotoxic cardiomyopathy Decreased ventricular preload Deep vein thrombosis Deep vein thrombosis postoperative Defect conduction intraventricular Delayed ischaemic neurological deficit Device embolisation Device occlusion Device related thrombosis Diabetic arteritis Diabetic cardiomyopathy Diabetic coronary microangiopathy Diastolic dysfunction Diffuse vasculitis Dilatation atrial Dilatation ventricular Diplegia Directional Doppler flow tests abnormal Dissecting coronary artery aneurysm Disseminated intravascular coagulation Disseminated intravascular coagulation in newborn Distributive shock Dural arteriovenous fistula Dysarthria Dyspnoea Dyspnoea paroxysmal nocturnal ECG P wave inverted
ECG electrically inactive area
ECG signs of myocardial infarction
ECG signs of myocardial ischaemia
ECG signs of ventricular hypertrophy


1.0 Final 17 of 152 Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Cardiovascular disorders Ejection fraction abnormal Ejection fraction decreased Electrocardiogram P wave abnormal Electrocardiogram PQ interval prolonged Electrocardiogram PQ interval shortened Electrocardiogram PR prolongation Electrocardiogram PR segment depression Electrocardiogram PR shortened Electrocardiogram Q wave abnormal Electrocardiogram QRS complex prolonged Electrocardiogram QT interval abnormal Electrocardiogram QT prolonged Electrocardiogram RR interval prolonged Electrocardiogram ST segment abnormal Electrocardiogram ST segment depression Electrocardiogram ST segment elevation Electrocardiogram ST-T segment abnormal Electrocardiogram ST-T segment depression Electrocardiogram ST-T segment elevation Electrocardiogram T wave abnormal Electrocardiogram T wave inversion Electrocardiogram U wave inversion Electrocardiogram U wave present Electrocardiogram U-wave abnormality Electrocardiogram abnormal Electrocardiogram ambulatory abnormal Electrocardiogram change Electrocardiogram delta waves abnormal Electrocardiogram repolarisation abnormality Embolia cutis medicamentosa Embolic cerebral infarction Embolic pneumonia Embolic stroke Embolism Embolism arterial Embolism venous Endarterectomy Endocardial fibroelastosis Endotoxic shock Eosinophilic granulomatosis with polyangiitis Eosinophilic myocarditis Epidural haemorrhage Erythema induratum Exercise electrocardiogram abnormal Exercise test abnormal External counterpulsation Extra-axial haemorrhage Extradural haematoma Extraischaemic cerebral haematoma Extrasystoles Femoral artery embolism Foetal arrhythmia Foetal cerebrovascular disorder Foetal heart rate acceleration abnormality Foetal heart rate deceleration abnormality Foetal heart rate disorder Foetal tachyarrhythmia Gonococcal heart disease Goodpasture's syndrome Graft thrombosis Granulomatosis with polyangiitis

Grey syndrome neonatal HIV cardiomyopathy


Final

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Haemorrhage coronary artery Haemorrhage intracranial

Cardiovascular disorders

Haemorrhagic adrenal infarction Haemorrhagic cerebral infarction Haemorrhagic infarction Haemorrhagic stroke Haemorrhagic transformation stroke Haemorrhagic vasculitis Haemorrhoids thrombosed Heart alternation Heart and lung transplant Heart block congenital Heart rate abnormal Heart rate decreased Heart rate increased Heart rate irregular Heart transplant Hemianaesthesia Hemiasomatognosia Hemihyperaesthesia Hemiparaesthesia Hemiparesis Hemiplegia Henoch-Schonlein purpura Henoch-Schonlein purpura nephritis Heparin-induced thrombocytopenia Hepatic artery embolism Hepatic artery occlusion Hepatic artery thrombosis Hepatic congestion Hepatic infarction Hepatic vascular thrombosis Hepatic vein dilatation Hepatic vein embolism Hepatic vein occlusion Hepatic vein thrombosis Hepatojugular reflux Hepatorenal failure
Homans' sign positive
Hyperdynamic left ventricle Hypersensitivity myocarditis Hypersensitivity vasculitis Hypertensive cardiomyopathy Hypertensive cerebrovascular disease Hypertrophic cardiomyopathy Hypoperfusion Hypothenar hammer syndrome Hypovolaemic shock Hypoxic-ischaemic encephalopathy Iliac artery  $\operatorname{embolism}$ Iliac artery occlusion Iliac vein occlusion Implant site thrombosis Incision site vessel occlusion Increased ventricular preload Infarction Inferior vena cava syndrome Inferior vena caval occlusion Infusion site thrombosis Infusion site vasculitis Injection site thrombosis

Injection site vasculitis


03 July 2019

Novo Nordisk 1.0 Final 19 of 152

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Cardiovascular disorders

Inner ear infarction Instillation site thrombosis Internal carotid artery kinking Intestinal infarction Intra-aortic balloon placement Intra-cerebral aneurysm operation Intracardiac mass Intracardiac pressure increased Intracardiac thrombus Intracerebral haematoma evacuation Intracranial aneurysm Intracranial artery dissection Intracranial haematoma Intracranial tumour haemorrhage Intracranial venous sinus thrombosis Intraoperative cerebral artery occlusion Intraventricular haemorrhage Intraventricular haemorrhage neonatal Irregular breathing
Ischaemic cardiomyopathy Ischaemic cerebral infarction Ischaemic mitral regurgitation Ischaemic stroke Jugular vein distension Jugular vein occlusion Jugular vein thrombosis Junctional ectopic tachycardia Kawasaki's disease Kounis syndrome Labile blood pressure Lacunar infarction Lacunar stroke Langerhans' cell histiocytosis Lateral medullary syndrome Lateropulsion Left atrial dilatation Left atrial enlargement Left ventricular diastolic collapse Left ventricular dilatation Left ventricular dysfunction Left ventricular end-diastolic pressure decreased Left ventricular enlargement Left ventricular failure Left ventricular heave Lenegre's disease Leriche syndrome Long QT syndrome Long QT syndrome congenital Loss of consciousness Low cardiac output syndrome Lower respiratory tract congestion Lown-Ganong-Levine syndrome Lupus myocarditis Lupus vasculitis Lyme carditis MAGIC syndrome Mahler sign Malarial myocarditis May-Thurner syndrome Medical device site thrombosis Medical device site vasculitis Meningorrhagia

Mental status changes


1.0 Final 20 of 152 Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Nodular vasculitis

Cardiovascular disorders

Mesenteric arterial occlusion Mesenteric arteriosclerosis Mesenteric artery embolism Mesenteric artery stenosis Mesenteric artery stent insertion Mesenteric artery thrombosis Mesenteric vascular insufficiency Mesenteric vascular occlusion Mesenteric vein thrombosis Mesenteric venous occlusion Metabolic cardiomyopathy Microembolism Microscopic polyangiitis Microvascular coronary artery disease Migrainous infarction Millard-Gubler syndrome Modified Rankin score decreased Modified Rankin score increased Monoparesis Monoplegia Moyamoya disease Multiple gated acquisition scan abnormal Multiple organ dysfunction syndrome Myocardiac abscess Myocardial calcification Myocardial depression Myocardial fibrosis Myocardial haemorrhage Myocardial hypoxia Myocardial infarction Myocardial ischaemia Mvocardial necrosis Myocardial necrosis marker increased Myocardial reperfusion injury Myocardial stunning Myocarditis Myocarditis bacterial Myocarditis helminthic Myocarditis infectious Myocarditis meningococcal Myocarditis mycotic Myocarditis post infection Myocarditis septic Myocarditis syphilitic Myocarditis toxoplasmal Myoglobinaemia Myoglobinuria N-terminal prohormone brain natriuretic peptide abnormal N-terminal prohormone brain natriuretic peptide increased NIH stroke scale abnormal NIH stroke scale score decreased NIH stroke scale score increased Neonatal anuria Neonatal cardiac failure Neonatal multi-organ failure Neonatal respiratory failure Neonatal tachycardia Neurogenic shock Nocturia Nocturnal dyspnoea Nodal arrhythmia Nodal rhythm


03 July 2019 Date: Version: Status: Page:

Novo Nordisk

1.0

Final


Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Cardiovascular disorders

Non-obstructive cardiomyopathy Nonreassuring foetal heart rate pattern Nuclear magnetic resonance imaging thoracic abnormal Obesity cardiomyopathy Obstetrical pulmonary embolism Obstructive shock Ocular vasculitis Oedema Oedema blister Oedema due to cardiac disease Oedema neonatal Oedema peripheral Ophthalmic artery thrombosis Ophthalmic vein thrombosis Optic nerve infarction Organ failure Orthopnoea Orthostatic hypotension Ovarian vein thrombosis Pacemaker generated arrhythmia Pacemaker syndrome Paget-Schroetter syndrome Palpable purpura Palpitations Pancreatic infarction Papillary muscle disorder Papillary muscle haemorrhage Papillary muscle infarction Paradoxical embolism Paralysis Paraneoplastic thrombosis Paraparesis Paraplegia Parasystole Paresis Paroxysmal arrhythmia Paroxysmal atrioventricular block Pelvic venous thrombosis Penile artery occlusion Penile vein thrombosis Percutaneous coronary intervention Perinatal stroke Peripartum cardiomyopathy Peripheral arterial occlusive disease Peripheral arterial reocclusion Peripheral artery angioplasty Peripheral artery bypass Peripheral artery occlusion Peripheral artery stent insertion Peripheral artery thrombosis Peripheral embolism Peripheral endarterectomy Peripheral oedema neonatal Peripheral revascularisation Peripheral swelling Periprocedural myocardial infarction Periventricular haemorrhage neonatal Phlebectomy Pituitary haemorrhage Pituitary infarction Placental infarction Plasma viscosity abnormal

Pneumatic compression therapy


Date: 03 July 2019 Version: 1.0 Status: Final

Final 22 of 152

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Cardiovascular disorders

Polyarteritis nodosa Polymyalgia rheumatica Popliteal artery entrapment syndrome Portal shunt procedure Portal vein cavernous transformation Portal vein occlusion Portal vein thrombosis Portosplenomesenteric venous thrombosis Post angioplasty restenosis Post cardiac arrest syndrome Post procedural myocardial infarction Post procedural pulmonary embolism
Post procedural stroke Post stroke depression Post thrombotic syndrome Posthaemorrhagic hydrocephalus Postinfarction angina Postoperative thrombosis Postpartum thrombosis Postpartum venous thrombosis Precerebral arteriosclerosis Precerebral artery occlusion Precerebral artery thrombosis Prerenal failure Primary familial brain calcification Prinzmetal angina Procedural shock Profundaplasty Prohormone brain natriuretic peptide abnormal Prohormone brain natriuretic peptide increased Propofol infusion syndrome Prosthetic cardiac valve thrombosis Prosthetic vessel implantation Pseudovasculitis Pulmonary arterial wedge pressure increased Pulmonary artery occlusion
Pulmonary artery therapeutic procedure Pulmonary artery thrombosis Pulmonary congestion Pulmonary embolism Pulmonary endarterectomy Pulmonary infarction Pulmonary microemboli
Pulmonary oedema
Pulmonary oedema neonatal
Pulmonary thrombosis Pulmonary tumour thrombotic microangiopathy Pulmonary vasculitis Pulmonary vein occlusion Pulmonary veno-occlusive disease Pulmonary venous thrombosis Pulse absent Pulseless electrical activity Putamen haemorrhage Quadriparesis Quadriplegia Radiation associated cardiac failure Radiation myocarditis Radiation vasculitis Rebound tachycardia Renal arteritis Renal artery angioplasty

Renal artery occlusion

Page:


Page:

Novo Nordisk

1.0

Final


Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Cardiovascular disorders

```
Renal artery thrombosis
Renal embolism
Renal failure
Renal failure neonatal
Renal infarct
Renal vascular thrombosis
Renal vasculitis
Renal vein embolism
Renal vein occlusion
Renal vein thrombosis
Reperfusion arrhythmia
Respiratory failure
Respiratory sinus arrhythmia magnitude abnormal
Respiratory sinus arrhythmia magnitude decreased
Respiratory sinus arrhythmia magnitude increased
Restrictive cardiomyopathy
Retinal artery embolism
Retinal artery occlusion
Retinal artery thrombosis
Retinal infarction
Retinal vascular thrombosis
Retinal vasculitis
Retinal vein occlusion
Retinal vein thrombosis
Retrograde p-waves
Reversible cerebral vasoconstriction syndrome
Reversible ischaemic neurological deficit
Rheumatoid vasculitis
Rhythm idioventricular
Right atrial dilatation
Right atrial enlargement
Right atrial pressure increased
Right hemisphere deficit syndrome
Right ventricle outflow tract obstruction
Right ventricular diastolic collapse
Right ventricular dilatation
Right ventricular dysfunction
Right ventricular ejection fraction decreased Right ventricular enlargement
Right ventricular failure
Right ventricular heave
Right ventricular systolic pressure decreased
Ruptured cerebral aneurysm
SI QIII TIII pattern
Scan myocardial perfusion abnormal 
Segmented hyalinising vasculitis
Septic shock
Shock
Shock haemorrhagic
Shock hypoglycaemic
Shock symptom
Shunt occlusion
Shunt thrombosis
Silent myocardial infarction
Sinoatrial block
Sinus arrest
Sinus arrhythmia
Sinus bradycardia
Sinus node dysfunction
Sinus tachycardia
Sneddon's syndrome
Spinal artery embolism
```

Spinal artery thrombosis


Page:

Novo Nordisk

1.0

Final


Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Spinal cord haematoma

Cardiovascular disorders

```
Spinal cord haemorrhage
Spinal cord infarction
Spinal cord ischaemia
Spinal epidural haematoma
Spinal epidural haemorrhage
Spinal subarachnoid haemorrhage
Spinal subdural haematoma
Spinal subdural haemorrhage
Spinal vascular disorder
Spinal vessel congenital anomaly
Splenic artery thrombosis
Splenic embolism
Splenic infarction
Splenic thrombosis
Splenic vein occlusion
Splenic vein thrombosis
Stoma site thrombosis
Stress cardiomyopathy
Stress echocardiogram abnormal
Stroke in evolution
Stroke volume decreased
Subarachnoid haematoma
Subarachnoid haemorrhage
Subarachnoid haemorrhage neonatal
Subclavian artery embolism Subclavian artery occlusion
Subclavian artery thrombosis
Subclavian coronary steal syndrome
Subclavian steal syndrome
Subclavian vein occlusion
Subclavian vein thrombosis
Subdural haematoma
Subdural haematoma evacuation
Subdural haemorrhage
Subdural haemorrhage neonatal
Subendocardial ischaemia
Sudden cardiac death
Sudden death
Superficial siderosis of central nervous system
Superior sagittal sinus thrombosis
Superior vena cava occlusion
Superior vena cava syndrome
Supraventricular extrasystoles
Supraventricular tachyarrhythmia
Supraventricular tachycardia
Surgical vascular shunt
Surgical ventricular restoration
Susac's syndrome
Syncope
Systolic anterior motion of mitral valve
Systolic dysfunction
Tachyarrhythmia
Tachycardia
Tachycardia foetal
Tachycardia induced cardiomyopathy
Tachycardia paroxysmal
Takayasu's arteritis
Temporal arteritis
Testicular infarction
Thalamic infarction
Thalamus haemorrhage
Thrombectomy
```


1.0 Final 25 of 152 Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Thromboangiitis obliterans

Cardiovascular disorders

Thromboembolectomy Thrombolysis Thrombophlebitis Thrombophlebitis migrans Thrombophlebitis neonatal Thrombophlebitis superficial Thrombosed varicose vein Thrombosis Thrombosis corpora cavernosa Thrombosis in device Thrombosis mesenteric vessel Thrombosis prophylaxis
Thrombotic cerebral infarction Thrombotic microangiopathy Thrombotic stroke Thrombotic thrombocytopenic purpura Thyroid infarction Thyrotoxic cardiomyopathy
Torsade de pointes Toxic shock syndrome Transient ischaemic attack Transverse sinus thrombosis Trifascicular block Troponin I increased Troponin T increased Troponin increased Truncus coeliacus thrombosis Tumour embolism Tumour thrombosis Type 2 lepra reaction Ultrasonic angiogram abnormal Ultrasound Doppler abnormal Umbilical cord occlusion Umbilical cord thrombosis Urticarial vasculitis Vaccination site thrombosis Vaccination site vasculitis Vascular access site thrombosis Vascular device occlusion Vascular encephalopathy Vascular graft Vascular graft occlusion Vascular graft thrombosis Vascular operation Vascular pseudoaneurysm thrombosis Vascular purpura Vascular resistance pulmonary increased Vascular stent insertion Vascular stent occlusion Vascular stent stenosis Vascular stent thrombosis Vasculitic rash Vasculitis Vasculitis gastrointestinal Vasculitis necrotising Vasodilation procedure Vein of Galen aneurysmal malformation Vena cava embolism Vena cava filter insertion Vena cava filter removal Vena cava thrombosis

Venogram abnormal

MedDRA version 21.1


Date: Version: Status: 03 July 2019 1.0

Novo Nordisk

Status: Final 

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Cardiovascular disorders Venoocclusive disease Venoocclusive liver disease Venous angioplasty Venous occlusion Venous operation Venous pressure increased Venous pressure jugular abnormal Venous pressure jugular increased Venous recanalisation Venous repair Venous stent insertion Venous thrombosis Venous thrombosis in pregnancy Venous thrombosis limb Venous thrombosis neonatal Ventricular arrhythmia Ventricular assist device insertion Ventricular asystole Ventricular compliance decreased Ventricular dysfunction Ventricular dyskinesia Ventricular dyssynchrony Ventricular enlargement Ventricular extrasystoles Ventricular failure Ventricular fibrillation Ventricular flutter Ventricular hyperkinesia Ventricular hypertrophy Ventricular hypokinesia Ventricular parasystole Ventricular pre-excitation Ventricular remodelling Ventricular septal defect acquired Ventricular tachyarrhythmia Ventricular tachycardia Vertebral artery aneurysm
Vertebral artery dissection
Vertebral artery occlusion
Vertebral artery perforation
Vertebral artery stenosis
Vertebral artery thrombosis
Vertebral artery thrombosis Vertebrobasilar dolichoectasia Vertebrobasilar insufficiency Vessel puncture site occlusion Vessel puncture site thrombosis Viral cardiomyopathy Viral myocarditis Viral vasculitis Visceral venous thrombosis Visual acuity reduced transiently Visual agnosia Visual midline shift syndrome Wall motion score index abnormal Wandering pacemaker Wellens' syndrome Withdrawal arrhythmia Wolff-Parkinson-White syndrome Wolff-Parkinson-White syndrome congenital Diabetic retinopathy Phase 3a search Amaurosis Cystoid macular oedema

Diabetic blindness


1.0 Final

Novo Nordisk

 ${\tt Pre-defined} \ {\tt MedDRA} \ {\tt search} \ {\tt -list} \ {\tt of} \ {\tt preferred} \ {\tt terms}$ 

Pre-defined MedDRA search Preferred term Diabetic retinopathy Phase 3a search Diabetic eye disease Diabetic glaucoma Diabetic retinal oedema Diabetic retinopathy Diabetic uveitis Exudative retinopathy Macular ischaemia Macular oedema Macular opacity Macular pseudohole Maculopathy Night blindness Papilloedema Papillophlebitis Retinal deposits Retinal detachment Retinal exudates Retinal haemorrhage Retinal ischaemia Retinal neovascularisation Retinal oedema Retinal pallor Retinal vascular occlusion Retinopathy Retinopathy proliferative Sudden visual loss Visual acuity reduced Visual acuity reduced transiently Vitreal cells Vitreous detachment Vitreous haemorrhage Vitreous opacities Gastrointestinal adverse events Abdominal adhesions Abdominal compartment syndrome Abdominal discomfort Abdominal distension Abdominal fat apron Abdominal hernia Abdominal hernia obstructive Abdominal hernia perforation Abdominal incarcerated hernia Abdominal mass Abdominal magraine Abdominal pain Abdominal pain lower Abdominal pain upper Abdominal rebound tenderness Abdominal rigidity
Abdominal strangulated hernia Abdominal symptom Abdominal tenderness Abdominal wall cyst Abdominal wall disorder Abdominal wall haematoma Abdominal wall haemorrhage Abdominal wall mass Abnormal faeces Acetonaemic vomiting Achlorhydria Acid peptic disease Acquired macroglossia Acquired oesophageal web


03 July 2019 Novo Nordisk 1.0

Final 28 of 152

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Gastrointestinal adverse events

Acute abdomen Acute haemorrhagic ulcerative colitis Acute oesophageal mucosal lesion Aerophagia Alcoholic pancreatitis Alcoholic pancreopathy Allergic colitis

Allergic gastroenteritis Allergic stomatitis Alveolar bone resorption

Amalgam tattoo Ampullary polyp Anal dilatation Anal erosion Anal fissure

Anal fissure haemorrhage Anal fistula

Anal haemorrhage Anal hypoaesthesia Anal incontinence Anal inflammation Anal leukoplakia Anal paraesthesia

Anal polyp Anal prolapse Anal pruritus Anal skin tags Anal spasm

Anal sphincter atony Anal sphincter hypertonia

Anal stenosis Anal trichiasis Anal ulcer

Anal ulcer haemorrhage Anastomotic ulcer perforation

Anastomotic ulcer, obstructive Angina bullosa haemorrhagica

Ankyloglossia acquired Anogenital dysplasia Anorectal discomfort Anorectal disorder Anorectal sensory loss

Anorectal squamous cell metaplasia

Anorectal stenosis Anorectal swelling Anorectal ulcer Anorectal varices

Anorectal varices haemorrhage Anovulvar fistula Aorto-oesophageal fistula

Aortoenteric fistula Aphthous ulcer Apical granuloma Apoptotic colonopathy Appendiceal mucocoele Appendicitis noninfective

Appendicolith Appendix disorder Aptyalism Ascites

Atrophic glossitis Auriculotemporal syndrome

Autoimmune colitis


Final

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Autoimmune enteropathy

Gastrointestinal adverse events

Autoimmune pancreatitis Barrett's oesophagus Bezoar Bile acid malabsorption Biliary ascites Bloody peritoneal effluent Bowel movement irregularity Breath odour Brunner's gland hyperplasia Buccal mucosal roughening Buccal polyp
Buccoglossal syndrome Burning mouth syndrome Cardiospasm Cascade stomach Cemento osseous dysplasia Change of bowel habit Chapped lips Cheilitis Cheilitis granulomatosa Cheilosis Chilaiditi's syndrome Chronic cheek biting Chronic gastritis Chronic gastrointestinal bleeding Coating in mouth Cobble stone tongue Coeliac artery aneurysm
Coeliac artery compression syndrome
Coeliac artery stenosis
Coeliac disease Colitis Colitis cystica profunda Colitis erosive Colitis ischaemic Colitis microscopic Colitis psychogenic Colitis ulcerative Colon dysplasia Colonic fistula Colonic haematoma Constipation Contact stomatitis Creatorrhoea Cricopharyngeal achalasia Crohn's disease Cronkhite-Canada syndrome Cryptitis Cyclic vomiting syndrome Defaecation disorder Defaecation urgency Dental abfraction
Dental alveolar anomaly Dental caries Dental cyst Dental discomfort Dental dysaesthesia Dental necrosis Dental paraesthesia Dental plaque Dental pulp disorder

Diabetic enteropathy


Date: Version: Status:

Page:

03 July 2019 Novo Nordisk 1.0 Final


Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Gastrointestinal adverse events Diabetic gastroenteropathy Diabetic gastroparesis Diabetic gastropathy Diaphragmatic hernia Diaphragmatic hernia, obstructive Diarrhoea Diarrhoea haemorrhagic Diarrhoea neonatal Diastema Dieulafoy's vascular malformation Discoloured vomit Distal intestinal obstruction syndrome Diverticular fistula Diverticular hernia Diverticular perforation Diverticulitis oesophageal Diverticuloma Diverticulum Diverticulum gastric Diverticulum intestinal Diverticulum intestinal haemorrhagic Diverticulum oesophageal Dolichocolon acquired Douglas' pouch mass Dry mouth Dumping syndrome Duodenal obstruction Duodenal papillitis Duodenal perforation Duodenal polyp Duodenal stenosis Duodenal ulcer Duodenal ulcer haemorrhage Duodenal ulcer perforation Duodenal ulcer perforation, obstructive Duodenal ulcer, obstructive Duodenal varices Duodenal vascular ectasia Duodenitis Duodenitis haemorrhagic Duodenogastric reflux Dysbactériosis Dyschezia Dyskinesia oesophageal Dyspepsia Dysphagia Dysphagia lusoria Entopic gastric mucosa
Enamel anomaly
Encapsulating peritoneal sclerosis Enlarged uvula Enteric neuropathy Enteritis Enteritis leukopenic Enterocele Enterochromaffin cell hyperplasia Enterocolitis Enterocolitis haemorrhagic Enterocolonic fistula Enterocutaneous fistula Enterovesical fistula Eosinophilic colitis

Eosinophilic oesophagitis


03 July 2019 Novo Nordisk 1.0

Final 31 of 152

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Epigastric discomfort

Gastrointestinal adverse events

Epiploic appendagitis Epulis Erosive duodenitis Erosive oesophagitis Eructation
Faecal vomiting Faecalith Faecaloma Faeces discoloured Faeces hard Faeces pale Faeces soft Feline oesophagus Femoral hernia Femoral hernia incarcerated Femoral hernia strangulated Femoral hernia, obstructive Fibrosing colonopathy
Fistula of small intestine Fixed bowel loop Flatulence Fluorosis dental Food poisoning Frequent bowel movements Functional gastrointestinal disorder Gallstone ileus Gastric antral vascular ectasia Gastric atony Gastric cyst Gastric dilatation Gastric disorder Gastric dysplasia Gastric fibrosis Gastric fistula Gastric haemorrhage Gastric hypermotility Gastric hypertonia Gastric hypomotility Gastric ileus Gastric mucosa erythema Gastric mucosal calcinosis Gastric mucosal hypertrophy Gastric mucosal lesion Gastric perforation Gastric pneumatosis Gastric polyps Gastric prolapse Gastric stenosis Gastric ulcer Gastric ulcer haemorrhage Gastric ulcer haemorrhage, obstructive Gastric ulcer perforation Gastric ulcer perforation, obstructive Gastric ulcer, obstructive Gastric varices Gastric varices haemorrhage Gastric volvulus Gastric xanthoma Gastritis Gastritis alcoholic Gastritis alcoholic haemorrhagic

Gastritis erosive

Pre-defined MedDRA search


Preferred term


Final 32 of 152

 ${\tt Pre-defined} \ {\tt MedDRA} \ {\tt search} \ {\tt -list} \ {\tt of} \ {\tt preferred} \ {\tt terms}$ 

Gastrointestinal adverse events Gastritis haemorrhagic Gastritis hypertrophic Gastrocoele Gastroduodenal haemorrhage Gastroduodenal ulcer Gastroenteritis eosinophilic Gastrointestinal amyloidosis Gastrointestinal angiectasia Gastrointestinal angiodysplasia Gastrointestinal disorder Gastrointestinal dysplasia Gastrointestinal erosion Gastrointestinal fistula Gastrointestinal haemorrhage Gastrointestinal hypermotility Gastrointestinal hypomotility Gastrointestinal inflammation Gastrointestinal ischaemia Gastrointestinal melanosis Gastrointestinal motility disorder Gastrointestinal mucocoele Gastrointestinal mucosa hyperaemia Gastrointestinal mucosal disorder Gastrointestinal mucosal exfoliation Gastrointestinal mucosal necrosis Gastrointestinal necrosis Gastrointestinal obstruction Gastrointestinal oedema Gastrointestinal pain Gastrointestinal perforation Gastrointestinal polyp Gastrointestinal polyp haemorrhage Gastrointestinal scarring
Gastrointestinal sounds abnormal Gastrointestinal stenosis Gastrointestinal toxicity Gastrointestinal tract irritation Gastrointestinal tract mucosal discolouration Gastrointestinal tract mucosal pigmentation Gastrointestinal ulcer Gastrointestinal ulcer haemorrhage Gastrointestinal ulcer perforation Gastrointestinal vascular malformation Gastrointestinal vascular malformation haemorrhagic Gastrointestinal wall abnormal Gastrointestinal wall thickening Gastrointestinal wall thinning Gastrolithiasis Gastrooesophageal reflux disease Gastrooesophageal sphincter insufficiency Gastropleural fistula Gastroptosis Gastrosplenic fistula Giant cell epulis

Gingival atrophy
Gingival bleeding
Gingival blister
Gingival cyst
Gingival discolouration
Gingival discomfort
Gingival disorder
Gingival erosion
Gingival erythema


03 July 2019 1.0

Final 33 of 152

Novo Nordisk

 ${\tt Pre-defined} \ {\tt MedDRA} \ {\tt search} \ {\tt -list} \ {\tt of} \ {\tt preferred} \ {\tt terms}$ 

Pre-defined MedDRA search Preferred term Gastrointestinal adverse events Gingival hyperpigmentation Gingival hypertrophy Gingival hypoplasia Gingival oedema Gingival pain Gingival polyp Gingival pruritus Gingival recession Gingival swelling Gingival ulceration Gingivitis ulcerative Glossitis Glossodynia Glossoptosis Glycogenic acanthosis Gut fermentation syndrome Haematemesis Haematochezia Haemorrhagic ascites Haemorrhagic erosive gastritis Haemorrhagic necrotic pancreatitis Haemorrhoidal haemorrhage Haemorrhoids Haemorrhoids thrombosed Hernial eventration Heyde's syndrome Hiatus hernia Hiatus hernia strangulated Hiatus hernia, obstructive Hypercementosis Hyperchlorhydria Hypergastrinaemia Hypertrophic anal papilla Hypertrophy of tongue papillae Hypoaesthesia oral Hypoaesthesia teeth Ileal perforation Ileal stenosis Ileal ulcer Ileal ulcer perforation Ileus Ileus paralytic Ileus spastic Impaired gastric emptying Incarcerated hiatus hernia Incarcerated inguinal hernia Incarcerated umbilical hernia Infantile colic Infantile spitting up Infantile vomiting Inflammatory bowel disease Infrequent bowel movements
Inguinal hernia
Inguinal hernia perforation Inguinal hernia strangulated Inguinal hernia, obstructive Internal hernia Intestinal angina Intestinal angioedema Intestinal calcification Intestinal congestion

Intestinal cyst

Intestinal diaphragm disease


 Date:
 03 July 2019

 Version:
 1.0

 Status:
 Final

2019 Novo Nordisk 1.0 Final


 ${\tt Pre-defined} \ {\tt MedDRA} \ {\tt search} \ {\tt -list} \ {\tt of} \ {\tt preferred} \ {\tt terms}$ 

Pre-defined MedDRA search Preferred term Gastrointestinal adverse events Intestinal dilatation Intestinal fibrosis Intestinal fistula Intestinal haematoma Intestinal haemorrhage Intestinal infarction Intestinal ischaemia Intestinal mass Intestinal metaplasia Intestinal mucosal atrophy Intestinal mucosal hypertrophy Intestinal obstruction Intestinal perforation Intestinal polyp Intestinal prolapse Intestinal pseudo-obstruction Intestinal smooth muscle hypertrophy Intestinal steatosis Intestinal stenosis Intestinal strangulation Intestinal ulcer Intestinal ulcer perforation Intestinal varices Intestinal varices haemorrhage
Intestinal villi atrophy
Intra-abdominal fluid collection
Intra-abdominal haematoma Intra-abdominal haemorrhage Intrinsic factor deficiency Intussusception Irritable bowel syndrome Ischaemic enteritis Ischaemic gastritis Ischaemic pancreatitis Ischiatic hernia Ischiorectal hernia Jejunal perforation Jejunal stenosis Jejunal ulcer Jejunal ulcer perforation Large intestinal haemorrhage Large intestinal obstruction Large intestinal stenosis Large intestinal ulcer Large intestinal ulcer haemorrhage Large intestinal ulcer perforation Large intestine erosion Large intestine perforation Large intestine polyp Leukoplakia oesophageal Leukoplakia oral Levator syndrome Lip blister Lip discolouration Lip disorder Lip dry Lip erosion Lip erythema Lip exfoliation Lip haematoma Lip haemorrhage Lip oedema Lip pain


2019 Novo Nordisk 1.0 Final

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Gastrointestinal adverse events Lip pruritus Lip swelling Lip ulceration Loose tooth Lower gastrointestinal haemorrhage Lower gastrointestinal perforation Lumbar hernia Lupus enteritis Lupus pancreatitis Lymphangiectasia intestinal Lymphocytic oesophagitis Lymphoid hyperplasia of intestine Malabsorption Malacoplakia gastrointestinal Malignant dysphagia Malignant gastrointestinal obstruction Mallory-Weiss syndrome Malocclusion Malpositioned teeth Mastocytic enterocolitis Mechanical ileus Meconium cyst Meconium ileus Meconium peritonitis Meconium plug syndrome Megacolon Meĺaena Melaena neonatal Melanoplakia oral Mesenteric arterial occlusion  $\begin{array}{ll} {\tt Mesenteric} \ \ {\tt arteriosclerosis} \\ {\tt Mesenteric} \ \ {\tt artery} \ \ {\tt aneurysm} \end{array}$ Mesenteric artery embolism Mesenteric artery stenosis Mesenteric artery thrombosis Mesenteric cyst Mesenteric fibrosis Mesenteric haematoma Mesenteric haemorrhage Mesenteric panniculitis Mesenteric phlebosclerosis Mesenteric vascular insufficiency Mesenteric vascular occlusion Mesenteric vein thrombosis Mesenteric venous occlusion Mesenteritis Mikulicz's disease Mikulicz's syndrome Mouth cyst Mouth haemorrhage Mouth swelling Mouth ulceration Mucous stools Myochosis Narcotic bowel syndrome Nausea Necrotising colitis Necrotising enterocolitis neonatal Necrotising gastritis Necrotising oesophagitis Neonatal gastrointestinal disorder Neonatal gastrointestinal haemorrhage

Neonatal intestinal dilatation


03 July 2019

1.0 Final 36 of 152 Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Neonatal intestinal obstruction

Gastrointestinal adverse events

Neonatal intestinal perforation Neurogenic bowel Neutropenic colitis Nicotinic stomatitis Noninfectious peritonitis Noninfective gingivitis Noninfective sialoadenitis Obstruction gastric Obstructive defaecation Obstructive pancreatitis Obturator hernia Odynophagia Oedema mouth Oedematous pancreatitis Oesophageal achalasia Oesophageal atony Oesophageal compression Oesophageal dilatation Oesophageal discomfort Oesophageal disorder Oesophageal dysplasia Oesophageal fibrosis Oesophageal fistula Oesophageal food impaction Oesophageal haemorrhage Oesophageal hypomotility Oesophageal intramural haematoma Oesophageal irritation Oesophageal mass Oesophageal motility disorder Oesophageal mucosa erythema Oesophageal mucosal blister Oesophageal mucosal dissection Oesophageal mucosal hyperplasia Oesophageal mucosal tear Oesophageal obstruction Oesophageal oedema Oesophageal pain Oesophageal perforation Oesophageal polyp Oesophageal rupture Oesophageal spasm Oesophageal stenosis
Oesophageal stent stenosis Oesophageal ulcer Oesophageal ulcer haemorrhage Oesophageal ulcer perforation Oesophageal varices haemorrhage Oesophagitis Oesophagitis haemorrhagic Oesophagitis ulcerative Oesophagopleural fistula Omental infarction Omental necrosis Oral cavity fistula Oral contusion Oral discharge Oral discomfort Oral disorder Oral dysaesthesia Oral hyperaesthesia Oral hyperkeratosis


Final

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Gastrointestinal adverse events Oral leukoedema Oral lichen planus Oral mucosa atrophy Oral mucosa erosion Oral mucosa haematoma Oral mucosal blistering Oral mucosal discolouration Oral mucosal eruption Oral mucosal erythema Oral mucosal exfoliation Oral mucosal hypertrophy Oral pain Oral papule Oral pigmentation Oral pruritus Oral submucosal fibrosis Oral toxicity Oroantral fistula Palatal disorder Palatal dysplasia Palatal oedema Palatal swelling Palatal ulcer Pancreatic atrophy Pancreatic calcification Pancreatic cyst Pancreatic cyst rupture Pancreatic disorder Pancreatic duct dilatation Pancreatic duct obstruction Pancreatic duct stenosis Pancreatic enlargement Pancreatic enzyme abnormality Pancreatic failure Pancreatic fibrosis Pancreatic fistula Pancreatic haemorrhage Pancreatic infarction Pancreatic mass Pancreatic necrosis Pancreatic phlegmon Pancreatic pseudoaneurysm Pancreatic pseudocyst Pancreatic steatosis
Pancreatic toxicity Pancreatitis Pancreatitis acute Pancreatitis chronic Pancreatitis haemorrhagic Pancreatitis necrotising Pancreatitis relapsing Pancreatolithiasis Papilla of Vater stenosis Paraesthesia oral Paresis anal sphincter Parotid duct obstruction Parotid gland enlargement Parotid gland haemorrhage Parotid lipomatosis Pelvic floor dyssynergia Peptic ulcer

Peptic ulcer haemorrhage Peptic ulcer perforation


1.0 Final 38 of 152 Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Rectal spasm

Gastrointestinal adverse events

Peptic ulcer perforation, obstructive Peptic ulcer, obstructive Perianal erythema Periodontal disease Periodontal inflammation Peripancreatic varices Peristalsis visible Peritoneal adhesions Peritoneal cloudy effluent Peritoneal cyst Peritoneal disorder Peritoneal fibrosis Peritoneal haematoma Peritoneal haemorrhage Peritoneal hernia Peritoneal lesion Peritoneal mesothelial hyperplasia Peritoneal necrosis Peritoneal perforation Peritoneocutaneous fistula Peritonitis lupus Pharyngo-oesophageal diverticulum Pigmentation lip Plicated tongue Pneumatosis intestinalis Pneumoperitoneum Pneumoretroperitoneum Poor dental condition Portal hypertensive colopathy Portal hypertensive enteropathy Portal hypertensive gastropathy Portal venous gas Post-tussive vomiting Pouchitis Prepyloric stenosis Presbyoesophagus Proctalgia Proctitis Proctitis haemorrhagic Proctitis ulcerative Proctoparalysis Protein-losing gastroenteropathy Protrusion tongue Pseudoachalasia Pseudodiverticular disease Pseudopolyposis Pudendal hernia Pyloric sphincter insufficiency Pylorospasm Pylorus dilatation Pyostomatitis vegetans Ranula Reactive gastropathy Rebound acid hypersecretion Rectal discharge Rectal fissure Rectal haemorrhage Rectal lesion Rectal obstruction Rectal perforation Rectal polyp Rectal prolapse


Final

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Rectal stenosis

Gastrointestinal adverse events

Rectal tenesmus Rectal ulcer Rectal ulcer haemorrhage Rectourethral fistula Reflux gastritis Regurgitation Retained deciduous tooth Retching Retroperitoneal effusion Retroperitoneal fibrosis Retroperitoneal haematoma Retroperitoneal haemorrhage Retroperitoneal hernia Retroperitoneal mass Retroperitoneal oedema Retroperitoneum cyst Richter's hernia Saliva altered Saliva discolouration Salivary duct inflammation Salivary duct obstruction Salivary duct stenosis Salivary gland atrophy Salivary gland calculus Salivary gland cyst Salivary gland disorder Salivary gland disorder Salivary gland enlargement Salivary gland fistula Salivary gland induration Salivary gland mass Salivary gland mucocoele Salivary gland pain Salivary hypersecretion Sandifer's syndrome Scalloped tongue Scaphoid abdomen Sciatic hernia Segmental diverticular colitis Sensitivity of teeth Short-bowel syndrome Sialadenosis Sialectasia Sialocele Sialodochitis fibrinosa Sialometaplasia Sideropenic dysphagia Small intestinal haemorrhage Small intestinal obstruction Small intestinal perforation Small intestinal stenosis Small intestinal ulcer haemorrhage Small intestinal ulcer perforation Small intestine polyp Small intestine ulcer Sordes Spigelian hernia Splenic artery aneurysm Splenic vein aneurysm Sprue-like enteropathy Stasis syndrome Steatorrĥoea

Stiff tongue


03 July 2019 1.0


Final

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Gastrointestinal adverse events

Stomach granuloma Stomach mass Stomatitis Stomatitis haemorrhagic Stomatitis necrotising Strangulated umbilical hernia Strawberry tongue Stress ulcer Subileus Submaxillary gland enlargement Superior mesenteric artery syndrome Supernumerary teeth Swollen tongue Teeth brittle Teething Thrombosis mesenteric vessel Tongue amyloidosis Tongue atrophy
Tongue blistering Tongue coated Tongue cyst Tongue discolouration Tongue discomfort Tongue disorder Tongue dry Tongue dysplasia Tongue eruption Tongue erythema Tongue exfoliation Tongue geographic Tongue haematoma Tongue haemorrhage Tongue infarction Tonque movement disturbance Tongue necrosis Tongue oedema Tongue pigmentation Tongue polyp Tongue pruritus Tongue spasm Tongue ulceration Tooth ankylosis Tooth delamination

Tooth demineralisation Tooth deposit Tooth development disorder Tooth discolouration

Tooth disorder Tooth erosion Tooth impacted

Tooth loss Tooth malformation

Tooth pulp haemorrhage Tooth resorption

Tooth socket haemorrhage

Toothache

Toxic dilatation of intestine Transient lingual papillitis Traumatic occlusion

Traumatic ulcerative granuloma with stromal eosinophilia

Trichoglossia

Truncus coeliacus thrombosis

Ulcerative duodenitis

MedDRA version 21.1


03 July 2019 1.0


Final

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Gastrointestinal adverse events

Ulcerative gastritis Ultrafiltration failure Umbilical hernia Umbilical hernia perforation Umbilical hernia, obstructive
Upper gastrointestinal haemorrhage Upper gastrointestinal perforation

Uraemic gastropathy Urinary ascites Uvulitis Varices oesophageal

Varicose veins of abdominal wall Varicose veins sublingual Vasculitis gastrointestinal Visceral venous thrombosis

Visceroptosis Volvulus

Volvulus of small bowel

Vomiting

Vomiting projectile White nipple sign Wischnewsky spots

Hepatic disorders

5'nucleotidase increased

Acquired antithrombin III deficiency Acquired hepatocerebral degeneration

Acquired protein S deficiency
Acute graft versus host disease in liver
Acute hepatic failure

Acute on chronic liver failure Acute yellow liver atrophy Alanine aminotransferase abnormal

Alanine aminotransferase increased

Allergic hepatitis Alloimmune hepatitis Ammonia abnormal Ammonia increased

Anorectal varices Anorectal varices haemorrhage Anti factor X activity abnormal Anti factor X activity decreased Anti factor X activity increased Antithrombin III decreased

Ascites

Aspartate aminotransferase abnormal Aspartate aminotransferase increased

Asterixis

Autoimmune hepatitis Bacterascites

Benign hepatic neoplasm Benign hepatobiliary neoplasm

Bile output abnormal Bile output decreased Biliary ascites Biliary cirrhosis Biliary fibrosis

Bilirubin conjugated abnormal Bilirubin conjugated increased Bilirubin excretion disorder

Bilirubin urine present Biopsy liver abnormal

Blood alkaline phosphatase abnormal Blood alkaline phosphatase increased

MedDRA version 21.1

Pre-defined MedDRA search


Preferred term


03 July 2019

1.0 Final 42 of 152

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Hepatic disorders Blood bilirubin abnormal Blood bilirubin increased Blood bilirubin unconjugated increased Blood cholinesterase abnormal Blood cholinesterase decreased Blood fibrinogen abnormal Blood fibrinogen decreased Blood thrombin abnormal Blood thrombin decreased Blood thromboplastin abnormal Blood thromboplastin decreased Bromosulphthalein test abnormal Child-Pugh-Turcotte score abnormal Child-Pugh-Turcotte score increased Cholaemia Cholangiosarcoma Cholestasis Cholestatic liver injury Cholestatic pruritus Chronic graft versus host disease in liver Chronic hepatic failure Chronic hepatitis Coagulation factor IX level abnormal Coagulation factor IX level decreased Coagulation factor V level abnormal Coagulation factor V level decreased Coagulation factor VII level abnormal Coagulation factor VII level decreased Coagulation factor X level abnormal Coagulation factor X level decreased Coagulation factor decreased Coma hepatic Computerised tomogram liver Computerised tomogram liver abnormal Cryptogenic cirrhosis Deficiency of bile secretion Diabetic hepatopathy

> Gastric variceal ligation Gastric varices

Gallbladder varices Gamma-glutamyltransferase abnormal Gamma-glutamyltransferase increased

Galactose elimination capacity test abnormal Galactose elimination capacity test decreased

Gastric variceal injection Gastric varices haemorrhage

Drug-induced liver injury Duodenal varices Focal nodular hyperplasia

Foetor hepaticus

Glutamate dehydrogenase increased Glycocholic acid increased Graft versus host disease in liver

Granulomatous liver disease Guanase increased

Haemorrhagic ascites Haemorrhagic hepatic cyst Hepaplastin abnormal

Haemangioma of liver

Hepaplastin decreased Hepatectomy

Hepatic adenoma Hepatic angiosarcoma


1.0 Final 43 of 152

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Hepatic disorders Hepatic artery flow decreased Hepatic atrophy Hepatic calcification Hepatic cancer Hepatic cancer metastatic Hepatic cancer recurrent Hepatic cancer stage I Hepatic cancer stage II Hepatic cancer stage III Hepatic cancer stage IV Hepatic cirrhosis Hepatic congestion Hepatic cyst Hepatic cyst ruptured Hepatic encephalopathy Hepatic encephalopathy prophylaxis Hepatic enzyme abnormal Hepatic enzyme decreased Hepatic enzyme increased Hepatic failure Hepatic fibrosis Hepatic fibrosis marker abnormal Hepatic fibrosis marker increased Hepatic function abnormal Hepatic haemangioma rupture Hepatic hamartoma Hepatic hydrothorax Hepatic hypertrophy Hepatic infiltration eosinophilic Hepatic lesion Hepatic lymphocytic infiltration Hepatic mass Hepatic necrosis Hepatic neoplasm Hepatic pain Hepatic sequestration Hepatic steato-fibrosis Hepatic steatosis Hepatic vascular resistance increased Hepatitis Hepatitis acute Hepatitis cholestatic Hepatitis chronic active Hepatitis chronic persistent Hepatitis fulminant Hepatitis toxic Hepatobiliary cancer Hepatobiliary cancer in situ Hepatobiliary cancer in Sitt Hepatobiliary cyst Hepatobiliary disease Hepatobiliary neoplasm Hepatobiliary scan abnormal Hepatoblastoma Hepatoblastoma recurrent Hepatocellular carcinoma Hepatocellular foamy cell syndrome Hepatocellular injury Hepatomegaly Hepatopulmonary syndrome Hepatorenal failure Hepatorenal syndrome Hepatosplenomegaly Hepatotoxicity


Date: Version: Status: 03 July 2019 A

Novo Nordisk

Status: Final 

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term
Hyperammonaemia

Periportal oedema

Hepatic disorders

Hyperbilirubinaemia Hypercholia Hyperfibrinolysis Hypertransaminasaemia Hypoalbuminaemia Hypocoagulable state Hypofibrinogenaemia Hypoprothrombinaemia Hypothrombinaemia Hypothromboplastinaemia Icterus index increased Immune-mediated hepatitis International normalised ratio abnormal International normalised ratio increased Intestinal varices Intestinal varices haemorrhage Intrahepatic portal hepatic venous fistula Ischaemic hepatitis Jaundice Jaundice cholestatic Jaundice hepatocellular Kayser-Fleischer ring Leucine aminopeptidase increased Liver ablation Liver and small intestine transplant Liver carcinoma ruptured Liver dialysis Liver disorder Liver function test abnormal Liver function test decreased Liver function test increased Liver induration Liver injury Liver iron concentration abnormal Liver iron concentration increased Liver operation Liver palpable Liver sarcoidosis Liver scan abnormal Liver tenderness Liver transplant Lupoid hepatic cirrhosis Lupus hepatitis Minimal hepatic encephalopathy Mitochondrial aspartate aminotransferase increased Mixed hepatocellular cholangiocarcinoma Mixed liver injury Model for end stage liver disease score abnormal Model for end stage liver disease score increased Molar ratio of total branched-chain amino acid to tyrosine Nodular regenerative hyperplasia Non-alcoholic fatty liver Non-alcoholic steatohepatitis Non-cirrhotic portal hypertension Nuclear magnetic resonance imaging liver abnormal Ocular icterus Oedema due to hepatic disease Oesophageal varices haemorrhage Parenteral nutrition associated liver disease Perihepatic discomfort Peripancreatic varices


Novo Nordisk

1.0

Final

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Peritoneal fluid protein abnormal Peritoneal fluid protein decreased Hepatic disorders Peritoneal fluid protein increased Peritoneovenous shunt Pneumobilia Portal fibrosis Portal hypertension Portal hypertensive colopathy Portal hypertensive enteropathy Portal hypertensive gastropathy Portal shunt Portal shunt procedure Portal tract inflammation Portal vein cavernous transformation Portal vein dilatation Portal vein flow decreased Portal vein pressure increased Portopulmonary hypertension Primary biliary cholangitis Protein C decreased Protein S abnormal Protein S decreased Prothrombin level abnormal Prothrombin level decreased Prothrombin time abnormal Prothrombin time prolonged Prothrombin time ratio abnormal Prothrombin time ratio increased Radiation hepatitis Regenerative siderotic hepatic nodule Renal and liver transplant Retinol binding protein decreased Retrograde portal vein flow Reye's syndrome Reynold's syndrome Small-for-size liver syndrome Spider naevus Splenic varices Splenic varices haemorrhage Splenorenal shunt Splenorenal shunt procedure Spontaneous intrahepatic portosystemic venous shunt Steatohepatitis Stomal varices Subacute hepatic failure Thrombin time abnormal Thrombin time prolonged Total bile acids increased Transaminases abnormal Transaminases increased Ultrasound liver abnormal Urine bilirubin increased Urobilinogen urine decreased Urobilinogen urine increased Varices oésophageal Varicose veins of abdominal wall White nipple sign X-ray hepatobiliary abnormal Yellow skin

> Acute motor axonal neuropathy Acute motor-sensory axonal neuropathy

Bickerstaff's encephalitis

Immune complex


Final 46 of 152

Novo Nordisk

```
Pre-defined MedDRA search
                                         Preferred term
                                          Chronic inflammatory demyelinating polyradiculoneuropathy
Immune complex
                                          Demyelinating polyneuropathy
                                          Guillain-Barre syndrome
                                          Miller Fisher syndrome
                                         Subacute inflammatory demyelinating polyneuropathy
Zika virus associated Guillain Barre syndrome
Injection site reactions
                                          Administration site abscess
                                          Administration site abscess sterile
                                          Administration site anaesthesia
                                          Administration site atrophy
                                          Administration site bruise
                                          Administration site calcification
                                          Administration site cellulitis
                                          Administration site coldness
                                          Administration site cyst
                                          Administration site dermatitis
                                          Administration site discharge
                                          Administration site discolouration
                                          Administration site discomfort
                                          Administration site dryness
                                          Administration site dysaesthesia
                                          Administration site eczema
                                          Administration site erosion
                                          Administration site erythema
                                          Administration site exfoliation
                                          Administration site extravasation
                                          Administration site fibrosis
                                          Administration site granuloma
                                          Administration site haematoma
                                          Administration site haemorrhage
                                          Administration site hyperaesthesia
                                          Administration site hypersensitivity
                                          Administration site hypertrichosis
                                          Administration site hypertrophy
                                          Administration site hypoaesthesia
                                          Administration site indentation
                                          Administration site induration
                                          Administration site infection
                                          Administration site inflammation
                                          Administration site injury
                                          Administration site irritation
                                          Administration site ischaemia
                                          Administration site joint discomfort
                                          Administration site joint effusion
                                          Administration site joint erythema
                                          Administration site joint infection
                                          Administration site
                                                              joint inflammation
                                          Administration site
                                                              joint movement impairment
                                          Administration site joint pain
                                          Administration site
                                                              joint warmth
                                          Administration site laceration
                                          Administration site lymphadenopathy
                                          Administration site macule
                                          Administration site mass
                                          Administration site movement impairment
                                          Administration site necrosis
                                          Administration site nerve damage
                                          Administration site nodule
                                          Administration site odour
                                          Administration site oedema
                                          Administration site pain
                                          Administration site pallor
```


 Date:
 03 July 2019

 Version:
 1.0

 Status:
 Final

Novo Nordisk

Status: Final 

```
Pre-defined MedDRA search
                                         Preferred term
Injection site reactions
                                         Administration site papule
                                         Administration site paraesthesia
                                         Administration site phlebitis
                                         Administration site photosensitivity reaction
                                         Administration site plaque
                                         Administration site pruritus
                                         Administration site pustule
                                         Administration site rash
                                         Administration site reaction
                                         Administration site recall reaction
                                         Administration site scab
                                         Administration site scar
                                         Administration site streaking
                                         Administration site swelling
                                         Administration site thrombosis
                                         Administration site ulcer
                                         Administration site urticaria
                                         Administration site vasculitis
                                         Administration site vesicles
                                         Administration site warmth
                                         Application site abscess
                                         Application site abscess sterile
                                         Application site acne
                                         Application site alopecia
                                         Application site anaesthesia
                                         Application site atrophy
                                         Application site bruise
                                         Application site burn
                                         Application site calcification
                                         Application site cellulitis
                                         Application site coldness
                                         Application site cvst
                                         Application site dermatitis
                                         Application site discharge
                                         Application site discolouration
                                         Application site discomfort
                                         Application site dryness
                                         Application site dysaesthesia
                                         Application site eczema
                                         Application site erosion
                                         Application site erythema
                                         Application site exfoliation
                                         Application site extravasation
                                         Application site fibrosis
                                         Application site fissure
                                         Application site folliculitis
                                         Application site granuloma
                                         Application site haematoma
                                         Application site haemorrhage
                                         Application site hyperaesthesia
                                         Application site hypersensitivity
                                         Application site hypertrichosis
Application site hypertrophy
                                         Application site hypoaesthesia
                                         Application site induration
                                         Application site
                                                           infection
                                         Application site inflammation
                                         Application site injury
                                         Application site irritation
                                         Application site ischaemia
                                         Application site joint discomfort
                                         Application site joint effusion
                                         Application site joint erythema
```


 Date:
 03 July 2019

 Version:
 1.0

 Status:
 Final

 Page:

Novo Nordisk

 ${\tt Pre-defined} \ {\tt MedDRA} \ {\tt search} \ {\tt -list} \ {\tt of} \ {\tt preferred} \ {\tt terms}$ 

Pre-defined MedDRA search Preferred term Injection site reactions Application site joint infection Application site joint inflammation Application site joint movement impairment Application site joint pain Application site joint swelling Application site joint warmth Application site laceration Application site lymphadenopathy Application site macule Application site mass Application site movement impairment Application site necrosis Application site nerve damage Application site nodule Application site odour Application site oedema Application site pain Application site pallor Application site papules Application site paraesthesia Application site perspiration Application site phlebitis Application site photosensitivity reaction Application site plaque Application site pruritus Application site purpura Application site pustules Application site rash Application site reaction Application site recall reaction Application site scab Application site scar Application site streaking Application site swelling Application site telangiectasia Application site thrombosis Application site ulcer Application site urticaria Application site vasculitis Application site vesicles Application site warmth Application site wound Embolia cutis medicamentosa Infusion site abscess Infusion site abscess sterile Infusion site anaesthesia Infusion site atrophy Infusion site bruising Infusion site calcification Infusion site cellulitis Infusion site coldness Infusion site cyst Infusion site dermatitis Infusion site discharge Infusion site discolouration Infusion site discomfort Infusion site dryness Infusion site dysaesthesia Infusion site eczema Infusion site erosion Infusion site erythema Infusion site exfoliation Infusion site extravasation


Novo Nordisk

1.0

Final

```
Pre-defined MedDRA search
                                          Preferred term
Injection site reactions
                                           Infusion site fibrosis
                                           Infusion site granuloma
                                           Infusion site haematoma
                                           Infusion site haemorrhage
                                           Infusion site hyperaesthesia
                                           Infusion site hypersensitivity
                                           Infusion site hypertrichosis
                                           Infusion site hypertrophy
                                           Infusion site hypoaesthesia
                                           Infusion site induration
                                           Infusion site infection
                                           Infusion site inflammation
                                           Infusion site injury
                                           Infusion site irritation
                                           Infusion site ischaemia
                                           Infusion site joint discomfort
                                           Infusion site joint effusion
                                           Infusion site joint erythema Infusion site joint infection
                                           Infusion site joint inflammation
                                           Infusion site joint movement impairment Infusion site joint pain
                                           Infusion site joint swelling
                                           Infusion site joint warmth Infusion site laceration
                                           Infusion site lymphadenopathy
                                           Infusion site macule
                                           Infusion site mass
                                           Infusion site mobility decreased
                                           Infusion site necrosis
                                           Infusion site nerve damage
                                           Infusion site nodule
                                           Infusion site oedema
                                           Infusion site pain
                                           Infusion site pallor
                                           Infusion site papule
                                           Infusion site paraesthesia
                                           Infusion site phlebitis
                                           Infusion site photosensitivity reaction
                                           Infusion site plaque
                                           Infusion site pruritus
                                           Infusion site pustule
                                           Infusion site rash
                                           Infusion site reaction
                                           Infusion site recall reaction
                                           Infusion site scab
                                           Infusion site scar
                                           Infusion site streaking
                                           Infusion site swelling
                                           Infusion site thrombosis
                                           Infusion site ulcer
                                           Infusion site urticaria
                                           Infusion site vasculitis
                                           Infusion site vesicles
                                           Infusion site warmth
                                           Injected limb mobility decreased
                                           Injection site abscess
                                           Injection site abscess sterile
                                           Injection site alopecia
                                           Injection site anaesthesia
                                           Injection site atrophy
                                           Injection site bruising
                                           Injection site calcification
```


Final 50 of 152

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Injection site reactions Injection site cellulitis Injection site coldness Injection site cyst Injection site deformation Injection site dermatitis Injection site discharge Injection site discolouration Injection site discomfort Injection site dryness Injection site dysaesthesia Injection site eczema Injection site erosion Injection site erythema Injection site exfoliation Injection site extravasation Injection site fibrosis Injection site granuloma Injection site haematoma Injection site haemorrhage Injection site hyperaesthesia Injection site hypersensitivity Injection site hypertrichosis Injection site hypertrophy Injection site hypoaesthesia Injection site indentation Injection site induration Injection site infection Injection site inflammation Injection site injury Injection site irritation Injection site ischaemia Injection site joint discomfort Injection site joint effusion Injection site joint erythema Injection site joint infection Injection site joint inflammation Injection site joint movement impairment Injection site joint pain Injection site joint swelling Injection site joint warmth Injection site laceration Injection site lymphadenopathy Injection site macule Injection site mass Injection site movement impairment Injection site necrosis Injection site nerve damage Injection site nodule Injection site oedema Injection site pain Injection site pallor Injection site papule
Injection site paraesthesia Injection site phlebitis Injection site photosensitivity reaction Injection site plaque Injection site pruritus Injection site pustule Injection site rash Injection site reaction Injection site recall reaction Injection site scab Injection site scar


Final

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Injection site reactions Injection site streaking Injection site swelling Injection site telangiectasia Injection site thrombosis Injection site ulcer Injection site urticaria Injection site vasculitis Injection site vesicles Injection site warmth Instillation site abscess Instillation site anaesthesia Instillation site atrophy Instillation site bruise Instillation site burn Instillation site coldness Instillation site complication Instillation site discharge Instillation site discolouration Instillation site discomfort Instillation site dryness Instillation site erosion Instillation site erythema Instillation site exfoliation Instillation site foreign body sensation Instillation site haematoma Instillation site haemorrhage Instillation site hyperaesthesia Instillation site hypersensitivity Instillation site hypoaesthesia Instillation site induration Instillation site infection Instillation site inflammation Instillation site irritation Instillation site lacrimation Instillation site necrosis Instillation site nodule Instillation site odour Instillation site oedema Instillation site pain Instillation site papules Instillation site paraesthesia Instillation site pruritus Instillation site pustules Instillation site rash Instillation site reaction Instillation site scab Instillation site swelling Instillation site thrombosis Instillation site ulcer Instillation site urticaria Instillation site vesicles Instillation site warmth Malabsorption from administration site Malabsorption from application site
Malabsorption from injection site Oral administration complication Puncture site abscess Puncture site discharge Puncture site erythema Puncture site haemorrhage Puncture site hernia Puncture site hypoaesthesia

Puncture site induration


Date: Version: Status:

Page:

03 July 2019 Novo Nordisk

1.0

Final


Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Injection site reactions Puncture site infection Puncture site oedema Puncture site pain Puncture site reaction Puncture site swelling Systemic leakage Vessel puncture site anaesthesia Vessel puncture site bruise Vessel puncture site cellulitis Vessel puncture site discharge Vessel puncture site erythema Vessel puncture site haematoma Vessel puncture site haemorrhage Vessel puncture site hypoaesthesia Vessel puncture site induration Vessel puncture site infection Vessel puncture site inflammation Vessel puncture site occlusion Vessel puncture site pain Vessel puncture site paraesthesia Vessel puncture site phlebitis Vessel puncture site pruritus Vessel puncture site rash Vessel puncture site reaction Vessel puncture site swelling Vessel puncture site thrombosis Vessel puncture site vesicles Malignant neoplasms 5q minus syndrome Abdominal wall neoplasm malignant Acinar cell carcinoma of pancreas Acinic cell carcinoma of salivary gland Acral lentiginous melanoma Acral lentiginous melanoma stage I Acral lentiginous melanoma stage II Acral lentiginous melanoma stage III Acral lentiginous melanoma stage IV Acute bilineal leukaemia Acute biphenotypic leukaemia Acute leukaemia Acute leukaemia in remission Acute lymphocytic leukaemia Acute lymphocytic leukaemia (in remission) Acute lymphocytic leukaemia recurrent Acute lymphocytic leukaemia refractory Acute megakaryocytic leukaemia Acute megakaryocytic leukaemia (in remission) Acute monocytic leukaemia Acute monocytic leukaemia (in remission) Acute myeloid leukaemia Acute myeloid leukaemia (in remission) Acute myeloid leukaemia recurrent Acute myeloid leukaemia refractory Acute myelomonocytic leukaemia Acute promyelocytic leukaemia Acute undifferentiated leukaemia Adenocarcinoma Adenocarcinoma gastric Adenocarcinoma of appendix Adenocarcinoma of colon Adenocarcinoma of salivary gland Adenocarcinoma of the cervix Adenocarcinoma pancreas


 Date:
 03 July 2019

 Version:
 1.0

 Status:
 Final

 Page:

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Malignant neoplasms

Adenoid cystic carcinoma
Adenoid cystic carcinoma of external auditory canal
Adenoid cystic carcinoma of salivary gland
Adenosquamous carcinoma of the cervix
Adenosquamous carcinoma of vagina
Adenosquamous cell carcinoma
Adenosquamous cell lung cancer
Adenosquamous cell lung cancer recurrent
Adenosquamous cell lung cancer stage 0

Adenosquamous cell lung cancer recurrent Adenosquamous cell lung cancer stage 0 Adenosquamous cell lung cancer stage I Adenosquamous cell lung cancer stage II Adenosquamous cell lung cancer stage III Adenosquamous cell lung cancer stage IV Adrenal gland cancer
Adrenal gland cancer metastatic Adrenocortical carcinoma Adult T-cell lymphoma leukaemia Adult T-cell lymphoma leukaemia recurrent Adult T-cell lymphoma leukaemia refractory Adult T-cell lymphoma leukaemia stage I Adult T-cell lymphoma leukaemia stage II Adult T-cell lymphoma

leukaemia stage I
Adult T-cell lymphoma
leukaemia stage II
Adult T-cell lymphoma
leukaemia stage III
Adult T-cell lymphoma
leukaemia stage IV
Aesthesioneuroblastoma
Aleukaemic leukaemia
Alveolar rhabdomyosarcoma
Alveolar soft part sarcoma
Alveolar soft part sarcoma
Alveolar soft part sarcoma recurrent
Anal cancer
Anal cancer metastatic
Anal cancer recurrent
Anal cancer stage I
Anal cancer stage II
Anal cancer stage III
Anal cancer stage IV

Anal squamous cell carcinoma
Anaplastic astrocytoma
Anaplastic large cell lymphoma T- and null-cell types
Anaplastic large cell lymphoma T- and null-cell types
recurrent
Anaplastic large cell lymphoma T- and null-cell types

refractory
Anaplastic large cell lymphoma T- and null-cell types stage
I
Anaplastic large cell lymphoma T- and null-cell types stage
I
Anaplastic large cell lymphoma T- and null-cell types stage

Anaplastic large cell lymphoma T- and null-cell types stage III
Anaplastic large cell lymphoma T- and null-cell types stage

Anaplastic large-cell lymphoma Anaplastic meningioma Anaplastic oligodendroglioma

Anaplastic thyroid cancer


Final 54 of 152

 ${\tt Pre-defined} \ {\tt MedDRA} \ {\tt search} \ {\tt -list} \ {\tt of} \ {\tt preferred} \ {\tt terms}$ 

Pre-defined MedDRA search Preferred term Malignant neoplasms Angiocentric glioma Angiocentric lymphoma Angiocentric lymphoma recurrent Angiocentric lymphoma refractory Angiocentric lymphoma stage I Angiocentric lymphoma stage II Angiocentric lymphoma stage III Angiocentric lymphoma stage IV Angioimmunoblastic T-cell lymphoma Angioimmunoblastic T-cell lymphoma recurrent Angioimmunoblastic T-cell lymphoma refractory Angioimmunoblastic T-cell lymphoma stage I Angioimmunoblastic T-cell lymphoma stage II Angioimmunoblastic T-cell lymphoma stage III Angioimmunoblastic T-cell lymphoma stage IV Angiosarcoma Angiosarcoma metastatic Angiosarcoma non-metastatic Angiosarcoma recurrent Apocrine breast carcinoma Appendix cancer Astrocytoma Astrocytoma malignant Atypical teratoid rhabdoid tumour of CNS B precursor type acute leukaemia B-cell lymphoma B-cell lymphoma recurrent B-cell lymphoma refractory B-cell lymphoma stage I B-cell lymphoma stage II B-cell lymphoma stage III B-cell lymphoma stage IV B-cell prolymphocytic leukaemia B-cell small lymphocytic lymphoma B-cell small lymphocytic lymphoma recurrent B-cell small lymphocytic lymphoma refractory B-cell small lymphocytic lymphoma stage I B-cell small lymphocytic lymphoma stage II B-cell small lymphocytic lymphoma stage III B-cell small lymphocytic lymphoma stage IV B-cell type acute leukaemia B-cell unclassifiable lymphoma high grade B-cell unclassifiable lymphoma low grade Basal cell carcinoma Basosquamous carcinoma Basosquamous carcinoma of skin Bile duct adenocarcinoma Bile duct adenosquamous carcinoma Bile duct cancer Bile duct cancer recurrent Bile duct cancer stage 0 Bile duct cancer stage I Bile duct cancer stage II Bile duct cancer stage III Bile duct cancer stage IV Bile duct squamous cell carcinoma Biliary cancer metastatic Biphasic mesothelioma Bladder adenocarcinoma recurrent Bladder adenocarcinoma stage 0 Bladder adenocarcinoma stage

Bladder adenocarcinoma stage II


 Date:
 03 July 2019

 Version:
 1.0

 Status:
 Final

 Page:

Novo Nordisk

```
Pre-defined MedDRA search
                                           Preferred term
                                           Bladder adenocarcinoma stage III
Malignant neoplasms
                                           Bladder adenocarcinoma stage IV
                                           Bladder adenocarcinoma stage unspecified
                                           Bladder cancer
                                           Bladder cancer recurrent
                                           Bladder cancer stage 0, with cancer in situ
Bladder cancer stage 0, without cancer in situ
                                           Bladder cancer stage I, with cancer in situ
                                           Bladder cancer stage I, without cancer in situ
Bladder cancer stage II
                                           Bladder cancer stage III
                                           Bladder cancer stage IV
                                           Bladder squamous cell carcinoma recurrent
                                           Bladder squamous cell carcinoma stage 0
                                           Bladder squamous cell carcinoma stage
                                           Bladder squamous cell carcinoma stage II
                                           Bladder squamous cell carcinoma stage III
                                           Bladder squamous cell carcinoma stage IV Bladder squamous cell carcinoma stage unspecified
                                           Bladder transitional cell carcinoma
                                           Bladder transitional cell carcinoma metastatic
                                           Bladder transitional cell carcinoma recurrent
                                           Bladder transitional cell carcinoma stage 0
                                           Bladder transitional cell carcinoma stage I
                                           Bladder transitional cell carcinoma stage II
                                           Bladder transitional cell carcinoma stage III
                                           Bladder transitional cell carcinoma stage IV
                                           Blast cell crisis
                                           Blast crisis in myelogenous leukaemia
                                           Blastic plasmacytoid dendritic cell neoplasia
                                           Bone cancer
                                           Bone cancer metastatic
                                           Bone giant cell tumour malignant
                                           Bone marrow leukaemic cell infiltration
                                           Bone marrow tumour cell infiltration
                                           Bone sarcoma
                                           Bowen's disease
                                           Brain cancer metastatic
                                           Brain neoplasm malignant
                                           Brain sarcoma
                                           Brain stem glioma
                                           Breast angiosarcoma
                                           Breast angiosarcoma metastatic
                                           Breast cancer
                                           Breast cancer female
                                           Breast cancer in situ
                                           Breast cancer male
                                           Breast cancer metastatic
                                           Breast cancer recurrent
                                           Breast cancer stage I
                                           Breast cancer stage II
                                           Breast cancer stage III
Breast cancer stage IV
                                           Breast sarcoma
                                           Breast sarcoma metastatic
                                           Breast sarcoma recurrent
                                           Bronchial carcinoma
                                           Bronchioloalveolar carcinoma
                                           Burkitt's leukaemia
                                           Burkitt's lymphoma
                                           Burkitt's lymphoma recurrent
                                           Burkitt's lymphoma refractory
                                           Burkitt's lymphoma stage I
```


 Date:
 03 July 2019

 Version:
 1.0

 Status:
 Final

 Page:

uly 2019 Novo Nordisk
1.0
Final

```
Pre-defined MedDRA search
                                             Preferred term
Malignant neoplasms
                                             Burkitt's lymphoma stage II
                                             Burkitt's lymphoma stage III
                                             Burkitt's lymphoma stage IV
                                             Buschke-Lowenstein's tumour
                                             CNS germinoma
                                             Cancer in remission
                                             Carcinoid tumour
                                             Carcinoid tumour of the appendix
                                             Carcinoid tumour of the caecum
                                             Carcinoid tumour of the duodenum
                                             Carcinoid tumour of the gastrointestinal tract
                                             Carcinoid tumour of the liver
                                             Carcinoid tumour of the ovary
                                             Carcinoid tumour of the pancreas
                                             Carcinoid tumour of the prostate
                                             Carcinoid tumour of the small bowel
                                             Carcinoid tumour of the stomach
                                             Carcinoid tumour pulmonary
                                             Carcinoma ex-pleomorphic adenoma Carcinoma in situ
                                             Carcinoma in situ of eye
                                             Carcinoma in situ of penis
                                             Carcinoma in situ of skin
                                             Carcinoma in situ of trachea
                                             Cardiac neoplasm malignant
                                             Central nervous system leukaemia
Central nervous system lymphoma
                                             Central nervous system melanoma
                                             Central nervous system neuroblastoma
                                             Cervix cancer metastatic
                                             Cervix carcinoma
                                             Cervix carcinoma recurrent
                                             Cervix carcinoma stage 0
                                             Cervix carcinoma stage I
                                             Cervix carcinoma stage II
                                             Cervix carcinoma stage III
                                             Cervix carcinoma stage IV
                                             Chloroma
                                             Chloroma (in remission)
                                             Cholangiocarcinoma
                                             Cholangiosarcoma
                                             Chondrosarcoma
                                             Chondrosarcoma metastatic
                                             Chondrosarcoma recurrent
                                             Chordoma
                                             Choriocarcinoma
                                             Choroid melanoma
                                             Choroid plexus carcinoma
                                             Chromophobe renal cell carcinoma
Chronic eosinophilic leukaemia
                                             Chronic leukaemia
                                             Chronic leukaemia in remission
Chronic lymphocytic leukaemia
                                             Chronic lymphocytic leukaemia (in remission)
                                             Chronic lymphocytic leukaemia recurrent
                                             Chronic lymphocytic leukaemia refractory
                                             Chronic lymphocytic leukaemia stage 0
                                             Chronic lymphocytic leukaemia stage 1
Chronic lymphocytic leukaemia stage 2
Chronic lymphocytic leukaemia stage 3
                                             Chronic lymphocytic leukaemia stage
                                             Chronic lymphocytic leukaemia transformation
                                             Chronic myeloid leukaemia
```


Final  Novo Nordisk

1.0

Pre-defined MedDRA search - list of preferred terms

```
Pre-defined MedDRA search
                                            Preferred term
                                             Chronic myeloid leukaemia (in remission)
Malignant neoplasms
                                             Chronic myeloid leukaemia recurrent
                                             Chronic myeloid leukaemia transformation
                                             Chronic myelomonocytic leukaemia
Chronic myelomonocytic leukaemia (in remission)
                                             Ciliary body melanoma
Clear cell carcinoma of cervix
                                             Clear cell endometrial carcinoma
                                             Clear cell renal cell carcinoma
                                             Clear cell sarcoma of soft tissue
                                             Clear cell sarcoma of the kidney
                                             Colon cancer
                                             Colon cancer metastatic
                                             Colon cancer recurrent
                                             Colon cancer stage 0
                                             Colon cancer stage I
                                             Colon cancer stage II
                                             Colon cancer stage III
                                             Colon cancer stage IV
                                             Colorectal adenocarcinoma
                                             Colorectal cancer
                                             Colorectal cancer metastatic
                                             Colorectal cancer recurrent
                                             Colorectal cancer stage I
                                             Colorectal cancer stage II
                                             Colorectal cancer stage III
Colorectal cancer stage IV
                                             Colorectal carcinoma stage 0
                                             Composite lymphoma
Congenital fibrosarcoma
                                             Congenital malignant neoplasm
Congenital retinoblastoma
                                             Conjunctival melanoma
                                             Cutaneous lymphoma
                                             Cystadenocarcinoma ovary
                                             Cystadenocarcinoma pancreas
                                             Dedifferentiated liposarcoma
                                             Dermatofibrosarcoma protuberans
                                             Dermatofibrosarcoma protuberans metastatic
                                             Desmoplastic melanoma
                                             Desmoplastic mesothelioma
                                             Desmoplastic small round cell tumour
                                             Diffuse large B-cell lymphoma
                                             Diffuse large B-cell lymphoma recurrent
                                             Diffuse large B-cell lymphoma refractory
                                             Diffuse large B-cell lymphoma stage I
                                             Diffuse large B-cell lymphoma stage II
                                             Diffuse large B-cell lymphoma stage III
                                             Diffuse large B-cell lymphoma stage IV
                                             Disseminated large cell lymphoma
                                             Double hit lymphoma
                                             Ductal adenocarcinoma of pancreas
Ear neoplasm malignant
                                             Eccrine carcinoma
Embryonal rhabdomyosarcoma
                                             Endocrine neoplasm malignant
                                             Endometrial adenocarcinoma
                                             Endometrial cancer
                                             Endometrial cancer metastatic
                                             Endometrial cancer recurrent
                                             Endometrial cancer stage 0
                                             Endometrial cancer stage I
```

Endometrial cancer stage II


Final 58 of 152

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Malignant neoplasms Endometrial cancer stage III Endometrial cancer stage IV Endometrial sarcoma Endometrial sarcoma metastatic Endometrial sarcoma recurrent Endometrial stromal sarcoma Endotheliomatosis Enteropathy-associated T-cell lymphoma Eosinophilic leukaemia Ependymoma malignant Epididymal cancer Epiglottic carcinoma Epithelioid mesothelioma Epithelioid sarcoma Epithelioid sarcoma metastatic Epithelioid sarcoma recurrent Epstein-Barr virus associated lymphoma Erythraemic myelosis (in remission) Erythroleukaemia Ewing's sarcoma Ewing's sarcoma metastatic Ewing's sarcoma recurrent Ewing-like sarcoma Extra-osseous Ewing's sarcoma Extra-osseous Ewing's sarcoma metastatic Extra-osseous Ewing's sarcoma recurrent Extra-osseous Ewing's sarcoma recurrent
Extragonadal primary embryonal carcinoma
Extragonadal primary germ cell tumour
Extragonadal primary germ cell tumour mixed
Extragonadal primary germ cell tumour mixed stage I
Extragonadal primary germ cell tumour mixed stage II
Extragonadal primary germ cell tumour mixed stage II
Extragonadal primary malignant teratoma
Extragonadal primary non-seminoma
Extragonadal primary non-seminoma Extragonadal primary non-seminoma stage I Extragonadal primary non-seminoma stage II Extragonadal primary non-seminoma stage III Extragonadal primary non-seminoma stage IV
Extragonadal primary seminoma (pure)
Extragonadal primary seminoma (pure) stage I
Extragonadal primary seminoma (pure) stage I
Extragonadal primary seminoma (pure) stage II Extragonadal primary seminoma (pure) stage III Extragonadal primary seminoma (pure) stage IV Extramammary Paget's disease Extranodal marginal zone B-cell lymphoma (BALT type) Extranodal marginal zone B-cell lymphoma (MALT type) Extranodal marginal zone B-cell lymphoma (MALT type) recurrent Extranodal marginal zone B-cell lymphoma (MALT type) refractory Extranodal marginal zone B-cell lymphoma (MALT type) stage I Extranodal marginal zone B-cell lymphoma (MALT type) stage Extranodal marginal zone B-cell lymphoma (MALT type) stage Extranodal marginal zone B-cell lymphoma (MALT type) stage T 7.7 Extraocular retinoblastoma Extraskeletal chondrosarcoma metastatic Extraskeletal chondrosarcoma recurrent Extraskeletal myxoid chondrosarcoma Extraskeletal osteosarcoma

Extraskeletal osteosarcoma metastatic


 Date:
 03 July 2019

 Version:
 1.0

 Status:
 Final

 Page:

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Malignant neoplasms Extraskeletal osteosarcoma recurrent Fallopian tube cancer Fallopian tube cancer metastatic Fallopian tube cancer stage I Fallopian tube cancer stage II Fallopian tube cancer stage III Fallopian tube cancer stage IV Familial medullary thyroid cancer Female reproductive tract carcinoma in situ Fibrosarcoma Fibrosarcoma metastatic Follicle centre lymphoma diffuse small cell lymphoma Follicle centre lymphoma diffuse small cell lymphoma recurrent Follicle centre lymphoma diffuse small cell lymphoma refractory Follicle centre lymphoma diffuse small cell lymphoma stage I Follicle centre lymphoma diffuse small cell lymphoma stage Follicle centre lymphoma diffuse small cell lymphoma stage Follicle centre lymphoma diffuse small cell lymphoma stage Follicle centre lymphoma, follicular grade I, II, III Follicle centre lymphoma, follicular grade I, II, III recurrent Follicle centre lymphoma, follicular grade I, II, III refractory Follicle centre lymphoma, follicular grade I, II, III stage Follicle centre lymphoma, follicular grade I, II, III stage Follicle centre lymphoma, follicular grade I, II, III stage Follicle centre lymphoma, follicular grade I, II, III stage ΙV Follicular dendritic cell sarcoma Follicular thyroid cancer Gallbladder adenocarcinoma Gallbladder adenosquamous carcinoma Gallbladder cancer Gallbladder cancer metastatic Gallbladder cancer recurrent Gallbladder cancer stage 0 Gallbladder cancer stage I Gallbladder cancer stage II Gallbladder cancer stage III Gallbladder cancer stage IV Gallbladder squamous cell carcinoma Ganglioglioma Ganglioneuroblastoma Gastric cancer Gastric cancer recurrent Gastric cancer stage 0 Gastric cancer stage Gastric cancer stage II Gastric cancer stage III Gastric cancer stage IV Gastric sarcoma Gastrinoma malignant Gastroenteropancreatic neuroendocrine tumour disease Gastrointestinal adenocarcinoma

Gastrointestinal cancer metastatic


Date: Version: Status: Page: 03 July 2019 1.0 Final

Final 60 of 152

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Gastrointestinal carcinoma

Malignant neoplasms

Gastrointestinal carcinoma in situ Gastrointestinal lymphoma Gastrointestinal melanoma Gastrointestinal stromal cancer Gastrooesophageal cancer Gastrooesophageal cancer recurrent Genital cancer male Genital cancer male in situ Genital neoplasm malignant female Genitourinary melanoma Germ cell cancer Germ cell cancer metastatic Gestational trophoblastic tumour Gingival cancer Glioblastoma Glioblastoma multiforme Glioma Gliomatosis cerebri Glioneuronal tumour Gliosarcoma Glottis carcinoma Glucagonoma HER-2 positive breast cancer HER-2 positive gastric cancer Haemangiopericytoma Haemangiopericytoma of meninges Haematological malignancy Hairy cell leukaemia
Hairy cell leukaemia recurrent Head and neck cancer Head and neck cancer metastatic Head and neck cancer stage I Head and neck cancer stage II Head and neck cancer stage III Head and neck cancer stage IV Hepatic angiosarcoma Hepatic cancer Hepatic cancer metastatic Hepatic cancer recurrent Hepatic cancer stage I Hepatic cancer stage II Hepatic cancer stage III Hepatic cancer stage IV Hepatobiliary cancer Hepatobiliary cancer in situ Hepatoblastoma Hepatoblastoma recurrent Hepatocellular carcinoma Hepatosplenic T-cell lymphoma Hereditary leiomyomatosis renal cell carcinoma Hereditary papillary renal carcinoma Hidradenocarcinoma High grade B-cell lymphoma Burkitt-like lymphoma High grade B-cell lymphoma Burkitt-like lymphoma lymphoma recurrent High grade B-cell lymphoma Burkitt-like lymphoma refractory High grade B-cell lymphoma Burkitt-like lymphoma stage I High grade B-cell lymphoma Burkitt-like lymphoma stage II High grade B-cell lymphoma Burkitt-like lymphoma stage III High grade B-cell lymphoma Burkitt-like lymphoma stage IV High-grade B-cell lymphoma Histiocytic medullary reticulosis Histiocytic sarcoma


03 July 2019 1.0 Final 61 of 152

Novo Nordisk

```
Pre-defined MedDRA search
                                                Preferred term
Malignant neoplasms
                                                Hodgkin's disease
                                                Hodgkin's disease lymphocyte depletion stage I site
                                                unspecified
                                                Hodgkin's disease lymphocyte depletion stage I subdiaphragm Hodgkin's disease lymphocyte depletion stage I
                                                supradiaphragm
                                                Hodgkin's disease lymphocyte depletion stage II site
                                                unspecified
                                                Hodgkin's disease lymphocyte depletion stage II subdiaphragm
                                                Hodgkin's disease lymphocyte depletion stage II
                                                supradiaphragm
                                                Hodgkin's disease lymphocyte depletion type recurrent
                                                Hodgkin's disease lymphocyte depletion type refractory
                                                Hodgkin's disease lymphocyte depletion type stage III
                                                Hodgkin's disease lymphocyte depletion type stage IV
                                                Hodgkin's disease lymphocyte depletion type stage
                                                unspecified
                                                Hodgkin's disease lymphocyte predominance stage I site
                                                unspec
                                                Hodgkin's disease lymphocyte predominance stage I
                                                subdiaphragm
                                                Hodgkin's disease lymphocyte predominance stage I
                                                supradiaphragm
                                                Hodgkin's disease lymphocyte predominance stage II site
                                                unspec
                                                Hodgkin's disease lymphocyte predominance stage II
                                                subdiaphragm
                                                Hodgkin's disease lymphocyte predominance stage II
                                                supradiaphragm
                                                Hodgkin's disease lymphocyte predominance type recurrent Hodgkin's disease lymphocyte predominance type refractory Hodgkin's disease lymphocyte predominance type stage III
                                                Hodgkin's disease lymphocyte predominance type stage IV Hodgkin's disease lymphocyte predominance type stage
                                                unspecified
                                                Hodgkin's disease mixed cellularity recurrent
                                                Hodgkin's disease mixed cellularity refractory
                                                Hodgkin's disease mixed cellularity stage I site unspecified Hodgkin's disease mixed cellularity stage I subdiaphragmatic Hodgkin's disease mixed cellularity stage I
                                                supradiaphragmatic
                                                Hodgkin's disease mixed cellularity stage II
                                                subdiaphragmatic
                                                Hodgkin's disease mixed cellularity stage II
                                                supradiaphragmatic
                                                Hodgkin's disease mixed cellularity stage III
                                                Hodgkin's disease mixed cellularity stage IV
                                                Hodgkin's disease mixed cellularity stage unspecified
                                                Hodgkin's disease nodular sclerosis
Hodgkin's disease nodular sclerosis recurrent
                                                Hodgkin's disease nodular sclerosis refractory
                                                Hodgkin's disease nodular sclerosis stage I
Hodgkin's disease nodular sclerosis stage II
                                                Hodgkin's disease nodular sclerosis stage III
                                                Hodgkin's disease nodular sclerosis stage IV
                                                Hodgkin's disease recurrent
                                                Hodgkin's disease refractory
                                                Hodgkin's disease stage I
                                                Hodgkin's disease stage II
                                                Hodgkin's disease stage III
                                                Hodgkin's disease stage IV
                                                Hodgkin's disease unclassifiable
                                                Hormone refractory breast cancer
```


Novo Nordisk

1.0

Final

```
Pre-defined MedDRA search
                                                    Preferred term
Malignant neoplasms
                                                    Hormone-dependent prostate cancer
                                                    Hormone-refractory prostate cancer Huerthle cell carcinoma
                                                    Hypopharyngeal cancer Hypopharyngeal cancer recurrent
                                                    Hypopharyngeal cancer stage 0
                                                    Hypopharyngeal cancer stage I
                                                    Hypopharyngeal cancer stage II
                                                    Hypopharyngeal cancer stage III
                                                    Hypopharyngeal cancer stage IV
                                                    Immune reconstitution inflammatory syndrome associated Kaposi's sarcoma Immunoblastic lymphoma
                                                    Inflammatory carcinoma of breast recurrent
                                                    Inflammatory carcinoma of breast stage III
                                                    Inflammatory carcinoma of breast stage IV
                                                    {\tt Inflammator}\bar{{\tt y}} \ {\tt carcinoma} \ {\tt of} \ {\tt the} \ {\tt breast}
                                                    Inflammatory malignant fibrous histiocytoma Inflammatory myofibroblastic tumour Intestinal T-cell lymphoma recurrent
                                                    Intestinal T-cell lymphoma refractory Intestinal T-cell lymphoma stage I
                                                    Intestinal T-cell lymphoma stage II
                                                    Intestinal T-cell lymphoma stage III
Intestinal T-cell lymphoma stage IV
                                                    Intestinal adenocarcinoma
Intestinal metastasis
                                                    Intracranial germ cell tumour
Intracranial meningioma malignant
                                                    Intraductal papillary breast neoplasm
                                                    Intraductal papillary-mucinous carcinoma of pancreas Intraductal proliferative breast lesion
                                                    Intraocular melanoma
                                                    Invasive breast carcinoma
                                                    Invasive ductal breast carcinoma
                                                    Invasive lobular breast carcinoma
                                                    Invasive papillary breast carcinoma
                                                    Iris melanoma
                                                    Juvenile chronic myelomonocytic leukaemia
                                                    Kaposi's sarcoma
                                                    Kaposi's sarcoma AIDS related
                                                    Kaposi's sarcoma classical type
                                                    Keratinising squamous cell carcinoma of nasopharynx
                                                    Keratoacanthoma
                                                    Langerhans cell sarcoma
Large cell lung cancer
                                                    Large cell lung cancer metastatic
                                                    Large cell lung cancer recurrent
                                                    Large cell lung cancer stage 0
Large cell lung cancer stage I
                                                    Large cell lung cancer stage II
                                                    Large cell lung cancer stage III
Large cell lung cancer stage IV
                                                    Laryngeal cancer
                                                    Laryngeal cancer metastatic
                                                    Laryngeal cancer recurrent
                                                    Laryngeal cancer stage 0
                                                    Laryngeal cancer stage I
                                                    Laryngeal cancer stage II
                                                    Larvngeal cancer stage III
                                                    Laryngeal cancer stage IV
                                                    Laryngeal squamous cell carcinoma
                                                    Leiomyosarcoma
```


Date: Version: Status: Page: 03 July 2019 | **Novo Nordisk**1.0 | Final |


Pre-defined MedDRA search - list of preferred terms

 ${\tt Pre-defined \ MedDRA \ search}$ 

Preferred term

Malignant neoplasms

```
Leiomyosarcoma metastatic
Leiomyosarcoma recurrent
Lentigo maligna
Lentigo maligna recurrent
Lentigo maligna stage I
Lentigo maligna stage II
Lentigo maligna stage III
Lentigo maligna stage IV
Leptomeningeal myelomatosis
Leukaemia
Leukaemia basophilic
Leukaemia cutis
Leukaemia granulocytic
Leukaemia in remission
Leukaemia monocytic
Leukaemia recurrent
Leukaemic cardiac infiltration
Leukaemic infiltration
Leukaemic infiltration extramedullary
Leukaemic infiltration gingiva
Leukaemic infiltration hepatic
Leukaemic infiltration ovary
Leukaemic infiltration pulmonary
Leukaemic infiltration renal
Leukaemic lymphoma
Leukaemic retinopathy
Leydig cell tumour of the testis
Linitis plastica
Lip and
or oral cavity cancer
Lip and or oral cavity cancer recurrent
Lip and
or oral cavity cancer stage 0
Lip and
or oral cavity cancer stage I
Lip and
or oral cavity cancer stage II
Lip and
or oral cavity cancer stage III
Lip and
or oral cavity cancer stage IV
Lip neoplasm malignant stage unspecified
Lip squamous cell carcinoma
Liposarcoma
Liposarcoma metastatic
Liposarcoma recurrent
Lobular breast carcinoma in situ
Lung adenocarcinoma
Lung adenocarcinoma recurrent
Lung adenocarcinoma stage 0
Lung adenocarcinoma stage I
Lung adenocarcinoma stage II
Lung adenocarcinoma stage III
Lung adenocarcinoma stage IV
Lung cancer metastatic
Lung carcinoma cell type unspecified recurrent
Lung carcinoma cell type unspecified stage O
Lung carcinoma cell type unspecified stage I
Lung carcinoma cell type unspecified stage II
Lung carcinoma cell type unspecified stage III
Lung carcinoma cell type unspecified stage IV
Lung infiltration malignant
```


Date: Version: Status: Page: 03 July 2019 1.0 Final 64 of 152

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Malignant neoplasms Lung neoplasm malignant Lung squamous cell carcinoma metastatic Lung squamous cell carcinoma recurrent Lung squamous cell carcinoma stage 0 Lung squamous cell carcinoma stage Lung squamous cell carcinoma stage II Lung squamous cell carcinoma stage III Lung squamous cell carcinoma stage IV Lymphangiosarcoma Lymphangiosis carcinomatosa Lymphocytic leukaemia Lymphocytic lymphoma Lymphoid leukaemia (in remission) Lymphoma Lymphoma AIDS related Lymphoma transformation Lymphoplasmacytoid lymphoma immunocytoma Lymphoplasmacytoid lymphoma immunocytoma recurrent Lymphoplasmacytoid lymphoma immunocytoma refractory Lymphoplasmacytoid lymphoma immunocytoma stage I Lymphoplasmacytoid lymphoma immunocytoma stage II Lymphoplasmacytoid lymphoma immunocytoma stage III Lymphoplasmacytoid lymphoma immunocytoma stage IV Malignant anorectal neoplasm Malignant blue naevus Malignant connective tissue neoplasm Malignant cranial nerve neoplasm Malignant fibrous histiocytoma Malignant fibrous histiocytoma metastatic Malignant fibrous histiocytoma of bone Malignant fibrous histiocytoma recurrent Malignant genitourinary tract neoplasm Malignant giant cell fibrous histiocytoma Malignant glioma Malignant haemangiopericytoma Malignant haemangiopericytoma metastatic Malignant haemangiopericytoma recurrent Malignant histiocytosis
Malignant hydatidiform mole Malignant joint neoplasm Malignant lymphoid neoplasm Malignant lymphoma unclassifiable high grade Malignant lymphoma unclassifiable low grade Malignant mast cell neoplasm Malignant mediastinal neoplasm Malignant melanoma Malignant melanoma in situ Malignant melanoma of eyelid Malignant melanoma of sites other than skin Malignant melanoma stage I Malignant melanoma stage II Malignant melanoma stage III Malignant melanoma stage IV Malignant meningioma metastatic Malignant mesenchymoma

Malignant mesenchymoma metastatic


Final

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Malignant neoplasms Malignant mesenchymoma recurrent Malignant mesenteric neoplasm Malignant middle ear neoplasm Malignant muscle neoplasm Malignant neoplasm of ampulla of Vater Malignant neoplasm of auricular cartilage Malignant neoplasm of choroid Malignant neoplasm of conjunctiva Malignant neoplasm of cornea Malignant neoplasm of eye Malignant neoplasm of eyelid Malignant neoplasm of islets of Langerhans Malignant neoplasm of lacrimal duct Malignant neoplasm of lacrimal gland Malignant neoplasm of orbit Malignant neoplasm of paraurethral glands Malignant neoplasm of placenta Malignant neoplasm of pleura Malignant neoplasm of pleura metastatic Malignant neoplasm of renal pelvis Malignant neoplasm of retina Malignant neoplasm of seminal vesicle Malignant neoplasm of spermatic cord Malignant neoplasm of spinal cord Malignant neoplasm of thorax Malignant neoplasm of thymus Malignant neoplasm of unknown primary site Malignant neoplasm of uterine adnexa Malignant neoplasm papilla of Vater Malignant nervous system neoplasm Malignant nipple neoplasm Malignant nipple neoplasm female Malignant nipple neoplasm male Malignant oligodendroglioma Malignant ovarian cyst Malignant palate neoplasm Malignant pericardial neoplasm Malignant peritoneal neoplasm Malignant pituitary tumour Malignant polyp Malignant respiratory tract neoplasm Malignant splenic neoplasm Malignant sweat gland neoplasm Malignant transformation Malignant urinary tract neoplasm Mantle cell lymphoma Mantle cell lymphoma recurrent Mantle cell lymphoma refractory Mantle cell lymphoma stage I Mantle cell lymphoma stage II Mantle cell lymphoma stage III Mantle cell lymphoma stage IV Marginal zone lymphoma Marginal zone lymphoma recurrent Marginal zone lymphoma refractory Marginal zone lymphoma stage I Marginal zone lymphoma stage II Marginal zone lymphoma stage III Marginal zone lymphoma stage IV Marjolin's ulcer Mastocytic leukaemia Maternal cancer in pregnancy

Mature B-cell type acute leukaemia


Final

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Malignant neoplasms

Medullary carcinoma of breast Medullary thyroid cancer Medulloblastoma Medulloblastoma recurrent Melanoma recurrent Meningioma malignant Mesothelioma malignant Mesothelioma malignant recurrent Metaplastic breast carcinoma Metastases to Eustachian tube Metastases to abdominal cavity Metastases to abdominal wall Metastases to adrenals Metastases to biliary tract Metastases to bladder Metastases to bone Metastases to bone marrow Metastases to breast Metastases to central nervous system Metastases to chest wall Metastases to diaphragm Metastases to eye Metastases to fallopian tube Metastases to gallbladder Metastases to gastrointestinal tract Metastases to heart Metastases to kidney Metastases to larynx Metastases to liver Metastases to lung Metastases to lymph nodes Metastases to meninges Metastases to mouth Metastases to muscle Metastases to nasal sinuses Metastases to neck Metastases to nervous system Metastases to oesophagus Metastases to ovary Metastases to pancreas Metastases to pelvis Metastases to penis Metastases to perineum Metastases to peripheral nervous system Metastases to peripheral vascular system Metastases to peritoneum Metastases to pharynx Metastases to pituitary gland Metastases to placenta Metastases to pleura Metastases to prostate Metastases to rectum Metastases to reproductive organ Metastases to retroperitoneum Metastases to salivary gland Metastases to skin Metastases to soft tissue Metastases to spinal cord Metastases to spine Metastases to spleen Metastases to stomach Metastases to testicle

Metastases to the mediastinum


Date: Version: Status: Page: 03 July 2019 1.0 Final


Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Malignant neoplasms Metastases to the respiratory system Metastases to thorax Metastases to thyroid Metastases to tonsils Metastases to trachea Metastases to urinary tract Metastases to uterus Metastases to vagina Metastasis Metastatic bronchial carcinoma Metastatic carcinoid tumour Metastatic carcinoma of the bladder Metastatic choriocarcinoma Metastatic gastric cancer Metastatic glioma Metastatic glucagonoma Metastatic 1ymphoma Metastatic malignant melanoma Metastatic neoplasm Metastatic nervous system neoplasm Metastatic ocular melanoma Metastatic renal cell carcinoma Metastatic salivary gland cancer Metastatic squamous cell carcinoma Metastatic uterine cancer Microsatellite instability cancer Minimal residual disease Mismatch repair cancer syndrome
Mixed adenoneuroendocrine carcinoma Mixed hepatocellular cholangiocarcinoma Mixed-type liposarcoma Monocytic leukaemia in remission Mucinous adenocarcinoma of appendix Mucinous breast carcinoma Mucinous cystadenocarcinoma ovary Mucinous endometrial carcinoma Mucoepidermoid carcinoma Mucoepidermoid carcinoma of salivary gland Musculoskeletal cancer Mycosis fungoides Mycosis fungoides recurrent Mycosis fungoides refractory Mycosis fungoides stage I Mycosis fungoides stage II Mycosis fungoides stage III Mycosis fungoides stage IV Myeloblastoma Myeloid leukaemia Myeloid leukaemia in remission Myxofibrosarcoma Myxoid liposarcoma NUT midline carcinoma Naevoid melanoma Nasal cavity cancer Nasal sinus cancer Nasopharyngeal cancer Nasopharyngeal cancer metastatic Nasopharyngeal cancer recurrent Nasopharyngeal cancer stage 0 Nasopharyngeal cancer stage I Nasopharyngeal cancer stage II Nasopharyngeal cancer stage III Nasopharyngeal cancer stage IV


 Date:
 03 July 2019

 Version:
 1.0

 Status:
 Final

 Page:

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Natural killer-cell leukaemia Malignant neoplasms Natural killer-cell lymphoblastic lymphoma Neonatal leukaemia Neonatal neuroblastoma Neoplasm malignant Nephroblastoma Neuroblastoma Neuroblastoma recurrent Neuroendocrine breast tumour Neuroendocrine carcinoma Neuroendocrine carcinoma metastatic Neuroendocrine carcinoma of the bladder Neuroendocrine carcinoma of the skin Neuroendocrine tumour Neuroendocrine tumour of the lung Neuroendocrine tumour of the lung metastatic Neurofibrosarcoma Neurofibrosarcoma metastatic Neurofibrosarcoma recurrent Nodal marginal zone B-cell lymphoma Nodal marginal zone B-cell lymphoma recurrent Nodal marginal zone B-cell lymphoma refractory Nodal marginal zone B-cell lymphoma stage I Nodal marginal zone B-cell lymphoma stage II Nodal marginal zone B-cell lymphoma stage III Nodal marginal zone B-cell lymphoma stage IV Nodular lymphocyte predominant Hodgkin lymphoma Nodular melanoma Non-Hodgkin's lymphoma
Non-Hodgkin's lymphoma metastatic
Non-Hodgkin's lymphoma recurrent
Non-Hodgkin's lymphoma refractory Non-Hodgkin's lymphoma stage I Non-Hodgkin's lymphoma stage II Non-Hodgkin's lymphoma stage III Non-Hodgkin's lymphoma stage IV Non-Hodgkin's lymphoma transformed recurrent Non-Hodgkin's lymphoma unspecified histology aggressive Non-Hodgkin's lymphoma unspecified histology aggressive recurrent Non-Hodgkin's lymphoma unspecified histology aggressive refractory Non-Hodgkin's lymphoma unspecified histology aggressive stage I Non-Hodgkin's lymphoma unspecified histology aggressive stage II Non-Hodgkin's lymphoma unspecified histology aggressive stage III Non-Hodgkin's lymphoma unspecified histology aggressive stage IV Non-Hodgkin's lymphoma unspecified histology indolent Non-Hodgkin's lymphoma unspecified histology indolent stage Non-Hodgkin's lymphoma unspecified histology indolent stage Non-Hodgkin's lymphoma unspecified histology indolent stage TTT Non-Hodgkin's lymphoma unspecified histology indolent stage ΤV Non-renal cell carcinoma of kidney Non-small cell lung cancer Non-small cell lung cancer metastatic

Non-small cell lung cancer recurrent


Date: Version: Status: Page: 03 July 2019 1.0 Final


Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Malignant neoplasms Non-small cell lung cancer stage 0 Non-small cell lung cancer stage I Non-small cell lung cancer stage II Non-small cell lung cancer stage III Non-small cell lung cancer stage IIIA Non-small cell lung cancer stage IIIB Non-small cell lung cancer stage IV Nongerminomatous germ cell tumour of the CNS Nonkeratinising carcinoma of nasopharynx Ocular cancer metastatic Ocular haemangiopericytoma Ocular lymphoma
Oesophageal adenocarcinoma Oesophageal adenocarcinoma recurrent Oesophageal adenocarcinoma stage 0 Oesophageal adenocarcinoma stage I Oesophageal adenocarcinoma stage II Oesophageal adenocarcinoma stage III Oesophageal adenocarcinoma stage IV Oesophageal cancer metastatic Oesophageal carcinoma Oesophageal carcinoma recurrent Oesophageal carcinoma stage 0 Oesophageal squamous cell carcinoma Oesophageal squamous cell carcinoma metastatic Oesophageal squamous cell carcinoma recurrent Oesophageal squamous cell carcinoma stage 0 Oesophageal squamous cell carcinoma stage Oesophageal squamous cell carcinoma stage Oesophageal squamous cell carcinoma stage III Oesophageal squamous cell carcinoma stage IV Oestrogen receptor positive breast cancer Oligoastrocytoma Oligodendroglioma Optic glioma Oral cavity cancer metastatic Oropharyngeal cancer Oropharyngeal cancer recurrent Oropharyngeal cancer stage 0 Oropharyngeal cancer stage I Oropharyngeal cancer stage II Oropharyngeal cancer stage III Oropharyngeal cancer stage IV Oropharyngeal lymphoepithelioma Oropharyngeal squamous cell carcinoma Osteosarcoma Osteosarcoma metastatic Osteosarcoma recurrent Otic cancer metastatic Ovarian cancer Ovarian cancer metastatic Ovarian cancer recurrent Ovarian cancer stage I Ovarian cancer stage II Ovarian cancer stage III Ovarian cancer stage IV Ovarian clear cell carcinoma Ovarian dysgerminoma stage I Ovarian dysgerminoma stage II Ovarian dysgerminoma stage III Ovarian dysgerminoma stage IV Ovarian dysgerminoma stage unspecified

Ovarian embryonal carcinoma


03 July 2019 | Novo Nordisk 1.0 Final 70 of 152

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Malignant neoplasms Ovarian endometrioid carcinoma Ovarian epithelial cancer Ovarian epithelial cancer metastatic Ovarian epithelial cancer recurrent Ovarian epithelial cancer stage I Ovarian epithelial cancer stage II Ovarian epithelial cancer stage III Ovarian epithelial cancer stage IV Ovarian germ cell cancer Ovarian germ cell cancer stage I Ovarian germ cell cancer stage II Ovarian germ cell cancer stage III Ovarian germ cell cancer stage IV Ovarian germ cell choriocarcinoma Ovarian germ cell choriocarcinoma stage I Ovarian germ cell choriocarcinoma stage II Ovarian germ cell choriocarcinoma stage III Ovarian germ cell choriocarcinoma stage IV Ovarian germ cell embryonal carcinoma stage I Ovarian germ cell embryonal carcinoma stage I Ovarian germ cell embryonal carcinoma stage III Ovarian germ cell embryonal carcinoma stage IV Ovarian germ cell endodermal sinus tumour Ovarian germ cell endodermal sinus tumour stage I Ovarian germ cell endodermal sinus tumour stage II Ovarian germ cell endodermal sinus tumour stage III Ovarian germ cell endodermal sinus tumour stage IV Ovarian germ cell polyembryoma Ovarian germ cell polyembryoma stage I Ovarian germ cell polyembryoma stage II Ovarian germ cell polyembryoma stage III Ovarian germ cell polyembryoma stage IV Ovarian germ cell teratoma Ovarian germ cell teratoma stage I Ovarian germ cell teratoma stage II Ovarian germ cell teratoma stage III Ovarian germ cell teratoma stage IV Ovarian germ cell tumour mixed Ovarian granulosa-theca cell tumour Ovarian low malignant potential tumour Ovarian stromal cancer Paget's disease of nipple Paget's disease of penis Paget's disease of the vulva Pancoast's tumour Pancreatic carcinoma Pancreatic carcinoma metastatic Pancreatic carcinoma recurrent Pancreatic carcinoma stage Pancreatic carcinoma stage I Pancreatic carcinoma stage II Pancreatic carcinoma stage III Pancreatic carcinoma stage IV Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour metastatic Pancreatic sarcoma Pancreatoblastoma Papillary renal cell carcinoma Papillary serous endometrial carcinoma Papillary thyroid cancer Paraganglion neoplasm malignant Paranasal sinus and nasal cavity malignant neoplasm


Novo Nordisk

1.0

Final

```
Pre-defined MedDRA search
                                                      Preferred term
                                                       Paranasal sinus and nasal cavity malignant neoplasm
Malignant neoplasms
                                                      Paranasal sinus and nasal cavity malignant neoplasm stage O
Paranasal sinus and nasal cavity malignant neoplasm stage I
Paranasal sinus and nasal cavity malignant neoplasm stage II
Paranasal sinus and nasal cavity malignant neoplasm stage
                                                       Paranasal sinus and nasal cavity malignant neoplasm stage IV
                                                       Parathyroid tumour malignant
                                                       Penile cancer
                                                       Penile squamous cell carcinoma
                                                       Penis carcinoma metastatic
                                                       Penis carcinoma recurrent
                                                       Penis carcinoma stage I
                                                       Penis carcinoma stage II
                                                       Penis carcinoma stage III
                                                       Penis carcinoma stage IV
                                                      Pericardial mesothelioma malignant
Pericardial mesothelioma malignant recurrent
Peripheral T-cell lymphoma unspecified
                                                       Peripheral T-cell lymphoma unspecified recurrent
                                                       Peripheral T-cell lymphoma unspecified refractory
                                                       Peripheral T-cell lymphoma unspecified stage I
                                                      Peripheral T-cell lymphoma unspecified stage II
Peripheral T-cell lymphoma unspecified stage III
Peripheral T-cell lymphoma unspecified stage IV
Peripheral neuroepithelioma of bone
Peripheral neuroepithelioma of bone metastatic
                                                       Peripheral neuroepithelioma of bone recurrent
                                                       Peripheral neuroepithelioma of soft tissue
                                                       Peripheral primitive neuroectodermal bone tumour
                                                       Peripheral primitive neuroectodermal tumour of soft tissue
                                                       Peritoneal carcinoma metastatic
                                                       Peritoneal mesothelioma malignant
                                                       Peritoneal mesothelioma malignant recurrent
                                                       Peritoneal sarcoma
                                                       Phaeochromocytoma malignant
                                                       Pharyngeal cancer
                                                       Pharyngeal cancer metastatic
                                                       Pharyngeal cancer recurrent
                                                       Pharyngeal cancer stage 0
                                                       Pharyngeal cancer stage
                                                       Pharyngeal cancer stage II
                                                       Pharyngeal cancer stage III
                                                       Pharyngeal cancer stage IV
                                                       Pilomatrix carcinoma
                                                       Pineal germinoma
                                                       Pineal parenchymal neoplasm malignant
                                                       Pinealoblastomā
                                                      Pituitary cancer metastatic
Pituitary neoplasm malignant recurrent
Plasma cell leukaemia
Plasma cell leukaemia in remission
                                                       Plasma cell myeloma
                                                       Plasma cell myeloma in remission
                                                       Plasma cell myeloma recurrent
                                                       Plasmablastic lymphoma
                                                       Plasmacytoma
                                                      Pleomorphic liposarcoma
Pleomorphic malignant fibrous histiocytoma
                                                       Pleural mesothelioma
Pleural mesothelioma malignant
                                                       Pleural mesothelioma malignant recurrent
```


03 July 2019 | Novo Nordisk 1.0 Final


```
Pre-defined MedDRA search
                                             Preferred term
Malignant neoplasms
                                             Pleural sarcoma
                                             Pleuropulmonary blastoma
                                             Poorly differentiated thyroid carcinoma
                                             Porocarcinoma
                                             Postcricoid cancer
                                             Precursor B-lymphoblastic lymphoma
                                             Precursor B-lymphoblastic lymphoma recurrent
                                             Precursor B-lymphoblastic lymphoma refractory
                                             Precursor B-lymphoblastic lymphoma stage I
                                             Precursor B-lymphoblastic lymphoma stage II
                                             Precursor B-lymphoblastic lymphoma stage III
                                             Precursor B-lymphoblastic lymphoma stage IV
                                             Precursor T-lymphoblastic lymphoma
                                             leukaemia
                                             Precursor T-lymphoblastic lymphoma
                                             leukaemia recurrent
                                             Precursor T-lymphoblastic lymphoma
                                             leukaemia refractory
Precursor T-lymphoblastic lymphoma
                                             leukaemia stage I
                                             Precursor T-lymphoblastic lymphoma
                                             leukaemia stage II
                                             Precursor T-lymphoblastic lymphoma
                                             leukaemia stage III
Precursor T-lymphoblastic lymphoma
leukaemia stage IV
Primary breast lymphoma
                                             Primary cardiac lymphoma
Primary effusion lymphoma
                                             Primary gastrointestinal follicular lymphoma
                                             Primary mediastinal large B-cell lymphoma
Primary mediastinal large B-cell lymphoma recurrent
                                             Primary mediastinal large B-cell lymphoma refractory
                                             Primary mediastinal large B-cell lymphoma stage I
                                             Primary mediastinal large B-cell lymphoma stage II
                                             Primary mediastinal large B-cell lymphoma stage III
                                             Primary mediastinal large B-cell lymphoma stage IV
                                             Primary pulmonary melanoma
Primitive neuroectodermal tumour
                                             Primitive neuroectodermal tumour metastatic
                                             Prolymphocytic leukaemia
                                             Prostate cancer
                                             Prostate cancer metastatic
                                             Prostate cancer recurrent
                                             Prostate cancer stage 0
                                             Prostate cancer stage
                                             Prostate cancer stage II
                                             Prostate cancer stage III
                                             Prostate cancer stage IV
                                             Pseudosarcoma
                                             Queyrat erythroplasia
                                             Rectal adenocarcinoma
Rectal cancer
                                             Rectal cancer metastatic
                                             Rectal cancer recurrent
                                             Rectal cancer stage 0
                                             Rectal cancer stage I
                                             Rectal cancer stage II
                                             Rectal cancer stage III
                                             Rectal cancer stage IV
                                             Rectosigmoid cancer
                                             Rectosigmoid cancer metastatic
                                             Rectosigmoid cancer recurrent
```


Date: Version: Status: Page: 03 July 2019 1.0 Final 73 of 152

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Malignant neoplasms Rectosigmoid cancer stage 0 Rectosigmoid cancer stage I Rectosigmoid cancer stage II Rectosigmoid cancer stage III Rectosigmoid cancer stage IV Recurrent cancer Refractory cancer Renal cancer Renal cancer metastatic Renal cancer recurrent Renal cancer stage I Renal cancer stage II Renal cancer stage III Renal cancer stage IV Renal cell carcinoma Renal cell carcinoma recurrent Renal cell carcinoma stage I Renal cell carcinoma stage II Renal cell carcinoma stage III Renal cell carcinoma stage IV Respiratory tract carcinoma in situ Retinal melanoma Retinoblastoma Retroperitoneal cancer Retroperitoneal neoplasm metastatic Rhabdoid tumour Rhabdoid tumour of the kidney Rhabdomyosarcoma Rhabdomyosarcoma recurrent Richter's syndrome Round cell liposarcoma Salivary gland cancer Salivary gland cancer recurrent Salivary gland cancer stage 0 Salivary gland cancer stage I Salivary gland cancer stage II Salivary gland cancer stage III Salivary gland cancer stage IV Sarcoma Sarcoma metastatic Sarcoma of skin Sarcoma uterus Sarcomatoid carcinoma Sarcomatoid carcinoma of the lung Sarcomatoid mesothelioma Sarcomatosis Scrotal cancer Sebaceous carcinoma Second primary malignancy Seminoma Serous cystadenocarcinoma ovary Signet-ring cell carcinoma Sinus cancer metastatic Skin angiosarcoma Skin cancer Skin cancer metastatic Skin squamous cell carcinoma metastatic Skin squamous cell carcinoma recurrent Small cell carcinoma Small cell carcinoma of the cervix Small cell lung cancer

Small cell lung cancer extensive stage Small cell lung cancer limited stage


03 July 2019 | Novo Nordisk 1.0 Final


Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Malignant neoplasms Small cell lung cancer metastatic Small cell lung cancer recurrent Small intestine adenocarcinoma Small intestine carcinoma Small intestine carcinoma metastatic Small intestine carcinoma recurrent Small intestine carcinoma stage 0 Small intestine carcinoma stage Small intestine carcinoma stage Small intestine carcinoma stage III Small intestine carcinoma stage IV Small intestine leiomyosarcoma Soft tissue sarcoma Solid pseudopapillary tumour of the pancreas Spermatocytic seminoma Spinal meningioma malignant Spindle cell sarcoma Splenic marginal zone lymphoma Splenic marginal zone lymphoma recurrent Splenic marginal zone lymphoma refractory Splenic marginal zone lymphoma stage I Splenic marginal zone lymphoma stage II Splenic marginal zone lymphoma stage III Splenic marginal zone lymphoma stage IV Squamous cell breast carcinoma Squamous cell carcinoma Squamous cell carcinoma of head and neck Squamous cell carcinoma of lung Squamous cell carcinoma of pharynx Squamous cell carcinoma of skin Squamous cell carcinoma of the cervix Squamous cell carcinoma of the hypopharynx Squamous cell carcinoma of the oral cavity Squamous cell carcinoma of the tonque Squamous cell carcinoma of the vagina Squamous cell carcinoma of the vulva Squamous endometrial carcinoma Stewart-Treves syndrome Superficial spreading melanoma stage I Superficial spreading melanoma stage II Superficial spreading melanoma stage III Superficial spreading melanoma stage IV Superficial spreading melanoma stage unspecified Synovial sarcoma Synovial sarcoma metastatic Synovial sarcoma recurrent T-cell chronic lymphocytic leukaemia T-cell lymphoma T-cell lymphoma recurrent T-cell lymphoma refractory T-cell lymphoma stage I T-cell lymphoma stage II T-cell lymphoma stage III T-cell lymphoma stage IV T-cell prolymphocytic leukaemia T-cell type acute leukaemia T-cell unclassifiable lymphoma high grade T-cell unclassifiable lymphoma low grade Testicular cancer metastatic Testicular choriocarcinoma Testicular choriocarcinoma recurrent Testicular choriocarcinoma stage I Testicular choriocarcinoma stage II


03 July 2019 1.0 Final


Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Testicular choriocarcinoma stage III Malignant neoplasms Testicular embryonal carcinoma Testicular embryonal carcinoma stage I Testicular embryonal carcinoma stage II Testicular embryonal carcinoma stage III Testicular germ cell cancer Testicular germ cell cancer metastatic Testicular germ cell tumour mixed Testicular germ cell tumour mixed stage I Testicular germ cell tumour mixed stage II Testicular germ cell tumour mixed stage III Testicular leiomyosarcoma Testicular malignant teratoma Testicular malignant teratoma stage I Testicular malignant teratoma stage II Testicular malignant teratoma stage III Testicular seminoma (pure) Testicular seminoma (pure) stage I Testicular seminoma (pure) stage II Testicular seminoma (pure) stage III Testicular yolk sac tumour Testicular yolk sac tumour stage I Testicular yolk sac tumour stage II Testicular yolk sac tumour stage III Testis cancer Testis cancer recurrent Throat cancer Thymic cancer metastatic Thymoma malignant Thymoma malignant recurrent Thyroid B-cell lymphoma Thyroid cancer Thyroid cancer metastatic Thyroid cancer recurrent Thyroid cancer stage 0 Thyroid cancer stage I Thyroid cancer stage II Thyroid cancer stage III Thyroid cancer stage IV Tonque cancer metastatic Tongue cancer recurrent Tongue carcinoma stage 0 Tongue carcinoma stage I Tongue carcinoma stage II Tonque carcinoma stage III Tonque carcinoma stage IV Tongue neoplasm malignant stage unspecified Tonsil cancer Tonsil cancer metastatic Tracheal cancer Transformation to acute myeloid leukaemia Transitional cell cancer of renal pelvis and ureter metastatic Transitional cell cancer of the renal pelvis and ureter Transitional cell cancer of the renal pelvis and ureter Transitional cell cancer of the renal pelvis and ureter recurrent Transitional cell cancer of the renal pelvis and ureter regional Transitional cell carcinoma Transitional cell carcinoma metastatic

Transitional cell carcinoma recurrent


03 July 2019 Date: Version: Final Status: 

Novo Nordisk

1.0

```
Pre-defined MedDRA search
                                            Preferred term
Malignant neoplasms
                                            Transitional cell carcinoma urethra
                                            Trichoblastic carcinoma
                                            Triple hit lymphoma
                                            Triple negative breast cancer
                                            Tubular breast carcinoma
                                            Tumour budding
                                            Undifferentiated carcinoma of colon
                                            Undifferentiated nasopharyngeal carcinoma
                                            Undifferentiated sarcoma
                                            Ureteric cancer
                                            Ureteric cancer local
                                            Ureteric cancer metastatic
                                            Ureteric cancer recurrent
                                            Ureteric cancer regional
                                            Urethral cancer
                                            Urethral cancer metastatic
                                            Urethral cancer recurrent
                                            Urethral melanoma metastatic
                                            Urinary bladder sarcoma
Urinary tract carcinoma in situ
                                            Uterine cancer
                                            Uterine carcinoma in situ
                                            Uterine leiomyosarcoma
                                            Uveal melanoma
                                            Vaginal adenocarcinoma
Vaginal cancer
                                            Vaginal cancer metastatic
                                            Vaginal cancer recurrent
                                            Vaginal cancer stage 0
                                            Vaginal cancer stage I
                                            Vaginal cancer stage II
                                            Vaginal cancer stage III
                                            Vaginal cancer stage IVA
                                            Vaginal cancer stage IVB
                                            Vuĺval cancer
                                            Vulval cancer metastatic
                                            Vulval cancer recurrent
                                            Vulval cancer stage 0
                                            Vulval cancer stage
                                            Vulval cancer stage II
                                            Vulval cancer stage III
                                            Vulval cancer stage IV
                                            Vulvar adenocarcinoma
                                            Waldenstrom's macroglobulinaemia
                                            Waldenstrom's macroglobulinaemia recurrent
Waldenstrom's macroglobulinaemia refractory
                                            Waldenstrom's macroglobulinaemia stage I
                                            Waldenstrom's macroglobulinaemia stage II
                                            Waldenstrom's macroglobulinaemia stage III
Waldenstrom's macroglobulinaemia stage IV
                                            Accidental device ingestion Accidental device ingestion by a child
Medication error and overdose
                                            Accidental exposure to product
                                            Accidental exposure to product by child
                                            Accidental exposure to product packaging
                                            Accidental exposure to product packaging by child
                                            Accidental overdose
                                            Accidental poisoning
                                            Accidental underdose
                                            Accidental use of placebo
                                            Assisted suicide
                                            Booster dose missed
```

 Date:
 03 July 2019

 Version:
 1.0

 Status:
 Final

 Page:

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Circumstance or information capable of leading to device Medication error and overdose Circumstance or information capable of leading to medication error Completed suicide Complication of device insertion Complication of device removal Complication of drug delivery system removal Contraindicated device used Contraindicated product administered Contraindicated product prescribed Contraindication to medical treatment Contraindication to vaccination Deprescribing error Device adhesion issue Device connection issue Device difficult to use Device dispensing error Device infusion issue Device malfunction Device monitoring procedure not performed Device programming error Device use error Device use issue Device used for unapproved schedule Device-device incompatibility Dietary supplement prescribing error Discontinued product administered
Documented hypersensitivity to administered product Dopamine dysregulation syndrome Dose calculation error Drug abuse Drug abuser Drug administered in wrong device Drug dependence Drug dependence, antepartum Drug dependence, postpartum Drug dispensed to wrong patient Drug dose omission by device Drug dose titration not performed Drug monitoring procedure incorrectly performed Drug monitoring procedure not performed Drug titration error Drug use disorder Drug use disorder, antepartum Drug use disorder, postpartum Duplicate therapy error Expired device used Expired product administered Exposure to contaminated device Exposure via contaminated device Exposure via direct contact Exposure via eye contact Exposure via ingestion Exposure via inhalation Exposure via partner Exposure via skin contact Exposure via unknown route Extra dose administered
Failure of child resistant mechanism for pharmaceutical product Failure to suspend medication Implantation complication


 Date:
 03 July 2019

 Version:
 1.0

 Status:
 Final

Page:

2019 Novo Nordisk 1.0 Final


Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Medication error and overdose

Inadequate aseptic technique in use of product Inappropriate schedule of product administration Incomplete course of vaccination Incorrect disposal of product Incorrect dosage administered Incorrect dose administered
Incorrect dose administered by device Incorrect dose administered by product Incorrect drug administration rate Incorrect product administration duration Incorrect product dosage form administered Incorrect product dosage form administered Incorrect product formulation administered Incorrect route of product administration Injury associated with device Intentional device misuse Intentional dose omission Intentional misuse of drug delivery system Intentional overdose Intentional product misuse Intentional self-injury Intercepted accidental exposure to product by child Intercepted medication error Intercepted product administration error Intercepted product dispensing error Intercepted product dispensing error
Intercepted product preparation error
Intercepted product prescribing error
Intercepted product selection error Intercepted product storage error Intercepted wrong patient selected Interchange of vaccine products
Labelled drug-disease interaction medication error Labelled drug-drug interaction medication error Labelled drug-food interaction medication error Lack of administration site rotation Lack of application site rotation Lack of infusion site rotation Lack of injection site rotation Lack of vaccination site rotation Maternal use of illicit drugs Medical device monitoring error Medication error Multiple use of single-use product Needle issue Neonatal complications of substance abuse Occupational exposure to product Occupational exposure to radiation Overdose Paravenous drug administration Performance enhancing product use Poisoning deliberate Poor quality device used Poor quality product administered Prescribed overdose Prescribed underdose Product adhesion issue Product administered at inappropriate site Product administered to patient of inappropriate age Product administration error Product administration interrupted Product appearance confusion Product barcode issue Product commingling


Page:

1.0 Final 79 of 152 Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

```
Pre-defined MedDRA search
                                               Preferred term
Medication error and overdose
                                               Product communication issue
                                               Product compounding quality issue
                                               Product design confusion
                                               Product dispensing error
                                               Product dispensing issue
                                               Product dosage form confusion
                                               Product dosage form issue
                                               Product dose omission
                                               Product dropper issue
                                               Product expiration date issue
                                               Product identification number issue
                                               Product label confusion
                                               Product label issue
                                               Product label on wrong product
                                               Product lot number issue
                                               Product monitoring error
                                               Product name confusion
                                               Product packaging confusion
Product packaging issue
Product preparation error
                                               Product preparation issue
                                               Product prescribing error
                                               Product prescribing issue
                                               Product reconstitution quality issue
                                               Product selection error
                                               Product storage error
Product substitution error
                                               Product use complaint
                                               Product use in unapproved indication
                                               Product use in unapproved therapeutic environment
                                               Product use issue
                                               Radiation overdose
                                               Radiation underdose
                                               Recalled product administered
                                               Single component of a two-component product administered
                                               Substance abuse
                                               Substance abuser
                                               Substance dependence
Substance use disorder
                                               Suicide attempt
                                               Suspected suicide attempt
                                               Syringe issue
                                               Therapeutic drug monitoring analysis incorrectly performed Therapeutic drug monitoring analysis not performed
                                               Transcription medication error Transfusion with incompatible blood
                                               Treatment noncompliance
                                               Underdose
                                               Unintentional medical device removal
                                               Unintentional use for unapproved indication
                                               Vaccination error
                                               Wrong device used Wrong dosage form
                                               Wrong dosage formulation
                                               Wrong dose
                                               Wrong drug
                                               Wrong patient received product
                                               Wrong product administered Wrong product procured
                                               Wrong product stored Wrong rate
                                               Wrong schedule
                                               Wrong strength
```


Final 80 of 152

Novo Nordisk

 ${\tt Pre-defined} \ {\tt MedDRA} \ {\tt search} \ {\tt -list} \ {\tt of} \ {\tt preferred} \ {\tt terms}$ 

Pre-defined MedDRA search Preferred term Wrong technique in device usage process Medication error and overdose Wrong technique in product usage process 5q minus syndrome ACTH-producing pituitary tumour Neoplasm APUDoma Abdominal neoplasm Abdominal wall cyst Abdominal wall neoplasm Abdominal wall neoplasm benign Abdominal wall neoplasm malignant Acanthoma Acanthosis nigricans Acinar cell carcinoma of pancreas Acinic cell carcinoma of salivary gland Acoustic neuroma Acquired C1 inhibitor deficiency Acquired bronchial cyst Acquired thalassaemia Acral lentiginous melanoma Acral lentiginous melanoma stage I Acral lentiginous melanoma stage II Acral lentiginous melanoma stage III Acral lentiginous melanoma stage IV Acrochordon Acrokeratosis paraneoplastica Actinic keratosis Acute bilineal leukaemia Acute biphenotypic leukaemia Acute leukaemia Acute leukaemia in remission Acute lymphocytic leukaemia Acute lymphocytic leukaemia (in remission) Acute lymphocytic leukaemia recurrent Acute lymphocytic leukaemia refractory Acute megakaryocytic leukaemia Acute megakaryocytic leukaemia (in remission) Acute monocytic leukaemia
Acute monocytic leukaemia (in remission)
Acute myeloid leukaemia Acute myeloid leukaemia (in remission) Acute myeloid leukaemia recurrent Acute myeloid leukaemia refractory Acute myelomonocytic leukaemia Acute promyelocytic leukaemia Acute undifferentiated leukaemia Adenocarcinoma Adenocarcinoma gastric Adenocarcinoma of appendix Adenocarcinoma of colon Adenocarcinoma of salivary gland Adenocarcinoma of the cervix Adenocarcinoma pancreas Adenoid cystic carcinoma Adenoid cystic carcinoma of external auditory canal Adenoid cystic carcinoma of salivary gland Adenolipoma Adenolymphoma Adenoma benign Adenomatous polyposis coli Adenosquamous carcinoma of the cervix Adenosquamous carcinoma of vagina Adenosquamous cell carcinoma


Final

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Neoplasm

Pre-defined MedDRA search

Preferred term

recurrent

refractory

Adenosquamous cell lung cancer

Adenosquamous cell lung cancer recurrent Adenosquamous cell lung cancer stage 0 Adenosquamous cell lung cancer stage I Adenosquamous cell lung cancer stage II Adenosquamous cell lung cancer stage III Adenosquamous cell lung cancer stage IV Administration site cyst Adnexa uteri cyst Adrenal adenoma Adrenal cyst Adrenal gland cancer Adrenal gland cancer metastatic Adrenal neoplasm Adrenocortical carcinoma Adult T-cell lymphoma leukaemia Adult T-cell lymphoma leukaemia recurrent Adult T-cell lymphoma leukaemia refractory Adult T-cell lymphoma leukaemia stage I Adult T-cell lymphoma leukaemia stage II Adult T-cell lymphoma leukaemia stage III Adult T-cell lymphoma leukaemia stage IV Aesthesioneuroblastoma Alcoholisation procedure Aleukaemic leukaemia Alpha 1 foetoprotein abnormal Alpha 1 foetoprotein increased Alpha interferon therapy Alpha-L-fucosidase increased Alveolar rhabdomyosarcoma Alveolar soft part sarcoma Alveolar soft part sarcoma metastatic Alveolar soft part sarcoma recurrent Ameloblastoma Ampullary polyp Amputation of penis Amyloidoma Anal cancer Anal cancer metastatic Anal cancer recurrent Anal cancer stage 0 Anal cancer stage Anal cancer stage II Anal cancer stage III Anal cancer stage IV Anal leukoplakia Anal neoplasm Anal polyp Anal polypectomy Anal squamous cell carcinoma Anaplastic astrocytoma Anaplastic large cell lymphoma T- and null-cell types Anaplastic large cell lymphoma T- and null-cell types

Anaplastic large cell lymphoma T- and null-cell types


Date: Version: Status: Page: 03 July 2019 1.0 Final


Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

```
Pre-defined MedDRA search
                                                 Preferred term
                                                 Anaplastic large cell lymphoma T- and null-cell types stage
Neoplasm
                                                 Anaplastic large cell lymphoma T- and null-cell types stage
                                                 Anaplastic large cell lymphoma T- and null-cell types stage
                                                 Anaplastic large cell lymphoma T- and null-cell types stage
                                                 Anaplastic large-cell lymphoma
                                                 Anaplastic lymphoma kinase gene and nucleophosmin gene
                                                 fusion overexpression
                                                 Anaplastic meningioma
Anaplastic oligodendroglioma
                                                 Anaplastic thyroid cancer
                                                 Androgen therapy
                                                 Aneurysmal bone cyst
                                                 Angiocentric glioma
                                                 Angiocentric lymphoma recurrent
                                                 Angiocentric lymphoma refractory
                                                 Angiocentric lymphoma stage I
                                                 Angiocentric lymphoma stage II
                                                 Angiocentric lymphoma stage III
                                                 Angiocentric lymphoma stage IV
                                                 Angiofibroma
                                                 Angiogenesis biomarker increased
Angioimmunoblastic T-cell lymphoma
Angioimmunoblastic T-cell lymphoma recurrent
                                                 Angioimmunoblastic T-cell lymphoma refractory
                                                 Angioimmunoblastic T-cell lymphoma stage I
Angioimmunoblastic T-cell lymphoma stage II
Angioimmunoblastic T-cell lymphoma stage III
                                                 Angioimmunoblastic T-cell lymphoma stage IV
                                                 Angiolipoma
                                                 Angiomyofibroblastoma
                                                 Angiomyolipoma
                                                 Angiomyxoma
                                                 Angiosarcoma
                                                 Angiosarcoma metastatic
                                                 Angiosarcoma non-metastatic
                                                 Angiosarcoma recurrent
                                                 Anogenital dysplasia
                                                 Anogenital warts
                                                 Anorectal haemangioma
Anti-NMDA antibody positive
Anti-VGCC antibody positive
                                                 Anti-androgen withdrawal syndrome
                                                 Antiandrogen therapy
                                                 Antioestrogen therapy
                                                 Apocrine breast carcinoma
                                                 Appendix adenoma
                                                 Appendix cancer
Application site cyst
                                                 Arachnoid cyst
Arsenical keratosis
                                                 Aspiration bone marrow abnormal
                                                 Astroblastoma
                                                 Astrocytoma
                                                 Astrocytoma malignant
                                                 Astrocytoma, low grade
Atypical fibroxanthoma
Atypical teratoid
                                                 rhabdoid tumour of CNS
```


 Date:
 03 July 2019

 Version:
 1.0

 Status:
 Final

 Page:

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Neoplasm Aural cystadenoma Aural polyp Autologous bone marrow transplantation therapy Axillary lymphadenectomy
B precursor type acute leukaemia
B-cell depletion therapy B-cell lymphoma B-cell lymphoma recurrent B-cell lymphoma refractory B-cell lymphoma stage I B-cell lymphoma stage II B-cell lymphoma stage III B-cell lymphoma stage IV B-cell prolymphocytic leukaemia B-cell small lymphocytic lymphoma B-cell small lymphocytic lymphoma recurrent B-cell small lymphocytic lymphoma refractory B-cell small lymphocytic lymphoma stage I B-cell small lymphocytic lymphoma stage II B-cell small lymphocytic lymphoma stage III B-cell small lymphocytic lymphoma stage IV B-cell type acute leukaemia B-cell unclassifiable lymphoma high grade B-cell unclassifiable lymphoma low grade Bannayan-Riley-Ruvalcaba syndrome Barrett's oesophagus Bartholin's cyst Basal cell carcinoma
Basal cell naevus syndrome Basosquamous carcinoma Basosquamous carcinoma of skin Becker's naevus Bence Jones proteinuria Benign abdominal neoplasm Benign anorectal neoplasm Benign biliary neoplasm Benign bone neoplasm Benign breast neoplasm Benign cardiac neoplasm Benign cartilage neoplasm Benign duodenal neoplasm Benign ear neoplasm Benign endocrine neoplasm Benign fallopian tube neoplasm Benign female reproductive tract neoplasm Benign gastric neoplasm Benign gastrointestinal neoplasm Benign genitourinary tract neoplasm Benign hepatic neoplasm Benign hepatobiliary neoplasm Benign hydatidiform mole Benign joint neoplasm Benign laryngeal neoplasm Benign lung neoplasm Benign lymph node neoplasm Benign male reproductive tract neoplasm Benign mediastinal neoplasm Benign mesenteric neoplasm Benign mesothelioma Benign middle ear neoplasm Benign muscle neoplasm Benign neoplasm Benign neoplasm of adrenal gland


Final

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Benign neoplasm of ampulla of Vater Benign neoplasm of bladder Neoplasm Benign neoplasm of cervix uteri Benign neoplasm of choroid Benign neoplasm of conjunctiva Benign neoplasm of cornea Benign neoplasm of epididymis Benign neoplasm of eye Benign neoplasm of eyelid Benign neoplasm of islets of Langerhans Benign neoplasm of lacrimal duct Benign neoplasm of lacrimal gland Benign neoplasm of optic nerve Benign neoplasm of orbit Benign neoplasm of pineal gland Benign neoplasm of prostate Benign neoplasm of retina Benign neoplasm of scrotum
Benign neoplasm of seminal vesicle Benign neoplasm of skin Benign neoplasm of spinal cord Benign neoplasm of testis Benign neoplasm of thymus Benign neoplasm of thyroid gland Benign neoplasm of ureter Benign neoplasm of urethra Benign nipple neoplasm Benign oesophageal neoplasm Benign ovarian tumour Benign pancreatic neoplasm Benign penile neoplasm Benign pericardium neoplasm Benign peritoneal neoplasm Benign pleural mesothelioma Benign pleural neoplasm Benign renal neoplasm Benign respiratory tract neoplasm Benign salivary gland neoplasm Benign small intestinal neoplasm Benign soft tissue neoplasm Benign spleen tumour Benign tracheal neoplasm Benign urinary tract neoplasm Benign uterine neoplasm Benign vaginal neoplasm Benign vascular neoplasm Benign vulval neoplasm Beta interferon therapy Bile duct adenocarcinoma Bile duct adenosquamous carcinoma Bile duct cancer Bile duct cancer recurrent Bile duct cancer stage 0 Bile duct cancer stage I Bile duct cancer stage II Bile duct cancer stage III Bile duct cancer stage IV Bile duct squamous cell carcinoma Biliary adenoma
Biliary cancer metastatic Biliary cyst Biliary hamartoma

Biliary neoplasm


03 July 2019

1.0 Final 85 of 152 Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Neoplasm Biliary polyp Bing-Neel syndrome Bing-Neel syndrome
Biopsy abdominal wall abnormal
Biopsy adrenal gland abnormal
Biopsy anus abnormal
Biopsy artery abnormal
Biopsy bile duct abnormal
Biopsy bladder abnormal Biopsy blood vessel abnormal Biopsy bone abnormal Biopsy bone marrow abnormal Biopsy brain abnormal Biopsy breast abnormal Biopsy bronchus abnormal Biopsy cartilage abnormal Biopsy cervix abnormal Biopsy chest wall abnormal Biopsy chorionic villous abnormal Biopsy colon abnormal Biopsy conjunctiva abnormal Biopsy cornea abnormal Biopsy diaphragm abnormal Biopsy diaphragm abnormal Biopsy ear abnormal Biopsy endometrium abnormal Biopsy epididymis abnormal Biopsy eyelid abnormal Biopsy fallopian tube abnormal Biopsy foetal abnormal Biopsy gallbladder abnormal Biopsy heart abnormal Biopsy intestine abnormal Biopsy kidney abnormal Biopsy larynx abnormal Biopsy ligament abnormal Biopsy lip abnormal Biopsy liver abnormal Biopsy lung abnormal Biopsy lymph gland abnormal Biopsy mucosa abnormal Biopsy muscle abnormal Biopsy oesophagus abnormal Biopsy ovary abnormal Biopsy palate abnormal Biopsy pancreas abnormal Biopsy parathyroid gland abnormal Biopsy penis abnormal Biopsy pericardium abnormal Biopsy peripheral nerve abnormal Biopsy perintoneum abnormal Biopsy pharynx abnormal Biopsy pleura abnormal Biopsy prostate abnormal Biopsy rectum abnormal Biopsy retina abnormal Biopsy salivary gland abnormal Biopsy sclera abnormal Biopsy sciera abnormal
Biopsy seminal vesicle abnormal
Biopsy site unspecified abnormal
Biopsy skin abnormal
Biopsy small intestine abnormal
Biopsy spinal cord abnormal
Biopsy spleen abnormal

Biopsy stomach abnormal


Final 86 of 152

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Neoplasm Biopsy tendon abnormal Biopsy testes abnormal Biopsy thymus gland abnormal Biopsy thyroid gland abnormal Biopsy tongue abnormal Biopsy trachea abnormal Biopsy urethra abnormal Biopsy uterus abnormal Biopsy vagina abnormal Biopsy vocal cord abnormal Biopsy vulva abnormal Biotherapy Biphasic mesothelioma Birt-Hogg-Dube syndrome Bladder adenocarcinoma recurrent Bladder adenocarcinoma stage 0 Bladder adenocarcinoma stage I Bladder adenocarcinoma stage II Bladder adenocarcinoma stage III Bladder adenocarcinoma stage IV Bladder adenocarcinoma stage unspecified Bladder cancer Bladder cancer recurrent Bladder cancer stage 0, with cancer in situ Bladder cancer stage 0, without cancer in situ Bladder cancer stage I, with cancer in situ Bladder cancer stage I, without cancer in situ Bladder cancer stage II Bladder cancer stage III Bladder cancer stage IV Bladder cyst Bladder dysplasia Bladder leukoplakia Bladder mapping Bladder neck resection Bladder neoplasm Bladder neoplasm surgery Bladder papilloma Bladder polypectomy Bladder squamous cell carcinoma recurrent Bladder squamous cell carcinoma stage 0 Bladder squamous cell carcinoma stage I Bladder squamous cell carcinoma stage II Bladder squamous cell carcinoma stage III Bladder squamous cell carcinoma stage IV Bladder squamous cell carcinoma stage unspecified Bladder transitional cell carcinoma Bladder transitional cell carcinoma metastatic Bladder transitional cell carcinoma recurrent Bladder transitional cell carcinoma stage 0 Bladder transitional cell carcinoma stage I Bladder transitional cell carcinoma stage II Bladder transitional cell carcinoma stage III Bladder transitional cell carcinoma stage IV Blast cell count increased Blast cell crisis Blast cell proliferation Blast cells present Blast crisis in myelogenous leukaemia Blastic plasmacytoid dendritic cell neoplasia Blepharal papilloma Blood chromogranin A increased

Bone cancer


Page:

1.0 Final 87 of 152 Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Neoplasm Bone cancer metastatic Bone cyst Bone giant cell tumour Bone giant cell tumour benign Bone giant cell tumour malignant Bone marrow infiltration Bone marrow leukaemic cell infiltration Bone marrow reticulin fibrosis Bone marrow tumour cell infiltration Bone neoplasm Bone sarcoma Bone scan abnormal Borderline mucinous tumour of ovary Borderline ovarian tumour Borderline serous tumour of ovary Bowen's disease Bowenoid papulosis Brachytherapy Brachytherapy to eye Brachytherapy to penis Brachytherapy to tongue Brachytherapy to tonsil Brain cancer metastatic Brain neoplasm Brain neoplasm benign Brain neoplasm malignant Brain sarcoma Brain scan abnormal Brain stem glioma Brain stem glioma benign Brain teratoma
Brain tumour operation Branchial cyst Breakthrough pain Breast adenoma Breast angiosarcoma Breast angiosarcoma metastatic Breast calcifications Breast cancer Breast cancer female Breast cancer in situ Breast cancer male Breast cancer metastatic Breast cancer recurrent Breast cancer stage I Breast cancer stage II Breast cancer stage III Breast cancer stage IV Breast capsulotomy Breast conserving surgery Breast cyst Breast cyst rupture Breast dysplasia Breast fibroma Breast neoplasm Breast proliferative changes Breast prosthesis implantation Breast reconstruction Breast sarcoma Breast sarcoma metastatic Breast sarcoma recurrent Breast tumour excision

Brenner tumour

Pre-defined MedDRA search


Preferred term


03 July 2019 1.0 Final


Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Neoplasm Bronchial carcinoma Bronchial neoplasm Bronchial neoplasm benign Bronchial polyp Bronchioloalveolar carcinoma Buccal polyp Burkitt's leukaemia Burkitt's lymphoma Burkitt's lymphoma recurrent Burkitt's lymphoma refractory Burkitt's lymphoma stage I Burkitt's lymphoma stage II Burkitt's lymphoma stage III Burkitt's lymphoma stage IV Buschke-Lowenstein's tumour C-kit gene negative CD20 antigen positive CD25 antigen positive CD30 expression CNS germinoma CSF lymphocyte count abnormal CSF lymphocyte count increased Cachexia Calcifying fibrous pseudotumour Cancer hormonal therapy Cancer in remission Cancer pain Cancer staging Cancer surgery Carbohydrate antigen 125 increased Carbohydrate antigen 15-3 increased Carbohydrate antigen 19-9 increased Carbohydrate antigen 27.29 increased Carbohydrate antigen 549 increased Carbohydrate antigen 72-4 Carcinoembryonic antigen decreased Carcinoembryonic antigen increased Carcinogenic effect in offspring Carcinoid crisis Carcinoid heart disease Carcinoid syndrome Carcinoid tumour Carcinoid tumour of the appendix Carcinoid tumour of the caecum Carcinoid tumour of the duodenum

Cardiac haemangioma benign

Carcinoma in situ
Carcinoma in situ of eye
Carcinoma in situ of penis
Carcinoma in situ of skin
Carcinoma in situ of trachea
Carcinomatous polyarthritis

Cardiac fibroma

Carcinoid tumour of the gastrointestinal tract

Carcinoid tumour of the liver
Carcinoid tumour of the ovary
Carcinoid tumour of the pancreas
Carcinoid tumour of the prostate
Carcinoid tumour of the small bowel
Carcinoid tumour of the stomach
Carcinoid tumour pulmonary
Carcinoma ex-pleomorphic adenoma


 Date:
 03 July 2019

 Version:
 1.0

 Status:
 Final

 Page:

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Neoplasm Cardiac myxoma Cardiac neoplasm malignant Cardiac neoplasm unspecified Cardiac neurofibroma Cardiac teratoma Cardiac valve fibroelastoma Carney complex Carotid body tumour Cartilage neoplasm Castleman's disease Cell marker increased Cell-free and concentrated ascites reinfusion therapy Cementoblastoma Cementoplasty Central nervous system dermoid tumour Central nervous system leukaemia Central nervous system lymphoma Central nervous system melanoma Central nervous system neoplasm Central nervous system neuroblastoma Cerebellar haemangioma Cerebellar tumour Cerebellopontine angle tumour Cerebral cyst Cerebral haemangioma Cervical cyst Cervical dysplasia Cervical polyp Cervix adenomatous polyp Cervix cancer metastatic Cervix carcinoma Cervix carcinoma recurrent Cervix carcinoma stage 0 Cervix carcinoma stage I Cervix carcinoma stage II Cervix carcinoma stage III Cervix carcinoma stage IV Cervix neoplasm Cervix tumour excision Cervix warts Chemical peel of skin Chemodectoma Chemotherapy Chemotherapy cardiotoxicity attenuation Chemotherapy cytokine prophylaxis
Chemotherapy extravasation management
Chemotherapy multiple agents systemic
Chemotherapy neurotoxicity attenuation Chemotherapy sensitivity and resistance assay Chemotherapy single agent systemic Chemotherapy urothelial toxicity attenuation Chest wall cyst Chest wall tumour Chiasma syndrome Chloroma Chloroma (in remission) Cholangioadenoma Cholangiocarcinoma Cholangiosarcoma Choledochal cyst Cholesteatoma Cholesterin granuloma of middle ear Cholesterol granuloma


Final 90 of 152

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Chondroblastoma Neoplasm Chondroma Chondromatosis Chondrosarcoma Chondrosarcoma metastatic Chondrosarcoma recurrent Chordoma Choriocarcinoma Choroid fissure cyst Choroid melanoma Choroid neoplasm Choroid plexus carcinoma Choroid plexus papilloma Choroid tumour excision Choroidal haemangioma Chromophobe renal cell carcinoma Chronic eosinophilic leukaemia Chronic leukaemia Chronic leukaemia in remission Chronic lymphocytic leukaemia Chronic lymphocytic leukaemia (in remission) Chronic lymphocytic leukaemia recurrent Chronic lymphocytic leukaemia refractory Chronic lymphocytic leukaemia stage 0 Chronic lymphocytic leukaemia stage 1 Chronic lymphocytic leukaemia stage 2 Chronic lymphocytic leukaemia stage 3 Chronic lymphocytic leukaemia stage Chronic lymphocytic leukaemia transformation Chronic myeloid leukaemia Chronic myeloid leukaemia (in remission) Chronic myeloid leukaemia recurrent Chronic myeloid leukaemia transformation Chronic myelomonocytic leukaemia Chronic myelomonocytic leukaemia (in remission) Chronic rhinosinusitis with nasal polyps Ciliary body melanoma Clear cell carcinoma of cervix Clear cell endometrial carcinoma Clear cell renal cell carcinoma Clear cell sarcoma of soft tissue Clear cell sarcoma of the kidney Clonal evolution Colectomy Colectomy total Colloid brain cyst Colon adenoma Colon cancer Colon cancer metastatic Colon cancer recurrent Colon cancer stage 0 Colon cancer stage I Colon cancer stage II Colon cancer stage III Colon cancer stage IV Colon dysplasia Colon neoplasm Colony stimulating factor therapy Colorectal adenocarcinoma Colorectal cancer Colorectal cancer metastatic Colorectal cancer recurrent Colorectal cancer stage I


03 July 2019 | **Novo Nordisk** 

Final 91 of 152

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Neoplasm Colorectal cancer stage II Colorectal cancer stage III Colorectal cancer stage IV Colorectal carcinoma stage 0 Composite lymphoma Computerised tomogram breast abnormal Computerised tomogram liver abnormal Congenital acrochordon Congenital benign neoplasm Congenital cerebral cyst Congenital cerebral haemangioma Congenital choroid plexus cyst Congenital cyst Congenital cystic disease of liver Congenital cystic kidney disease Congenital eye naevus Congenital fibrosarcoma Congenital malignant neoplasm Congenital melanocytic naevus Congenital naevus Congenital neoplasm Congenital renal cyst Congenital retinoblastoma Congenital teratoma Congenital vaginal cyst Conjunctival cyst
Conjunctival melanoma Conjunctival neoplasm Conjunctival primary acquired melanosis Connective tissue neoplasm Corneal cyst
Corneoconjunctival intraepithelial neoplasia
Cowden's disease
Cranial nerve neoplasm benign Craniopharyngioma Craniopharyngioma benign Crohn's disease Cronkhite-Canada syndrome Cutaneous T-cell dyscrasia Cutaneous lymphoma Cyclotron therapy Cyst Cyst rupture Cystadenocarcinoma ovary Cystadenocarcinoma pancreas Cystadenofibroma of fallopian tube Cystic angiomatosis Cystic eyeball, congenital Cystic lymphangioma Cystoprostatectomy Cytokeratin 18 increased Dedifferentiated liposarcoma Dental cyst Denys-Drash syndrome Dermal cyst Dermatofibrosarcoma protuberans Dermatofibrosarcoma protuberans metastatic Dermoid cyst Desmoid tumour Desmoplastic melanoma Desmoplastic mesothelioma Desmoplastic small round cell tumour Diaphragm neoplasm


Final 92 of 152

 ${\tt Pre-defined} \ {\tt MedDRA} \ {\tt search} \ {\tt -list} \ {\tt of} \ {\tt preferred} \ {\tt terms}$ 

Pre-defined MedDRA search Preferred term Neoplasm Differentiation syndrome Diffuse large B-cell lymphoma Diffuse large B-cell lymphoma recurrent Diffuse large B-cell lymphoma refractory Diffuse large B-cell lymphoma stage I Diffuse large B-cell lymphoma stage II Diffuse large B-cell lymphoma stage III Diffuse large B-cell lymphoma stage IV Diffuse uveal melanocytic proliferation Disseminated large cell lymphoma Double hit lymphoma Ductal adenocarcinoma of pancreas Duodenal neoplasm Duodenal polyp Duodenectomy Dysplasia Dysplastic naevus Dysplastic naevus syndrome Ear neoplasm Ear neoplasm malignant Eastern Cooperative Oncology Group performance status Eastern Cooperative Oncology Group performance status worsened Eccrine carcinoma Ectopic ACTH syndrome Ectopic aldosterone secretion Ectopic antidiuretic hormone secretion Ectopic calcitonin production Ectopic chorionic gonadotrophin secretion Ectopic growth hormone secretion Ectopic hormone secretion Ectopic parathyroid hormone production Ectopic prolactin secretion Ectopic renin secretion Elastofibroma Electron radiation therapy Electron radiation therapy to bladder Electron radiation therapy to blood Electron radiation therapy to bone Electron radiation therapy to brain Electron radiation therapy to breast Electron radiation therapy to colon Electron radiation therapy to ear, nose, or throat Electron radiation therapy to liver Electron radiation therapy to lung Electron radiation therapy to pancreas Electron radiation therapy to prostate Electron radiation therapy to skin
Electron radiation therapy to soft tissue Electron radiation therapy to uterus Elephantiasis nostras verrucosa Embryonal rhabdomyosarcoma Encephalitis autoimmune Enchondromatosis Endobronchial lipoma Endocrine neoplasm Endocrine neoplasm malignant Endometrial adenocarcinoma Endometrial adenoma Endometrial cancer Endometrial cancer metastatic Endometrial cancer recurrent


 Date:
 03 July 2019

 Version:
 1.0

 Status:
 Final

 Page:

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Neoplasm Endometrial cancer stage 0 Endometrial cancer stage I Endometrial cancer stage II Endometrial cancer stage III Endometrial cancer stage IV Endometrial dysplasia Endometrial hyperplasia Endometrial neoplasm Endometrial sarcoma Endometrial sarcoma metastatic Endometrial sarcoma recurrent Endometrial stromal sarcoma Endotheliomatosis Enteropathy-associated T-cell lymphoma Eosinophilic leukaemia Ependymoma Ependymoma benign Ependymoma malignant Epidermal naevus syndrome Epidermodysplasia verruciformis Epididymal cancer Epididymal cyst Epididymal neoplasm Epiglottic carcinoma Epiglottic cyst Epiglottic mass Epiglottidectomy Epithelioid mesothelioma Epithelioid sarcoma Epithelioid sarcoma metastatic Epithelioid sarcoma recurrent Epithelioma adenoides cysticum Epstein Barr virus positive mucocutaneous ulcer Epstein-Barr virus associated lymphoma Epstein-Barr virus associated lymphoproliferative disorder Epulis Erdheim-Chester disease Erythraemic myelosis (in remission) Erythroleukaemia Erythroplasia Erythroplasia of lip Erythroplasia of penis Erythroplasia of vulva Essential thrombocythaemia Ewing's sarcoma Ewing's sarcoma metastatic Ewing's sarcoma recurrent Ewing-like sarcoma Ex vivo gene therapy Exploratory operation Extended radical mastectomy Extra-osseous Ewing's sarcoma
Extra-osseous Ewing's sarcoma metastatic Extra-osseous Ewing's sarcoma recurrent Extradural neoplasm Extragonadal primary embryonal carcinoma Extragonadal primary embryonal carchoma
Extragonadal primary germ cell tumour
Extragonadal primary germ cell tumour mixed
Extragonadal primary germ cell tumour mixed stage I
Extragonadal primary germ cell tumour mixed stage II
Extragonadal primary germ cell tumour mixed stage III
Extragonadal primary malignant teratoma Extragonadal primary non-seminoma


 Date:
 03 July 2019

 Version:
 1.0

 Status:
 Final

 Page:

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

```
Pre-defined MedDRA search
                                                       Preferred term
Neoplasm
                                                       Extragonadal primary non-seminoma stage I
                                                       Extragonadal primary non-seminoma stage II
                                                       Extragonadal primary non-seminoma stage III
                                                       Extragonadal primary non-seminoma stage IV
Extragonadal primary seminoma (pure)
Extragonadal primary seminoma (pure) stage I
Extragonadal primary seminoma (pure) stage II
Extragonadal primary seminoma (pure) stage II
Extragonadal primary seminoma (pure) stage III
                                                       Extragonadal primary seminoma (pure) stage IV Extramammary Paget's disease
                                                       Extranodal marginal zone B-cell lymphoma (BALT type)
Extranodal marginal zone B-cell lymphoma (MALT type)
Extranodal marginal zone B-cell lymphoma (MALT type)
                                                       recurrent
                                                       Extranodal marginal zone B-cell lymphoma (MALT type)
                                                       refractory
                                                       Extranodal marginal zone B-cell lymphoma (MALT type) stage I Extranodal marginal zone B-cell lymphoma (MALT type) stage
                                                       Extranodal marginal zone B-cell lymphoma (MALT type) stage
                                                       Extranodal marginal zone B-cell lymphoma (MALT type) stage
                                                       Extraocular retinoblastoma
                                                       Extraskeletal chondrosarcoma metastatic Extraskeletal chondrosarcoma recurrent
                                                       Extraskeletal myxoid chondrosarcoma
                                                       Extraskeletal osteosarcoma
                                                       Extraskeletal osteosarcoma metastatic
                                                       Extraskeletal osteosarcoma recurrent
                                                       Eye haemangioma
                                                       Eve naevus
                                                       Evelid haemangioma
                                                       Eyelid naevus
                                                       Eyelid tumour
                                                       Fallopian tube cancer
                                                       Fallopian tube cancer metastatic
                                                       Fallopian tube cancer stage I
                                                       Fallopian tube cancer stage II
                                                       Fallopian tube cancer stage III
                                                       Fallopian tube cancer stage IV
                                                       Fallopian tube cyst
                                                       Fallopian tube leiomyoma
                                                       Fallopian tube neoplasm
                                                       Familial acromegaly
Familial gigantiform cementoma
                                                       Familial haemophagocytic lymphohistiocytosis
                                                       Familial medullary thyroid cancer
Familial multiple lipomatosis
                                                       Female reproductive neoplasm
                                                       Female reproductive tract carcinoma in situ
                                                       Fibroadenoma of breast
Fibrocystic breast disease
                                                       Fibroma
                                                       Fibromatosis
                                                       Fibrosarcoma
                                                       Fibrosarcoma excision
                                                       Fibrosarcoma metastatic
                                                       Fibrous cortical defect
                                                       Fibrous histiocytoma
                                                       Fiducial marker placement
Fms-like tyrosine kinase 3 positive
                                                       Focal nodular hyperplasia
```


 Date:
 03 July 2019

 Version:
 1.0

 Status:
 Final

 Page:

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Neoplasm Foetal cystic hygroma Follicle centre lymphoma diffuse small cell lymphoma Follicle centre lymphoma diffuse small cell lymphoma recurrent. Follicle centre lymphoma diffuse small cell lymphoma refractory Follicle centre lymphoma diffuse small cell lymphoma stage I Follicle centre lymphoma diffuse small cell lymphoma stage Follicle centre lymphoma diffuse small cell lymphoma stage TTT Follicle centre lymphoma diffuse small cell lymphoma stage Follicle centre lymphoma, follicular grade I, II, III Follicle centre lymphoma, follicular grade I, II, III recurrent Follicle centre lymphoma, follicular grade I, II, III refractory
Follicle centre lymphoma, follicular grade I, II, III stage Follicle centre lymphoma, follicular grade I, II, III stage Follicle centre lymphoma, follicular grade I, II, III stage Follicle centre lymphoma, follicular grade I, II, III stage Follicular dendritic cell sarcoma Follicular thyroid cancer Frasier syndrome Free prostate-specific antigen increased Free prostate-specific antigen positive Fungating wound Gallbladder adenocarcinoma Gallbladder adenoma Gallbladder adenosquamous carcinoma Gallbladder cancer Gallbladder cancer metastatic Gallbladder cancer recurrent Gallbladder cancer stage 0 Gallbladder cancer stage I Gallbladder cancer stage II Gallbladder cancer stage III Gallbladder cancer stage IV Gallbladder neoplasm Gallbladder papilloma Gallbladder polyp Gallbladder squamous cell carcinoma Gamma interferon therapy Gamma radiation therapy Gamma radiation therapy to bladder Gamma radiation therapy to blood Gamma radiation therapy to bone Gamma radiation therapy to brain Gamma radiation therapy to breast Gamma radiation therapy to colon Gamma radiation therapy to ear, nose, or throat Gamma radiation therapy to liver Gamma radiation therapy to lung Gamma radiation therapy to pancreas Gamma radiation therapy to pleura Gamma radiation therapy to prostate Gamma radiation therapy to skin Gamma radiation therapy to soft tissue


Date: Version: Status: Page: 03 July 2019 1.0 Final


Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Gamma radiation therapy to thyroid Neoplasm Gamma radiation therapy to uterus Gammopathy Ganglioglioma Ganglioneuroblastoma Ganglioneuroma Garcin syndrome Gastrectomy Gastric adenoma Gastric cancer Gastric cancer recurrent Gastric cancer stage 0 Gastric cancer stage I Gastric cancer stage II Gastric cancer stage III Gastric cancer stage IV Gastric cyst Gastric dysplasia Gastric haemangioma Gastric leiomyoma Gastric neoplasm Gastric polypectomy Gastric polyps Gastric sarcoma Gastric stent insertion Gastrinoma Gastrinoma malignant Gastroenteropancreatic neuroendocrine tumour disease Gastrointestinal adenocarcinoma Gastrointestinal cancer metastatic Gastrointestinal carcinoma Gastrointestinal carcinoma in situ Gastrointestinal dysplasia Gastrointestinal lymphoma Gastrointestinal melanoma Gastrointestinal neoplasm Gastrointestinal polyp Gastrointestinal polyp haemorrhage Gastrointestinal stromal cancer Gastrointestinal stromal tumour Gastrointestinal submucosal tumour Gastrointestinal tract adenoma Gastrooesophageal cancer Gastrooesophageal cancer recurrent Genital cancer male Genital cancer male in situ Genital cyst Genital neoplasm malignant female Genitourinary melanoma Genitourinary tract neoplasm Germ cell cancer Germ cell cancer metastatic Germ cell neoplasm Gestational trophoblastic tumour Giant cell epulis Giant cell tumour of tendon sheath Gingival cancer Gingival cyst Gingival polyp Glioblastoma Glioblastoma multiforme Glioma

Gliomatosis cerebri


Page:

Novo Nordisk

1.0

Final


Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Neoplasm Glioneuronal tumour Gliosarcoma Glomus jugulare tumour Glomus tumour Glomus tympanicum tumour Glossectomy Glottis carcinoma Glucagonoma Good syndrome Gorham's disease Granular cell tumour Granulosa cell tumour of the testis Growth hormone-producing pituitary tumour HER-2 positive breast cancer HER-2 positive gastric cancer Haemangioblastoma Haemangioma Haemangioma congenital Haemangioma of bone Haemangioma of breast Haemangioma of liver Haemangioma of retina Haemangioma of skin Haemangioma of spleen Haemangioma-thrombocytopenia syndrome Haemangiopericytoma Haemangiopericytoma of meninges Haematological malignancy Haematopoietic neoplasm Haemophagocytic lymphohistiocytosis Haemophilic pseudotumour Haemorrhagic breast cyst Haemorrhagic cyst Haemorrhagic hepatic cyst Haemorrhagic ovarian cyst Haemorrhagic thyroid cyst Haemorrhagic tumour necrosis Hair follicle tumour benign
Hairy cell leukaemia
Hairy cell leukaemia recurrent
Hamartoma Hamartoma vascular Head and neck cancer Head and neck cancer metastatic Head and neck cancer stage I Head and neck cancer stage II Head and neck cancer stage III Head and neck cancer stage IV Heavy chain disease Hemicorporectomy Hemipelvectomy Hepatectomy Hepatic adenoma Hepatic angiosarcoma Hepatic cancer Hepatic cancer metastatic Hepatic cancer recurrent Hepatic cancer stage I Hepatic cancer stage II Hepatic cancer stage III Hepatic cancer stage IV Hepatic cyst

Hepatic cyst infection


Date: Version: Status: Page: 03 July 2019 1.0 Final 98 of 152

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Neoplasm Hepatic cyst ruptured Hepatic haemangioma rupture Hepatic hamartoma Hepatic neoplasm Hepatobiliary cancer Hepatobiliary cancer in situ Hepatobiliary cyst Hepatobiliary neoplasm Hepatoblastoma Hepatoblastoma recurrent Hepatocellular carcinoma Hepatosplenic T-cell lymphoma Hereditary leiomyomatosis renal cell carcinoma Hereditary multiple osteochondromas Hereditary non-polyposis colorectal cancer syndrome Hereditary papillary renal carcinoma Hidradenocarcinoma High frequency ablation High grade B-cell lymphoma Burkitt-like lymphoma High grade B-cell lymphoma Burkitt-like lymphoma recurrent High grade B-cell lymphoma Burkitt-like lymphoma refractory High grade B-cell lymphoma Burkitt-like lymphoma stage I High grade B-cell lymphoma Burkitt-like lymphoma stage II High grade B-cell lymphoma Burkitt-like lymphoma stage II High grade B-cell lymphoma Burkitt-like lymphoma stage IV High intensity focused ultrasound High-grade B-cell lymphoma lymphoma stage III Histiocytic medullary reticulosis Histiocytic necrotising lymphadenitis Histiocytic sarcoma Histiocytosis Hodgkin's disease Hodgkin's disease lymphocyte depletion stage I site unspecified Hodgkin's disease lymphocyte depletion stage I subdiaphragm Hodgkin's disease lymphocyte depletion stage I supradiaphragm Hodgkin's disease lymphocyte depletion stage II site unspecified Hodgkin's disease lymphocyte depletion stage II subdiaphragm Hodgkin's disease lymphocyte depletion stage II supradiaphragm Hodgkin's disease lymphocyte depletion type recurrent Hodgkin's disease lymphocyte depletion type refractory Hodgkin's disease lymphocyte depletion type stage III Hodgkin's disease lymphocyte depletion type stage IV Hodgkin's disease lymphocyte depletion type stage unspecified Hodgkin's disease lymphocyte predominance stage I site unspec Hodgkin's disease lymphocyte predominance stage I subdiaphragm Hodgkin's disease lymphocyte predominance stage I supradiaphragm Hodgkin's disease lymphocyte predominance stage II site Hodgkin's disease lymphocyte predominance stage II subdiaphragm Hodgkin's disease lymphocyte predominance stage II supradiaphragm Hodgkin's disease lymphocyte predominance type recurrent Hodgkin's disease lymphocyte predominance type refractory Hodgkin's disease lymphocyte predominance type stage III


Final 99 of 152

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Hodgkin's disease lymphocyte predominance type stage IV Neoplasm Hodgkin's disease lymphocyte predominance type stage unspecified Hodgkin's disease mixed cellularity recurrent Hodgkin's disease mixed cellularity refractory Hodgkin's disease mixed cellularity stage I site unspecified Hodgkin's disease mixed cellularity stage I subdiaphragmatic Hodgkin's disease mixed cellularity stage I supradiaphragmatic Hodgkin's disease mixed cellularity stage II subdiaphragmatic Hodgkin's disease mixed cellularity stage II supradiaphragmatic Hodgkin's disease mixed cellularity stage III Hodgkin's disease mixed cellularity stage IV Hodgkin's disease mixed cellularity stage unspecified Hodgkin's disease nodular sclerosis Hodgkin's disease nodular sclerosis recurrent Hodgkin's disease nodular sclerosis refractory Hodgkin's disease nodular sclerosis stage I Hodgkin's disease nodular sclerosis stage II Hodgkin's disease nodular sclerosis stage III Hodgkin's disease nodular sclerosis stage IV Hodgkin's disease recurrent Hodgkin's disease refractory Hodgkin's disease stage I Hodgkin's disease stage II Hodgkin's disease stage III Hodgkin's disease stage IV Hodgkin's disease unclassifiable Hormone refractory breast cancer Hormone suppression therapy Hormone therapy Hormone-dependent prostate cancer Hormone-refractory prostate cancer Hormone-secreting ovarian tumour Horner's syndrome Huerthle cell carcinoma
Human chorionic gonadotropin increased
Human chorionic gonadotropin positive
Human epidermal growth factor receptor increased Hygroma colli Hypercalcaemia of malignancy Hypercalcitoninaemia Hypergammaglobulinaemia benign monoclonal Hyperleukocytosis Hyperreactio luteinalis Hyperthermia therapy Hyperthermic chemotherapy Hypertrophic osteoarthropathy Hypopharyngeal cancer Hypopharyngeal cancer recurrent Hypopharyngeal cancer stage 0 Hypopharyngeal cancer stage I Hypopharyngeal cancer stage II Hypopharyngeal cancer stage III Hypopharyngeal cancer stage IV Hypopharyngeal neoplasm Hypopharyngeal neoplasm benign Hypophosphataemic osteomalacia Hypophysectomy Hypothalamic hamartoma Hysterectomy


 Date:
 03 July 2019

 Version:
 1.0

 Status:
 Final

Page:

Final 100 of 152

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Neoplasm Hysterosalpingectomy Hysterosalpingo-oophorectomy Ileectomy Ileocolectomy Imaging procedure abnormal Immune enhancement therapy Immune reconstitution inflammatory syndrome associated Kaposi's sarcoma Immunoblastic lymphoma Immunochemotherapy Immunoglobulin clonality assay Implant site cyst In vivo gene therapy Infantile fibromatosis Infantile haemangioma Infantile septic granulomatosis Infected cyst Infected dermal cyst Infected lymphocele Infected naevus Infected neoplasm Inferior vena cava syndrome Inflammatory carcinoma of breast recurrent Inflammatory carcinoma of breast stage III Inflammatory carcinoma of breast stage IV Inflammatory carcinoma of the breast Inflammatory malignant fibrous histiocytoma Inflammatory myofibroblastic tumour Inflammatory pseudotumour Infusion site cyst Injection site cyst Insulinoma Interleukin therapy Intestinal T-cell lymphoma recurrent Intestinal T-cell lymphoma refractory Intestinal T-cell lymphoma stage I Intestinal T-cell lymphoma stage II Intestinal T-cell lymphoma stage III Intestinal T-cell lymphoma stage IV Intestinal adenocarcinoma Intestinal angioma Intestinal cyst Intestinal metastasis Intestinal polyp
Intestinal polypectomy
Intestinal resection Intra-abdominal haemangioma Intracranial germ cell tumour Intracranial haemangioma Intracranial meningioma malignant Intracranial tumour haemorrhage Intracystic breast papilloma
Intraductal papillary breast neoplasm
Intraductal papillary mucinous neoplasm
Intraductal papillary-mucinous carcinoma of pancreas Intraductal papilloma of breast Intraductal proliferative breast lesion Intraneural cyst Intraocular melanoma Intraosseous angioma Intratumoural aneurysm Intravascular lipoma

Intravascular papillary endothelial hyperplasia


1.0 Final 101 of 152 Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Leiomyoma Leiomyosarcoma

Intravenous leiomyomatosis

Neoplasm

Intravesical immunotherapy Invasive breast carcinoma
Invasive ductal breast carcinoma
Invasive lobular breast carcinoma Invasive papillary breast carcinoma Iris cyst Iris hamartoma Iris melanoma Iris neoplasm Trreversible electroporation
Isocitrate dehydrogenase gene mutation Jaw cyst Jejunectomy Joint neoplasm Juvenile angiofibroma Juvenile chronic myelomonocytic leukaemia Juvenile melanoma benign Kaposi's sarcoma
Kaposi's sarcoma AIDS related Kaposi's sarcoma classical type Keratinising squamous cell carcinoma of nasopharynx Keratoacanthoma Kidney angiomyolipoma Knuckle pads Lacrimal cyst Lacrimal duct neoplasm Langerhans cell sarcoma Langerhans' cell histiocytosis Large cell lung cancer Large cell lung cancer metastatic Large cell lung cancer recurrent Large cell lung cancer stage 0 Large cell lung cancer stage I Large cell lung cancer stage Large cell lung cancer stage III Large cell lung cancer stage IV Large granular lymphocytosis Large intestinal polypectomy Large intestine benign neoplasm Large intestine fibroma Large intestine polyp Laryngeal cancer Laryngeal cancer metastatic Laryngeal cancer recurrent Laryngeal cancer stage 0 Laryngeal cancer stage I Laryngeal cancer stage II Laryngeal cancer stage III Laryngeal cancer stage IV Laryngeal cyst Laryngeal dysplasia Laryngeal leukoplakia Laryngeal neoplasm Laryngeal papilloma Laryngeal polyp Laryngeal polypectomy Laryngeal squamous cell carcinoma Laryngectomy Laryngopharyngectomy Laser brain ablation


1.0 Final 102 of 152 Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Liposarcoma recurrent

Neoplasm

```
Leiomyosarcoma metastatic
Leiomyosarcoma recurrent
Lentigo maligna
Lentigo maligna recurrent
Lentigo maligna stage I
Lentigo maligna stage II
Lentigo maligna stage III
Lentigo maligna stage IV
Leptomeningeal myelomatosis
Leser-Trelat sign
Leukaemia
Leukaemia basophilic
Leukaemia cutis
Leukaemia granulocytic
Leukaemia in remission
Leukaemia monocytic
Leukaemia recurrent
Leukaemic cardiac infiltration Leukaemic infiltration
Leukaemic infiltration extramedullary
Leukaemic infiltration gingiva
Leukaemic infiltration hepatic
Leukaemic infiltration ovary
Leukaemic infiltration pulmonary
Leukaemic infiltration renal
Leukaemic lymphoma
Leukaemic retinopathy
Leukoerythroblastosis
Leukoplakia
Leukoplakia oesophageal
Leukoplakia of penis
Leukoplakia oral
Leukostasis syndrome
Leydig cell tumour of the testis
Light chain disease
Limbic encephalitis
Linitis plastica
Lip and or oral cavity cancer
Lip and
or oral cavity cancer recurrent
Lip and
or oral cavity cancer stage 0
Lip and
or oral cavity cancer stage I
Lip and
or oral cavity cancer stage II
Lip and
or oral cavity cancer stage III
Lip and
or oral cavity cancer stage IV
Lip neoplasm Lip neoplasm benign
Lip neoplasm malignant stage unspecified Lip squamous cell carcinoma
Lipoblastoma
Lipodermoid tumour
Lipofibroma
Lipoma
Lipoma of breast
Liposarcoma
Liposarcoma metastatic
```


Date: Version: Status: Page: 03 July 2019 1.0 Final 103 of 152

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Neoplasm Liver ablation Liver carcinoma ruptured Liver scan abnormal Lobular breast carcinoma in situ Lung adenocarcinoma Lung adenocarcinoma recurrent Lung adenocarcinoma stage 0 Lung adenocarcinoma stage I Lung adenocarcinoma stage Lung adenocarcinoma stage III Lung adenocarcinoma stage IV Lung cancer metastatic Lung carcinoma cell type unspecified recurrent Lung carcinoma cell type unspecified stage 0 Lung carcinoma cell type unspecified stage I Lung carcinoma cell type unspecified stage II Lung carcinoma cell type unspecified stage III Lung carcinoma cell type unspecified stage IV Lung cyst Lung infiltration malignant Lung lobectomy Lung neoplasm Lung neoplasm malignant Lung neoplasm surgery
Lung squamous cell carcinoma metastatic
Lung squamous cell carcinoma recurrent
Lung squamous cell carcinoma stage 0 Lung squamous cell carcinoma stage I Lung squamous cell carcinoma stage II Lung squamous cell carcinoma stage III Lung squamous cell carcinoma stage IV Lymph nodes scan abnormal Lymphadenectomy Lymphangioma Lymphangiosarcoma Lymphangiosis carcinomatosa Lymphatic mapping Lymphatic system neoplasm Lymphocele Lymphocyte adoptive therapy Lymphocyte morphology abnormal Lymphocytic leukaemia Lymphocytic lymphoma Lymphoid leukaemia (in remission) Lymphoid tissue operation Lymphoma Lymphoma AIDS related Lymphoma operation Lymphoma transformation Lymphoplasmacytoid lymphoma immunocytoma Lymphoplasmacytoid lymphoma immunocytoma recurrent Lymphoplasmacytoid lymphoma immunocytoma refractory Lymphoplasmacytoid lymphoma immunocytoma stage I Lymphoplasmacytoid lymphoma immunocytoma stage II Lymphoplasmacytoid lymphoma immunocytoma stage III Lymphoplasmacytoid lymphoma immunocytoma stage IV


03 July 2019 Date: Version: Status: Page:

1.0 Final 104 of 152 Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Neoplasm Lymphoproliferative disorder Lymphoproliferative disorder in remission Male reproductive tract neoplasm Malignant anorectal neoplasm Malignant ascites Malignant biliary obstruction Malignant blue naevus Malignant connective tissue neoplasm Malignant cranial nerve neoplasm Malignant dysphagia Malignant exophthalmos Malignant fibrous histiocytoma Malignant fibrous histiocytoma metastatic Malignant fibrous histiocytoma of bone Malignant fibrous histiocytoma recurrent Malignant gastrointestinal obstruction Malignant genitourinary tract neoplasm Malignant giant cell fibrous histiocytoma Malignant glioma Malignant haemangiopericytoma Malignant haemangiopericytoma metastatic Malignant haemangiopericytoma recurrent Malignant histiocytosis Malignant hydatidiform mole Malignant joint neoplasm
Malignant lymphoid neoplasm
Malignant lymphoma unclassifiable high grade Malignant lymphoma unclassifiable low grade Malignant mast cell neoplasm Malignant mediastinal neoplasm Malignant melanoma Malignant melanoma in situ Malignant melanoma of eyelid Malignant melanoma of sites other than skin Malignant melanoma stage I Malignant melanoma stage II Malignant melanoma stage III Malignant melanoma stage IV Malignant meningioma metastatic Malignant mesenchymoma Malignant mesenchymoma metastatic Malignant mesenchymoma recurrent Malignant mesenteric neoplasm Malignant middle ear neoplasm Malignant muscle neoplasm Malignant neoplasm of ampulla of Vater Malignant neoplasm of auricular cartilage Malignant neoplasm of choroid Malignant neoplasm of conjunctiva Malignant neoplasm of cornea Malignant neoplasm of eye
Malignant neoplasm of eyelid
Malignant neoplasm of islets of Langerhans Malignant neoplasm of lacrimal duct Malignant neoplasm of lacrimal gland Malignant neoplasm of orbit Malignant neoplasm of paraurethral glands Malignant neoplasm of placenta Malignant neoplasm of pleura Malignant neoplasm of pleura metastatic Malignant neoplasm of renal pelvis Malignant neoplasm of retina

Malignant neoplasm of seminal vesicle


Final

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Neoplasm Malignant neoplasm of spermatic cord Malignant neoplasm of spinal cord Malignant neoplasm of thorax
Malignant neoplasm of thymus
Malignant neoplasm of unknown primary site
Malignant neoplasm of uterine adnexa Malignant neoplasm papilla of Vater Malignant neoplasm progression Malignant nervous system neoplasm Malignant nipple neoplasm Malignant nipple neoplasm female Malignant nipple neoplasm male Malignant oligodendroglioma Malignant ovarian cyst Malignant palate neoplasm Malignant pericardial neoplasm Malignant peritoneal neoplasm Malignant pituitary tumour Malignant pleural effusion Malignant polyp Malignant psoas syndrome Malignant respiratory tract neoplasm Malignant splenic neoplasm Malignant sweat gland neoplasm Malignant transformation Malignant urinary tract neoplasm
Malignant urinary tract obstruction Mantíe cell lymphoma Mantle cell lymphoma recurrent Mantle cell lymphoma refractory Mantle cell lymphoma stage I Mantle cell lymphoma stage II Mantle cell lymphoma stage III Mantle cell lymphoma stage IV Marginal zone lymphoma Marginal zone lymphoma recurrent Marginal zone lymphoma refractory Marginal zone lymphoma stage I Marginal zone lymphoma stage II Marginal zone lymphoma stage III Marginal zone lymphoma stage IV Marjolin's ulcer Marrow hyperplasia Mastectomy Mastocytic leukaemia Mastocytoma Mastoid cyst Mastoidectomy Maternal cancer in pregnancy Mature B-cell type acute leukaemia Maxillofacial sinus neoplasm Mazabraud's syndrome Mediastinal biopsy abnormal Mediastinal cyst Mediastinum neoplasm Medical device site cyst Medullary carcinoma of breast Medullary thyroid cancer Medulloblastoma Medulloblastoma recurrent Megaloblasts increased Meigs' syndrome

Melanocytic naevus


2019 Novo Nordisk 1.0 Final

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Melanoma recurrent

Metastases to skin Metastases to soft tissue

Neoplasm

Melanoplakia oral Meningeal neoplasm Meningioma Meningioma benign Meningioma malignant Meniscus cyst Mesenteric cyst Mesenteric neoplasm Mesoblastic nephroma Mesonephric duct cyst Mesothelioma Mesothelioma malignant Mesothelioma malignant recurrent Metaplastic breast carcinoma Metastases to Eustachian tube Metastases to abdominal cavity Metastases to abdominal wall Metastases to adrenals Metastases to biliary tract Metastases to bladder Metastases to bone Metastases to bone marrow Metastases to breast Metastases to central nervous system Metastases to chest wall Metastases to diaphragm Metastases to eye Metastases to fallopian tube Metastases to gallbladder Metastases to gastrointestinal tract Metastases to heart Metastases to kidnev Metastases to larynx Metastases to liver Metastases to lung Metastases to lymph nodes Metastases to meninges Metastases to mouth Metastases to muscle Metastases to nasal sinuses Metastases to neck Metastases to nervous system Metastases to oesophagus Metastases to ovary Metastases to pancreas Metastases to pelvis Metastases to penis Metastases to perineum Metastases to peripheral nervous system Metastases to peripheral vascular system Metastases to peritoneum Metastases to pharynx Metastases to pituitary gland Metastases to placenta Metastases to pleura Metastases to prostate Metastases to rectum Metastases to reproductive organ Metastases to retroperitoneum Metastases to salivary gland


Page:

Final 107 of 152

1.0

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Neoplasm Metastases to spinal cord Metastases to spine Metastases to spleen Metastases to stomach Metastases to testicle Metastases to the mediastinum Metastases to the respiratory system Metastases to thorax Metastases to thyroid Metastases to tonsils Metastases to trachea Metastases to urinary tract Metastases to uterus Metastases to vagina Metastasis Metastatic bronchial carcinoma Metastatic carcinoid tumour Metastatic carcinoma of the bladder Metastatic choriocarcinoma Metastatic gastric cancer Metastatic glioma Metastatic glucagonoma Metastatic lymphoma Metastatic malignant melanoma Metastatic neoplasm Metastatic nervous system neoplasm Metastatic ocular melanoma Metastatic pulmonary embolism Metastatic renal cell carcinoma Metastatic salivary gland cancer Metastatic squamous cell carcinoma Metastatic uterine cancer Micrographic skin surgery Microsatellite instability cancer Minimal residual disease Mismatch repair cancer syndrome Mixed adenoneuroendocrine carcinoma Mixed hepatocellular cholangiocarcinoma Mixed-type liposarcoma Modified radical mastectomy Monoclonal gammopathy Monocytic leukaemia in remission Mouth cyst Mucinous adenocarcinoma of appendix Mucinous breast carcinoma Mucinous cystadenocarcinoma ovary Mucinous endometrial carcinoma Mucoepidermoid carcinoma Mucoepidermoid carcinoma of salivary gland Mucosal cyst of postmastoidectomy cavity Mueller's mixed tumour Muir-Torre syndrome Multicentric reticulohistiocytosis Multinucleate cell angiohistiocytoma Multiple cutaneous and uterine leiomyomatosis Multiple endocrine neoplasia Multiple endocrine neoplasia Type 1
Multiple endocrine neoplasia Type 2
Multiple endocrine neoplasia Type 2A
Multiple endocrine neoplasia Type 2A
Multiple endocrine neoplasia Type 2B
Multiple gated acquisition scan abnormal Muscle neoplasm

Musculoskeletal cancer


Date: 03 July 2019 Version: 1.0 Status: Final

Page:

Final 108 of 152

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Neoplasm Myasthenic syndrome Mycosis fungoides Mycosis fungoides recurrent Mycosis fungoides refractory Mycosis fungoides stage I Mycosis fungoides stage II Mycosis fungoides stage III Mycosis fungoides stage IV Myectomy Myeloblast present Myeloblastoma Myelodysplastic syndrome Myelodysplastic syndrome transformation Myelodysplastic syndrome unclassifiable Myelofibrosis Myeloid leukaemia Myeloid leukaemia in remission Myeloid metaplasia Myelolipoma
Myeloma cast nephropathy Myeloproliferative neoplasm Myolipoma Myxofibrosarcoma Myxoid liposarcoma NMP22 test abnormal NUT midline carcinoma Naevoid melanoma Naevus haemorrhage Naevus lipomatosus cutaneous superficialis Nasal cavity cancer Nasal cyst Nasal neoplasm Nasal neoplasm benign Nasal polyps Nasal sinus cancer Nasopharyngeal cancer Nasopharyngeal cancer metastatic Nasopharyngeal cancer recurrent Nasopharyngeal cancer stage 0 Nasopharyngeal cancer stage I Nasopharyngeal cancer stage II Nasopharyngeal cancer stage III Nasopharyngeal cancer stage IV Nasopharyngeal neoplasm benign Nasopharyngeal polyp Natural killer-cell leukaemia Natural killer-cell lymphoblastic lymphoma Neck dissection Necrolytic migratory erythema Needle biopsy site unspecified abnormal Neoadjuvant therapy Neobladder surgery Neonatal leukaemia Neonatal neuroblastoma Neoplasm Neoplasm malignant Neoplasm of appendix Neoplasm of cornea unspecified malignancy Neoplasm of orbit Neoplasm of thymus Neoplasm progression Neoplasm prostate

Neoplasm recurrence


Novo Nordisk

1.0

Final

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term

Neoplasm

Neoplasm skin Neoplasm swelling Nephrectomy Nephroblastoma Nephroureterectomy Nervous system cyst Nervous system neoplasm Nervous system neoplasm benign Nervous system neoplasm surgery Neurilemmoma benign Neuroblastoma Neuroblastoma recurrent Neuroectodermal neoplasm Neuroendocrine breast tumour Neuroendocrine carcinoma Neuroendocrine carcinoma metastatic Neuroendocrine carcinoma of the bladder Neuroendocrine carcinoma of the skin Neuroendocrine tumour Neuroendocrine tumour of the lung Neuroendocrine tumour of the lung metastatic Neuroendoscopy Neurofibroma Neurofibromatosis Neurofibrosarcoma Neurofibrosarcoma metastatic Neurofibrosarcoma recurrent Neurogenic tumour Neuroma Neuromyotonia Neurotensinoma Nipple neoplasm Nipple resection Nodal marginal zone B-cell lymphoma Nodal marginal zone B-cell lymphoma recurrent Nodal marginal zone B-cell lymphoma refractory Nodal marginal zone B-cell lymphoma stage I Nodal marginal zone B-cell lymphoma stage II Nodal marginal zone B-cell lymphoma stage III Nodal marginal zone B-cell lymphoma stage IV Nodular fasciitis Nodular lymphocyte predominant Hodgkin lymphoma Nodular melanoma Non-Hodgkin's lymphoma Non-Hodgkin's lymphoma metastatic Non-Hodgkin's lymphoma recurrent Non-Hodgkin's lymphoma refractory Non-Hodgkin's lymphoma stage I Non-Hodgkin's lymphoma stage II Non-Hodgkin's lymphoma stage III Non-Hodgkin's lymphoma stage IV Non-Hodgkin's lymphoma transformed recurrent Non-Hodgkin's lymphoma unspecified histology aggressive Non-Hodgkin's lymphoma unspecified histology aggressive recurrent Non-Hodgkin's lymphoma unspecified histology aggressive refractory Non-Hodgkin's lymphoma unspecified histology aggressive stage T Non-Hodgkin's lymphoma unspecified histology aggressive Non-Hodgkin's lymphoma unspecified histology aggressive stage III


Date: Version: Status: Page: 03 July 2019 | Novo Nordisk 1.0 Final 110 of 152

 ${\tt Pre-defined\ MedDRA\ search\ -\ list\ of\ preferred\ terms}$ 

Pre-defined MedDRA search Preferred term Non-Hodgkin's lymphoma unspecified histology aggressive Neoplasm Non-Hodgkin's lymphoma unspecified histology indolent Non-Hodgkin's lymphoma unspecified histology indolent stage Non-Hodgkin's lymphoma unspecified histology indolent stage Non-Hodgkin's lymphoma unspecified histology indolent stage Non-Hodgkin's lymphoma unspecified histology indolent stage Non-renal cell carcinoma of kidney Non-secretory adenoma of pituitary Non-small cell lung cancer Non-small cell lung cancer metastatic Non-small cell lung cancer recurrent Non-small cell lung cancer stage 0 Non-small cell lung cancer stage I Non-small cell lung cancer stage II Non-small cell lung cancer stage III Non-small cell lung cancer stage IIIA Non-small cell lung cancer stage IIIB Non-small cell lung cancer stage IV Nongerminomatous germ cell tumour of the CNS Nonkeratinising carcinoma of nasopharynx Numb chin syndrome Ocular cancer metastatic Ocular haemangiopericytoma Ocular lymphoma Ocular neoplasm Odontogenic cyst Oesophageal adenocarcinoma Oesophageal adenocarcinoma recurrent Oesophageal adenocarcinoma stage 0 Oesophageal adenocarcinoma stage I Oesophageal adenocarcinoma stage II Oesophageal adenocarcinoma stage III Oesophageal adenocarcinoma stage IV Oesophageal cancer metastatic Oesophageal carcinoma Oesophageal carcinoma recurrent Oesophageal carcinoma stage 0 Oesophageal cyst Oesophageal dysplasia Oesophageal neoplasm Oesophageal papilloma Oesophageal polyp Oesophageal polypectomy Oesophageal prosthesis insertion
Oesophageal squamous cell carcinoma Oesophageal squamous cell carcinoma metastatic Oesophageal squamous cell carcinoma recurrent Oesophageal squamous cell carcinoma stage 0 Oesophageal squamous cell carcinoma stage I Oesophageal squamous cell carcinoma stage II Oesophageal squamous cell carcinoma stage III Oesophageal squamous cell carcinoma stage IV Oesophagectomy Oesophagogastrectomy Oestrogen receptor assay positive Oestrogen receptor positive breast cancer Oligoastrocytoma Oligodendroglioma


03 July 2019 1.0 Final


Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Oligodendroglioma benign Neoplasm Omenn syndrome Omentectomy Oncocytoma Oncologic complication Oophorectomy Oophorectomy bilateral Optic glioma
Optic nerve neoplasm Oral cavity cancer metastatic Oral cavity neoplasm surgery Oral fibroma Oral haemangioma Oral hairy leukoplakia Oral neoplasm Oral neoplasm benign Oral papilloma Oral polypectomy Orbital exenteration Orchidectomy Orchidotomy Oropharyngeal cancer Oropharyngeal cancer recurrent Oropharyngeal cancer stage 0 Oropharyngeal cancer stage I Oropharyngeal cancer stage II Oropharyngeal cancer stage III Oropharyngeal cancer stage IV Oropharyngeal dysplasia Oropharyngeal lymphoepithelioma Oropharyngeal neoplasm Oropharyngeal neoplasm benign Oropharyngeal squamous cell carcinoma Ostectomy Osteochondroma Osteofibroma Osteoma Osteoma cutis Osteosarcoma Osteosarcoma metastatic Osteosarcoma recurrent Ota's naevus Otic cancer metastatic Ovarian Sertoli-Leydig cell tumour Ovarian adenoma Ovarian cancer Ovarian cancer metastatic Ovarian cancer recurrent Ovarian cancer stage I Ovarian cancer stage II Ovarian cancer stage III Ovarian cancer stage IV Ovarian clear cell carcinoma Ovarian cyst Ovarian cyst ruptured Ovarian cyst torsion Ovarian dysgerminoma stage I Ovarian dysgerminoma stage II Ovarian dysgerminoma stage III Ovarian dysgerminoma stage IV Ovarian dysgerminoma stage unspecified Ovarian dysplasia

Ovarian embryonal carcinoma


1.0 Final

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Neoplasm Ovarian endometrioid carcinoma Ovarian epithelial cancer Ovarian epithelial cancer metastatic Ovarian epithelial cancer recurrent Ovarian epithelial cancer stage I Ovarian epithelial cancer stage II Ovarian epithelial cancer stage III Ovarian epithelial cancer stage IV Ovarian fibroma Ovarian germ cell cancer Ovarian germ cell cancer stage I Ovarian germ cell cancer stage II Ovarian germ cell cancer stage III Ovarian germ cell cancer stage IV Ovarian germ cell choriocarcinoma Ovarian germ cell choriocarcinoma stage I Ovarian germ cell choriocarcinoma stage II Ovarian germ cell choriocarcinoma stage III Ovarian germ cell choriocarcinoma stage IV Ovarian germ cell embryonal carcinoma stage I Ovarian germ cell embryonal carcinoma stage II Ovarian germ cell embryonal carcinoma stage III Ovarian germ cell embryonal carcinoma stage IV Ovarian germ cell endodermal sinus tumour Ovarian germ cell endodermal sinus tumour stage I Ovarian germ cell endodermal sinus tumour stage II Ovarian germ cell endodermal sinus tumour stage III Ovarian germ cell endodermal sinus tumour stage IV Ovarian germ cell polyembryoma Ovarian germ cell polyembryoma stage 1 Ovarian germ cell polyembryoma stage II Ovarian germ cell polyembryoma stage III Ovarian germ cell polyembryoma stage IV Ovarian germ cell teratoma Ovarian germ cell teratoma benign Ovarian germ cell teratoma stage I Ovarian germ cell teratoma stage II Ovarian germ cell teratoma stage III Ovarian germ cell teratoma stage IV Ovarian germ cell tumour Ovarian germ cell tumour mixed Ovarian granulosa cell tumour Ovarian granulosa-theca cell tumour Ovarian low malignant potential tumour Ovarian neoplasm Ovarian stromal cancer Ovarian stromal hyperplasia Ovarian theca cell tumour PHACES syndrome PMT. RAR alpha expression POEMS syndrome Paget's disease of nipple Paget's disease of penis Paget's disease of the vulva Palliative care Palmar fasciitis Pancoast's syndrome Pancoast's tumour Pancreastatin abnormal Pancreastatin increased

Pancreatectomy Pancreatic carcinoma


1.0 Final 113 of 152 Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Neoplasm Pancreatic carcinoma metastatic Pancreatic carcinoma recurrent Pancreatic carcinoma stage 0 Pancreatic carcinoma stage Pancreatic carcinoma stage II Pancreatic carcinoma stage III Pancreatic carcinoma stage IV Pancreatic cyst Pancreatic cyst rupture Pancreatic neoplasm Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour metastatic Pancreatic sarcoma Pancreaticoduodenectomy Pancreaticosplenectomy Pancreatoblastoma Papillary cystadenoma lymphomatosum
Papillary renal cell carcinoma
Papillary serous endometrial carcinoma
Papillary thyroid cancer Papillary tumour of renal pelvis Papilloma Papilloma conjunctival Paracancerous pneumonia Paraganglion neoplasm
Paraganglion neoplasm benign
Paraganglion neoplasm malignant Paranasal biopsy abnormal Paranasal cyst Paranasal sinus and nasal cavity malignant neoplasm Paranasal sinus and nasal cavity malignant neoplasm recurrent. Paranasal sinus and nasal cavity malignant neoplasm stage O Paranasal sinus and nasal cavity malignant neoplasm stage I Paranasal sinus and nasal cavity malignant neoplasm stage II Paranasal sinus and nasal cavity malignant neoplasm stage III Paranasal sinus and nasal cavity malignant neoplasm stage IV Paranasal sinus benign neoplasm Paranasal sinus neoplasm Paraneoplastic arthritis Paraneoplastic dermatomyositis Paraneoplastic dermatosis Paraneoplastic encephalomyelitis Paraneoplastic glomerulonephritis Paraneoplastic myelopathy Paraneoplastic nephrotic syndrome Paraneoplastic neurological syndrome Paraneoplastic pemphigus Paraneoplastic pleural effusion Paraneoplastic rash Paraneoplastic retinopathy Paraneoplastic syndrome Paraneoplastic thrombosis Paraproteinaemia Parapsoriasis Parathyroid cyst Parathyroid scan abnormal Parathyroid tumour Parathyroid tumour benign Parathyroid tumour malignant Parathyroidectomy Parotidectomy


1.0 Final 114 of 152

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Pathological fracture Neoplasm Pearly penile papules Pelvic cyst Pelvic neoplasm Penile cancer Penile dysplasia Penile neoplasm Penile operation Penile squamous cell carcinoma Penile wart Penile warts excision Penis carcinoma metastatic Penis carcinoma recurrent Penis carcinoma stage Penis carcinoma stage II Penis carcinoma stage III Penis carcinoma stage IV Pepsinogen test positive Percutaneous ethanol injection therapy Pericardial cyst Pericardial effusion malignant Pericardial mesothelioma malignant Pericardial mesothelioma malignant recurrent Pericardial neoplasm Pericarditis malignant Perineal cyst Perineurial cyst Peripheral T-cell lymphoma unspecified Peripheral T-cell lymphoma unspecified recurrent Peripheral T-cell lymphoma unspecified refractory Peripheral T-cell lymphoma unspecified stage I Peripheral T-cell lymphoma unspecified stage II Peripheral T-cell lymphoma unspecified stage III Peripheral T-cell lymphoma unspecified stage IV Peripheral nervous system neoplasm Peripheral neuroepithelioma of bone Peripheral neuroepithelioma of bone metastatic Peripheral neuroepithelioma of bone recurrent Peripheral neuroepithelioma of soft tissue Peripheral primitive neuroectodermal bone tumour Peripheral primitive neuroectodermal tumour of soft tissue Peritoneal carcinoma metastatic Peritoneal cyst Peritoneal fluid protein increased Peritoneal gliomatosis Peritoneal mesothelioma malignant Peritoneal mesothelioma malignant recurrent Peritoneal neoplasm Peritoneal sarcoma Peritonectomy Peritumoural oedema Peutz-Jeghers syndrome Phaeochromocytoma Phaeochromocytoma crisis Phaeochromocytoma excision Phaeochromocytoma malignant Phakomatosis Pharyngeal cancer Pharyngeal cancer metastatic Pharvngeal cancer recurrent Pharyngeal cancer stage 0 Pharyngeal cancer stage I

Pharyngeal cancer stage II


Final

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Neoplasm Pharyngeal cancer stage III Pharyngeal cancer stage IV Pharyngeal cyst Pharyngeal leukoplakia Pharyngeal mass Pharyngeal neoplasm Pharyngeal neoplasm benign Pharyngeal polyp Pharyngectomy Philadelphia chromosome positive Phosphaturic mesenchymal tumour Photodynamic diagnostic procedure Photon radiation therapy Photon radiation therapy to bladder Photon radiation therapy to blood Photon radiation therapy to bone Photon radiation therapy to brain Photon radiation therapy to breast Photon radiation therapy to colon Photon radiation therapy to ear, nose, or throat Photon radiation therapy to liver Photon radiation therapy to lung Photon radiation therapy to pancreas Photon radiation therapy to pleura Photon radiation therapy to prostate Photon radiation therapy to skin
Photon radiation therapy to soft tissue Photon radiation therapy to thyroid Photon radiation therapy to uterus Phyllodes tumour Pilomatrix carcinoma Pineal germinoma Pineal gland cyst Pineal neoplasm Pineal parenchymal neoplasm malignant Pinealoblastoma Pinealoma Pineocytoma Pituitary cancer metastatic Pituitary cyst Pituitary gland radiotherapy Pituitary neoplasm malignant recurrent Pituitary tumour Pituitary tumour benign Pituitary tumour recurrent Placental chorioangioma Placental neoplasm Placental polyp Plasma cell leukaemia Plasma cell leukaemia in remission Plasma cell myeloma Plasma cell myeloma in remission Plasma cell myeloma recurrent Plasmablastic lymphoma Plasmacytoma Pleomorphic adenoma Pleomorphic liposarcoma Pleomorphic malignant fibrous histiocytoma Pleural cyst Pleural mesothelioma Pleural mesothelioma malignant Pleural mesothelioma malignant recurrent Pleural neoplasm


Date: Version: Status: Page: 03 July 2019 1.0 Final


Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Neoplasm Pleural sarcoma Pleurectomy Pleuropulmonary blastoma Pneumonectomy Polycythaemia vera Polyneuropathy in malignant disease Polvp Poorly differentiated thyroid carcinoma Porocarcinoma Portal vein embolisation
Post breast therapy pain syndrome Post transplant lymphoproliferative disorder Postcricoid cancer Posterior fossa syndrome Postmastectomy lymphoedema syndrome Precancerous lesion excision Precancerous mucosal lesion Precancerous skin lesion Precursor B-lymphoblastic lymphoma Precursor B-lymphoblastic lymphoma recurrent Precursor B-lymphoblastic lymphoma refractory Precursor B-lymphoblastic lymphoma stage I Precursor B-lymphoblastic lymphoma stage II Precursor B-lymphoblastic lymphoma stage III Precursor B-lymphoblastic lymphoma stage IV Precursor T-lymphoblastic lymphoma leukaemia Precursor T-lymphoblastic lymphoma leukaemia recurrent Precursor T-lymphoblastic lymphoma leukaemia refractory Precursor T-lymphoblastic lymphoma leukaemia stage I Precursor T-lymphoblastic lymphoma leukaemia stage II Precursor T-lymphoblastic lymphoma leukaemia stage III Precursor T-lymphoblastic lymphoma leukaemia stage IV Primary breast lymphoma Primary cardiac lymphoma Primary effusion lymphoma Primary gastrointestinal follicular lymphoma Primary mediastinal large B-cell lymphoma Primary mediastinal large B-cell lymphoma recurrent Primary mediastinal large B-cell lymphoma refractory Primary mediastinal large B-cell lymphoma stage I Primary mediastinal large B-cell lymphoma stage II Primary mediastinal large B-cell lymphoma stage III Primary mediastinal large B-cell lymphoma stage IV Primary myelofibrosis Primary pulmonary melanoma Primitive neuroectodermal tumour Primitive neuroectodermal tumour metastatic Proctectomy Proctocolectomy Progesterone receptor assay positive Prolactin-producing pituitary tumour Prolymphocytic leukaemia Prophylactic chemotherapy Prostate ablation Prostate cancer

Prostate cancer metastatic


03 July 2019 Date: Version: 1.0 Status:

Page:

Final 117 of 152 Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

```
Pre-defined MedDRA search
                                                     Preferred term
Neoplasm
                                                      Prostate cancer recurrent
                                                      Prostate cancer stage 0
                                                      Prostate cancer stage
                                                      Prostate cancer stage
                                                      Prostate cancer stage III
Prostate cancer stage IV
                                                      Prostate cryoablation
                                                      Prostate interstitial hyperthermia therapy
                                                      Prostatectomy
                                                      Prostatic adenoma
                                                      Prostatic cyst
                                                      Prostatic dysplasia
                                                      Prostatic polyp
Prostatic specific antigen abnormal
                                                      Prostatic specific antigen increased
                                                      Pseudoachalasia
                                                      Pseudocirrhosis
                                                      Pseudomyxoma peritonei
                                                      Pseudosarcoma
                                                      Pulmonary resection
                                                      Pulmonary tumour thrombotic microangiopathy
                                                      Pylorectomy
                                                      Pyoderma gangrenosum
                                                      Pyogenic granuloma
                                                      Queyrat erythroplasia
                                                      Radiation therapy to ear, nose, or throat Radical cystectomy
                                                      Radical hysterectomy
                                                      Radical mastectomy
                                                      Radical parametrectomy
                                                      Radical prostatectomy
Radioactive iodine therapy
                                                      Radioembolisation
                                                      Radiofrequency ablation of oesophagus
Radiofrequency-induced thermochemotherapeutic effect
                                                      Radioisotope scan abnormal
                                                      Radiosensitisation therapy
                                                      Radiotherapy
Radiotherapy to abdomen
                                                      Radiotherapy to adrenal gland
Radiotherapy to blood
                                                      Radiotherapy to bone
                                                      Radiotherapy to brain
                                                      Radiotherapy to breast
Radiotherapy to colon
Radiotherapy to ear
                                                      Radiotherapy to eye
                                                      Radiotherapy to gallbladder
                                                      Radiotherapy to gastrointestinal tract
Radiotherapy to head and neck
                                                     Radiotherapy to joint
Radiotherapy to kidney
Radiotherapy to liver
Radiotherapy to lung
Radiotherapy to lymph nodes
                                                      Radiotherapy to mediastinum
Radiotherapy to nose
                                                      Radiotherapy to oesophagus
Radiotherapy to oral cavity
                                                      Radiotherapy to ovary
                                                      Radiotherapy to pancreas
Radiotherapy to pleura
                                                      Radiotherapy to prostate
```


Final 118 of 152

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

```
Pre-defined MedDRA search
                                              Preferred term
Neoplasm
                                               Radiotherapy to rectum
                                               Radiotherapy to skin
                                               Radiotherapy to soft tissue
                                               Radiotherapy to spleen Radiotherapy to stomach
                                               Radiotherapy to throat
                                               Radiotherapy to thymus
Radiotherapy to thyroid
                                               Radiotherapy to urinary bladder
                                               Radiotherapy to uterus
                                               Radiotherapy to vagina
                                               Rectal adenocarcinoma
Rectal adenoma
                                               Rectal cancer
                                               Rectal cancer metastatic
                                               Rectal cancer recurrent
                                               Rectal cancer stage 0
                                              Rectal cancer stage I
Rectal cancer stage II
                                               Rectal cancer stage III
                                               Rectal cancer stage IV
                                               Rectal neoplasm
                                               Rectal polyp
                                               Rectal polypectomy
                                               Rectosigmoid cancer
Rectosigmoid cancer metastatic
                                               Rectosigmoid cancer recurrent
                                               Rectosigmoid cancer stage 0
                                               Rectosigmoid cancer stage I
                                               Rectosigmoid cancer stage II
                                               Rectosigmoid cancer stage III
                                               Rectosigmoid cancer stage IV
                                               Recurrent cancer
                                               Refractory anaemia with an excess of blasts
Refractory anaemia with ringed sideroblasts
                                               Refractory cancer
                                               Refractory cytopenia with multilineage dysplasia
                                               Refractory cytopenia with unilineage dysplasia Regional chemotherapy
                                               Renal adenoma
                                               Renal cancer
                                               Renal cancer metastatic
                                               Renal cancer recurrent
                                               Renal cancer stage I
                                               Renal cancer stage II
                                               Renal cancer stage III
                                               Renal cancer stage IV
                                               Renal cell carcinoma
                                               Renal cell carcinoma recurrent
                                               Renal cell carcinoma stage I
                                               Renal cell carcinoma stage II
                                               Renal cell carcinoma stage III
Renal cell carcinoma stage IV
                                               Renal cell dysplasia
                                               Renal cyst
                                               Renal cyst haemorrhage
                                               Renal cyst infection
                                               Renal cyst ruptured
                                               Renal haemangioma
                                               Renal neoplasm
                                               Renal oncocytoma
                                               Renal scan abnormal
                                               Renal tumour excision
```


Final 119 of 152

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

 ${\tt Pre-defined\ MedDRA\ search}$ 

Preferred term

Neoplasm

Respiratory papilloma Respiratory tract carcinoma in situ Respiratory tract neoplasm Retention cyst Retinal melanocytoma Retinal melanoma Retinal neoplasm Retinal tumour excision Retinoblastoma Retro-orbital neoplasm Retro-pubic prostatectomy Retroperitoneal cancer Retroperitoneal neoplasm Retroperitoneal neoplasm metastatic Retroperitoneum cyst Rhabdoid tumour Rhabdoid tumour of the kidney Rhabdomyoma Rhabdomyosarcoma Rhabdomyosarcoma recurrent Richter's syndrome Rosai-Dorfman syndrome Round cell liposarcoma Sacrectomy
Salivary bypass tube insertion
Salivary gland adenoma
Salivary gland cancer Salivary gland cancer recurrent Salivary gland cancer stage 0 Salivary gland cancer stage I Salivary gland cancer stage II Salivary gland cancer stage III Salivary gland cancer stage IV Salivary gland cyst Salivary gland induration Salivary gland neoplasm
Salivary gland resection
Salivary gland scan abnormal
Salpingectomy Salpingo-oophorectomy Salpingo-oophorectomy bilateral Salpingo-oophorectomy unilateral Sarcomá Sarcoma excision Sarcoma metastatic Sarcoma of skin Sarcoma uterus Sarcomatoid carcinoma Sarcomatoid carcinoma of the lung Sarcomatoid mesothelioma Sarcomatosis Scan abdomen abnormal Scan abnormal Scan adrenal gland abnormal Scan bone marrow abnormal Scan gallium abnormal Scan myocardial perfusion abnormal Scan with contrast abnormal Schwannoma Sclerosing pneumocytoma Scrotal cancer Scrotal cyst

Sebaceous adenoma


2019 Novo Nordisk 1.0 Final

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Sebaceous carcinoma

Spinal synovial cyst

Neoplasm

Sebaceous naevus Seborrhoeic keratosis Second primary malignancy Secondary cerebellar degeneration Secretory adenoma of pituitary Seminal vesicular cyst Seminoma Serous cystadenocarcinoma ovary Sertoli cell testicular tumour Sezary cells increased Sigmoidectomy Signet-ring cell carcinoma Silicon granuloma Simple mastectomy Sinonasal papilloma Sinus cancer metastatic Sinus polyp Sinus polyp degeneration Skin angiosarcoma Skin cancer Skin cancer metastatic Skin cryotherapy Skin neoplasm bleeding Skin neoplasm excision Skin papilloma Skin squamous cell carcinoma metastatic Skin squamous cell carcinoma recurrent Small cell carcinoma Small cell carcinoma of the cervix Small cell lung cancer Small cell lung cancer extensive stage Small cell lung cancer limited stage Small cell lung cancer metastatic Small cell lung cancer recurrent Small intestinal polypectomy Small intestinal resection Small intestine adenocarcinoma Small intestine carcinoma Small intestine carcinoma metastatic Small intestine carcinoma recurrent Small intestine carcinoma stage 0 Small intestine carcinoma stage Small intestine carcinoma stage II Small intestine carcinoma stage III Small intestine carcinoma stage IV Small intestine leiomyosarcoma Small intestine polyp Smooth muscle cell neoplasm Soft tissue neoplasm Soft tissue sarcoma Solid pseudopapillary tumour of the pancreas Solitary epithelioid histiocytoma Somatostatin receptor scan abnormal Somatostatinoma Spermatocele Spermatocytic seminoma Spinal cord lipoma Spinal cord neoplasm Spinal meningeal cyst Spinal meningioma benign Spinal meningioma malignant


Final 121 of 152

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Neoplasm Spindle cell sarcoma Spleen scan abnormal Splenectomy Splenic cyst Splenic hamartoma Splenic marginal zone lymphoma Splenic marginal zone lymphoma recurrent Splenic marginal zone lymphoma refractory Splenic marginal zone lymphoma stage I Splenic marginal zone lymphoma stage II Splenic marginal zone lymphoma stage III Splenic marginal zone lymphoma stage IV Splenic neoplasm malignancy unspecified Squamous cell breast carcinoma Squamous cell carcinoma Squamous cell carcinoma of head and neck Squamous cell carcinoma of lung Squamous cell carcinoma of pharynx Squamous cell carcinoma of skin Squamous cell carcinoma of the cervix Squamous cell carcinoma of the hypopharynx Squamous cell carcinoma of the oral cavity Squamous cell carcinoma of the tongue Squamous cell carcinoma of the vagina Squamous cell carcinoma of the vulva Squamous endometrial carcinoma Stauffer's syndrome Steatocystoma multiplex Stem cell therapy Stem cell transplant Stewart-Treves syndrome Stoma site polyp Stomach scan abnormal Superficial spreading melanoma stage I Superficial spreading melanoma stage II Superficial spreading melanoma stage III Superficial spreading melanoma stage IV Superficial spreading melanoma stage unspecified Superior vena cava occlusion Superior vena cava syndrome Suprapubic prostatectomy Sweat gland tumour Synovial cyst Synovial sarcoma Synovial sarcoma metastatic Synovial sarcoma recurrent Systemic mastocytosis T-cell chronic lymphocytic leukaemia T-cell lymphoma T-cell lymphoma recurrent T-cell lymphoma refractory T-cell lymphoma stage I T-cell lymphoma stage II T-cell lymphoma stage III T-cell lymphoma stage T-cell prolymphocytic leukaemia T-cell type acute leukaemia T-cell unclassifiable lymphoma high grade T-cell unclassifiable lymphoma low grade TEMPI syndrome Targeted cancer therapy Tendon neoplasm Teratoma


Final 122 of 152

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Neoplasm Teratoma benign Testicle adenoma Testicular cancer metastatic Testicular choriocarcinoma Testicular choriocarcinoma recurrent Testicular choriocarcinoma stage I Testicular choriocarcinoma stage II Testicular choriocarcinoma stage III Testicular cyst Testicular embryonal carcinoma Testicular embryonal carcinoma stage I Testicular embryonal carcinoma stage II Testicular embryonal carcinoma stage III Testicular germ cell cancer Testicular germ cell cancer metastatic Testicular germ cell tumour Testicular germ cell tumour mixed Testicular germ cell tumour mixed stage I Testicular germ cell tumour mixed stage II Testicular germ cell tumour mixed stage III Testicular leiomyosarcoma Testicular malignant teratoma Testicular malignant teratoma stage I Testicular malignant teratoma stage II Testicular malignant teratoma stage III Testicular neoplasm Testicular papilloma Testicular scan abnormal Testicular seminoma (pure) Testicular seminoma (pure) stage I Testicular seminoma (pure) stage II Testicular seminoma (pure) stage III Testicular teratoma benign Testicular yolk sac tumour Testicular yolk sac tumour stage I Testicular yolk sac tumour stage II Testicular yolk sac tumour stage III Testis cancer Testis cancer recurrent Therapeutic ovarian suppression Throat cancer Thymic cancer metastatic Thymic cyst Thymoma Thymoma malignant Thymoma malignant recurrent Thyroglossal cyst Thyroid B-cell lymphoma Thyroid C-cell hyperplasia Thyroid adenoma Thyroid cancer Thyroid cancer metastatic Thyroid cancer recurrent Thyroid cancer stage 0 Thyroid cancer stage Thyroid cancer stage II Thyroid cancer stage III Thyroid cancer stage IV Thyroid cyst Thyroid electron radiation therapy Thyroid gland scan abnormal Thyroid neoplasm Thyroid stimulating hormone-producing pituitary tumour


03 July 2019 Date: Version: Status: Page:

1.0 Final 123 of 152

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

```
Pre-defined MedDRA search
                                              Preferred term
Neoplasm
                                              Thyroidectomy
                                              Tissue polypeptide antigen increased
                                              Tongue cancer metastatic
                                              Tongue cancer recurrent
                                              Tongue carcinoma stage 0
                                              Tongue carcinoma stage I
                                              Tonque carcinoma stage II
                                              Tongue carcinoma stage III
                                              Tongue carcinoma stage IV
                                              Tongue cyst
                                              Tongue dysplasia
                                              Tongue neoplasm
Tongue neoplasm benign
                                              Tongue neoplasm malignant stage unspecified
                                              Tongue polyp
Tonsil cancer
Tonsil cancer metastatic
                                              Tonsillar cyst
                                              Tonsillar neoplasm
                                              Tonsillar neoplasm benign
                                              Tornwaldt cyst
                                              Total adrenalectomy
                                              Tracheal cancer
                                              Tracheal neoplasm
                                              Tracheal papilloma
Tracheal resection
                                              Transcatheter arterial chemoembolisation
                                              Transcranial electrical motor evoked potential monitoring
                                              Transdifferentiation of neoplasm
                                              Transformation to acute myeloid leukaemia
Transitional cell cancer of renal pelvis and ureter
                                              metastatic
                                              Transitional cell cancer of the renal pelvis and ureter
Transitional cell cancer of the renal pelvis and ureter
                                              localised
                                              Transitional cell cancer of the renal pelvis and ureter
                                              recurrent
                                              Transitional cell cancer of the renal pelvis and ureter
                                              regional
                                              Transitional cell carcinoma
                                              Transitional cell carcinoma metastatic
                                              Transitional cell carcinoma recurrent
                                              Transitional cell carcinoma urethra
                                              Transurethral bladder resection
                                              Transurethral prostatectomy
                                              Trichoblastic carcinoma
                                              Triple hit lymphoma
                                              Triple negative breast cancer
                                              Trisomy 12
                                              Trousseau's syndrome
                                              Tuberous sclerosis complex
Tubular breast carcinoma
                                              Tumour associated fever
Tumour budding
                                              Tumour cavitation
                                              Tumour cell mobilisation
                                              Tumour compression
                                              Tumour embolism
                                              Tumour excision
                                              Tumour exudation
                                              Tumour fistulisation
                                              Tumour flare
```


03 July 2019 Date: Version: 1.0 Status: Page:

Final 124 of 152 Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

```
Pre-defined MedDRA search
                                                 Preferred term
Neoplasm
                                                 Tumour haemorrhage
                                                  Tumour hyperprogression
                                                 Tumour inflammation
                                                 Tumour invasion
                                                 Tumour lysis syndrome
                                                 Tumour marker abnormal
                                                 Tumour marker decreased
                                                 Tumour marker increased
                                                 Tumour necrosis
                                                 Tumour obstruction
                                                 Tumour of ampulla of Vater
                                                 Tumour pain
Tumour perforation
                                                 Tumour pruritus
                                                 Tumour pseudoprogression
                                                 Tumour rupture
                                                 Tumour thrombosis
                                                 Tumour treating fields therapy
Tumour ulceration
Tumour vaccine therapy
                                                 Ulcerated haemangioma
                                                 Ultrasound pancreas abnormal
                                                 Ultrasound scan abnormal
                                                 Ultrasound scan vagina abnormal
                                                 Umbilical cord cyst
Undifferentiated carcinoma of colon
Undifferentiated nasopharyngeal carcinoma
                                                 Undifferentiated sarcoma
                                                 Ureteral cyst
                                                 Ureteral neoplasm
                                                 Ureteral polyp
Ureteric cancer
                                                 Ureteric cancer local
                                                 Ureteric cancer metastatic
                                                 Ureteric cancer recurrent
                                                 Ureteric cancer regional
                                                 Ureteric papilloma
                                                 Urethral adenoma
Urethral cancer
                                                 Urethral cancer metastatic
                                                 Urethral cancer recurrent
                                                 Urethral cyst
                                                 Urethral melanoma metastatic
                                                 Urethral neoplasm
                                                 Urethral papilloma
Urethral polyp
                                                 Urethrectomy
                                                 Urinary bladder adenoma
                                                 Urinary bladder polyp
Urinary bladder sarcoma
                                                 Urinary cystectomy
Urinary tract carcinoma in situ
Urinary tract neoplasm
                                                 Urinary tract polyp
Uterine cancer
                                                 Uterine carcinoma in situ
                                                 Uterine cyst
Uterine leiomyoma
                                                 Uterine leiomyosarcoma
                                                 Uterine myoma expulsion
                                                 Uterine neoplasm
                                                 Uterine polyp
                                                 Uterine tumour excision
```


Final 125 of 152

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Uveal melanoma

Uvulectomy

Neoplasm

Vaccination site cyst Vaginal adenocarcinoma Vaginal cancer Vaginal cancer metastatic Vaginal cancer recurrent Vaginal cancer stage 0 Vaginal cancer stage I Vaginal cancer stage II Vaginal cancer stage III Vaginal cancer stage IVA Vaginal cancer stage IVB Vaginal cyst Vaginal dysplasia Vaginal neoplasm Vaginal polyp Vaginectomy Vascular neoplasm Venous angioma of brain Vipoma Viral acanthoma Vitreous cyst Vocal cord cyst
Vocal cord leukoplakia
Vocal cord neoplasm
Vocal cord polyp Vocal cordectomy Vulva cyst Vulval cancer Vulval cancer metastatic Vulval cancer recurrent Vulval cancer stage 0 Vulval cancer stage Vulval cancer stage II Vulval cancer stage III Vulval cancer stage IV Vulval neoplasm Vulval operation Vulval polyp Vulval warts removal Vulvar adenocarcinoma Vulvar dysplasia Vulvectomy Vulvovaginal adenosis Vulvovaginal warts Waldenstrom's macroglobulinaemia Waldenstrom's macroglobulinaemia recurrent Waldenstrom's macroglobulinaemia refractory Waldenstrom's macroglobulinaemia stage I Waldenstrom's macroglobulinaemia stage II Waldenstrom's macroglobulinaemia stage III Waldenstrom's macroglobulinaemia stage IV Warty dyskeratoma White sponge naevus X-linked lymphoproliferative syndrome X-ray therapy to bladder X-ray therapy to blood X-ray therapy to bone X-ray therapy to brain X-ray therapy to breast X-ray therapy to colon

X-ray therapy to ear, nose, or throat


 Date:
 03 July 2019
 Novo Nordisk

 Version:
 1.0

 Status:
 Final

Page:

Final 126 of 152

Pre-defined MedDRA search - list of preferred terms

| Pre-defined MedDRA search | Preferred term |
|---|---|
| Neoplasm | X-ray therapy to joint |
| | X-ray therapy to liver |
| | X-ray therapy to lung |
| | X-ray therapy to pancreas |
| | X-ray therapy to pleura |
| | X-ray therapy to prostate |
| | X-ray therapy to skin |
| | X-ray therapy to soft tissue |
| | X-ray therapy to thyroid |
| | X-ray therapy to uterus |
| | X-ray treatment<br>Xanthogranuloma |
| | Yolk sac tumour site unspecified |
| Pancreatitis | Alcoholic pancreatitis |
| | Alcoholic pancreopathy |
| | Autoimmune pancreatitis |
| | Cullen's sign |
| | Cytomegalovirus pancreatitis |
| | Grey Turner's sign |
| | Haemorrhagic necrotic pancreatitis Hereditary pancreatitis |
| | Ischaemic pancreatitis |
| | Lupus pancreatitis |
| | Obstructive pancreatitis |
| | Oedematous pancreatitis |
| | Pancreas infection |
| | Pancreatic abscess |
| | Pancreatic haemorrhage |
| | Pancreatic necrosis |
| | Pancreatic phlegmon |
| | Pancreatic pseudoaneurysm |
| | Pancreatic pseudocyst |
| | Pancreatic pseudocyst drainage |
| | Pancreatitis |
| | Pancreatitis acute |
| | Pancreatitis bacterial |
| | Pancreatitis chronic |
| | Pancreatitis fungal |
| | Pancreatitis haemorrhagic |
| | Pancreatitis helminthic |
| | Pancreatitis mumps Pancreatitis necrotising |
| | Pancreatitis relapsing |
| | Pancreatitis viral |
| | Pancreatorenal syndrome |
| | Radiation pancreatitis |
| | Traumatic pancreatitis |
| | ridamacio panoreacicio |
| Rare | 11-beta-hydroxylase deficiency |
| | 17,20-desmolase deficiency |
| | 17-alpha-hydroxylase deficiency |
| | 18q minus syndrome |
| | 2-Hydroxyglutaric aciduria |
| | 20,22-desmolase deficiency |
| | 21-hydroxylase deficiency |
| | 3-hydroxyacetyl-coenzyme A dehydrogenase deficiency |
| | 3M syndrome |
| | 5-alpha-reductase deficiency |
| | ABO haemolytic disease of newborn |
| | ACAD9 deficiency |
| | Aase syndrome<br>Abdominal transposition |

Pre-defined MedDRA search


Preferred term


Page:

1.0 Final 127 of 152 Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Abdominal wall anomaly Rare Abnormal palmar plantar creases Acardia Accessory auricle Accessory breast Accessory breast
Accessory carpal bone
Accessory kidney
Accessory liver lobe
Accessory muscle
Accessory navicular syndrome
Accessory salivary gland
Accessory spleen Acetylcholinesterase deficiency Achromotrichia congenital Acquired amegakaryocytic thrombocytopenia Acral peeling skin syndrome Acrodermatitis enteropathica Acrodysostosis Acrokeratosis verruciformis Activated PI3 kinase delta syndrome Acute focal bacterial nephritis Adactyly Adams-Oliver syndrome Adenine phosphoribosyl transferase deficiency Adenylosuccinate lyase deficiency Adrenal insufficiency neonatal Adrenogenital syndrome Adrenoleukodystrophy Adult polyglucosan body disease Aglossia Agranulocytosis Aicardi's syndrome Alagille syndrome Albinism Albright's disease Alkaptonuria Allan-Herndon-Dudley syndrome Alpers' disease Alpha-1 anti-trypsin deficiency Alport's syndrome Alstroem syndrome Alternating hemiplegia of childhood Alveolar capillary dysplasia Amblyopia congenital Amegakaryocytic thrombocytopenia Amelogenesis imperfecta Aminoaciduria Amniotic band syndrome Amyotrophic lateral sclerosis gene carrier Anal atresia Androgen insensitivity syndrome Anencephaly Angelman's syndrome Angiotensin converting enzyme inhibitor foetopathy

Aniridia

Ankyloglossia congenital

Anomalous arrangement of pancreaticobiliary duct

Anomalous pulmonary venous connection Anomaly of external ear congenital Anomaly of middle ear congenital

Annular pancreas Anodontia


1.0 Final

Novo Nordisk


Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Benjamin syndrome Berdon's syndrome

Anomaly of orbit, congenital

Rare

Anophthalmos Anorchism Anorectal agenesis Anotia Anterior chamber cleavage syndrome Anterior displaced anus Antithrombin III deficiency Aorta hypoplasia Aortic valve atresia Aorticopulmonary septal defect Apert's syndrome Aphakia congenital Aplasia Aplasia cutis congenita Aplastic anaemia Apparent mineralocorticoid excess Arachnodactyly Arcuate foramen
Arginase deficiency Argininosuccinate lyase deficiency Argininosuccinate synthetase deficiency Arnold-Chiari malformation Arterial tortuosity syndrome Arteriovenous malformation Ash leaf macule Aspartate-glutamate-transporter deficiency Aspartylglucosaminuria Asphyxiating thoracic dystrophy Asplenia Asymptomatic gene carrier Ataxia telangiectasia Atrial septal defect Atrioventricular septal defect Auditory neuropathy spectrum disorder Autoimmune aplastic anaemia Autoimmune lymphoproliferative syndrome Autoimmune nephritis Autosomal chromosome anomaly Azygos lobe B-lymphocyte abnormalities B-lymphocyte count abnormal B-lymphocyte count decreased BPES syndrome Baltic myoclonic epilepsy
Band neutrophil count decreased
Band neutrophil percentage decreased Baraitser Rodeck Garner syndrome Barakat syndrome Barth syndrome
Bartter's syndrome
Basophil count abnormal
Basophil count decreased Basophil percentage decreased Basophilopenia Becker's muscular dystrophy Beckwith-Wiedemann syndrome Benign congenital hypotonia Benign familial haematuria Benign familial neonatal convulsions Benign familial pemphigus


 Date:
 03 July 2019

 Version:
 1.0

 Status:
 Final

Page:

Final 129 of 152

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Cervical auricle

Rare

Bergmeister's papilla Beta ketothiolase deficiency Bicuspid aortic valve Bicuspid pulmonary valve Bicytopenia Biotinidase deficiency Birth mark Bladder agenesis Blau syndrome Blepharophimosis congenital Blindness congenital Bloch-Sulzberger syndrome Blood count abnormal Blood disorder Blood incompatibility haemolytic anaemia of newborn Bloom syndrome Bone marrow disorder Bone marrow failure Bone marrow myelogram abnormal Bone marrow necrosis Bone marrow toxicity Brachycephaly Brachydactyly Brachymetatarsia Brain malformation Branchial cleft sinus Branchio-oto-renal syndrome Branchiogenic syndrome Breast malformation Bronchial atresia Bronchogenic cyst Brunner syndrome Bruton's agammaglobulinaemia Bulbospinal muscular atrophy congenital Buried penis syndrome Clq nephropathy C3 glomerulopathy CANDLE syndrome CHARGE syndrome CTLA4 deficiency Camptodactyly congenital Camptomelia Canavan disease Cancer gene carrier Carbamoyl phosphate synthetase deficiency Carbohydrate metabolism disorder Cardiac malposition Cardiac septal defect Carnitine palmitoyltransferase deficiency Carnitine-acylcarnitine translocase deficiency Carpenter syndrome Carpus curvus Cartilage-hair hypoplasia Cataract congenital Caudal regression syndrome Central core disease Cerebellar dysplasia Cerebellar hypoplasia Cerebral atrophy congenital Cerebral dysgenesis Cerebral palsy Cerebrohepatorenal syndrome


2019 Novo Nordisk 1.0 Final

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Rare Cervical rib Chediak-Higashi syndrome Chiari network Chimerism Choanal atresia Choanal stenosis Cholangiectasis congenital Chondrodystrophy Chondroectodermal dysplasia Chordee Chorea-acanthocytosis Chorioretinal degeneration congenital Choroidal coloboma Chromosomal deletion Chromosomal mutation Chronic autoimmune glomerulonephritis Chronic granulomatous disease Chronic infantile neurological cutaneous and articular svndrome Citrate transporter deficiency Cleft lip Cleft lip and palate Cleft palate Cleft uvula Cleidocranial dysostosis Clinodactyly Cloacal exstrophy Clostridial infection Clostridial sepsis Clostridium bacteraemia Clostridium colitis Clostridium difficile colitis Clostridium difficile infection Clostridium test positive Coagulation factor mutation Coarctation of the aorta Cobb syndrome Cockayne's syndrome Cohen syndrome Collodion baby Coloboma Colour blindness Combined immunodeficiency Complement deficiency disease Congenital Eustachian tube anomaly Congenital HIV infection Congenital Horner's syndrome Congenital Zika syndrome Congenital abdominal hernia
Congenital absence of bile ducts
Congenital absence of cranial vault
Congenital absence of vertebra
Congenital adrenal gland hypoplasia Congenital amputation Congenital anaemia Congenital androgen deficiency Congenital anomalies of ear ossicles Congenital anomaly Congenital anomaly in offspring Congenital anomaly of adrenal gland Congenital anomaly of inner ear Congenital anosmia

Congenital aortic anomaly

Pre-defined MedDRA search


2019 Novo Nordisk 1.0 Final

Pre-defined MedDRA search - list of preferred terms

Rare

Preferred term

Congenital aortic atresia

```
Congenital aortic dilatation
Congenital aortic stenosis
Congenital aortic valve incompetence
Congenital aortic valve stenosis
Congenital aplastic anaemia
Congenital aqueductal stenosis
Congenital arterial malformation
Congenital arteriovenous fistula
Congenital astigmatism
Congenital aural fistula
Congenital bladder anomaly
Congenital bladder diverticulum
Congenital bladder neck obstruction
Congenital bowing of long bones
Congenital brain damage
Congenital bronchiectasis
Congenital bronchomalacia
Congenital calyceal diverticulum
Congenital cardiovascular anomaly
Congenital carnitine deficiency
Congenital central diabetes insipidus
Congenital central hypoventilation syndrome
Congenital central nervous system anomaly
Congenital cerebellar agenesis
Congenital choroidal anomaly
Congenital chylothorax
Congenital clavicular agenesis
Congenital claw toe
Congenital coagulopathy
Congenital condyloma
Congenital corneal anomaly
Congenital coronary artery malformation
Congenital cranial nerve paralysis
Congenital cutis laxa
Congenital cystic lung
Congenital cytomegalovirus infection
Congenital deformity of clavicle
Congenital dermal sinus
Congenital diaphragmatic anomaly
Congenital diaphragmatic eventration
Congenital diaphragmatic hernia
Congenital disorder of glycosylation
Congenital dyserythropoietic anaemia
Congenital dysfibrinogenaemia
Congenital dyskeratosis
Congenital ectodermal dysplasia
Congenital ectopic bladder
Congenital ectopic pancreas
Congenital elevation of scapula
Congenital emphysema
Congenital endocrine anomaly Congenital epiblepharon
Congenital epiglottal anomaly
Congenital eye disorder
Congenital eyelid malformation
Congenital facial nerve hypoplasia
Congenital fallopian tube anomaly
Congenital flaccid paralysis
Congenital flat feet
Congenital floppy infant
Congenital foot malformation
```

Congenital gastric anomaly


03 July 2019 | **Novo Nordisk**1.0 | Final


Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Congenital gastrointestinal vessel anomaly Rare Congenital generalised lipodystrophy Congenital genital malformation Congenital genital malformation female Congenital genital malformation male Congenital genitourinary abnormality Congenital great vessel anomaly Congenital haematological disorder Congenital hair disorder Congenital hand malformation Congenital hearing disorder Congenital heart valve disorder Congenital heart valve incompetence Congenital hepatic fibrosis Congenital hepatitis B infection Congenital hepatobiliary anomaly Congenital hepatomegaly Congenital herpes simplex infection Congenital hiatus hernia Congenital high airway obstruction syndrome Congenital hydrocele renalis Congenital hydrocephalus Congenital hydronephrosis Congenital hypercoagulation Congenital hyperextension of knee Congenital hyperextension of spine Congenital hypertrichosis Congenital hypogammaglobulinaemia Congenital hypoparathyroidism Congenital hypoplasia of depressor angularis oris muscle Congenital infection Congenital inguinal hernia Congenital intestinal malformation Congenital intestinal obstruction Congenital intrinsic factor deficiency Congenital iris anomaly Congenital jaw malformation Congenital joint malformation Congenital knee deformity Congenital knee dislocation Congenital kyphoscoliosis Congenital labia pudendi adhesions Congenital lacrimal gland anomaly Congenital lacrimal passage anomaly Congenital large intestinal atresia Congenital laryngeal stridor Congenital lenticonus Congenital limb hyperextension Congenital lip fistula Congenital lymphoedema Congenital malaria Congenital megacolon Congenital megaureter Congenital melanosis Congenital methaemoglobinaemia Congenital midline defect Congenital mitochondrial cytopathy Congenital mitral valve incompetence Congenital mitral valve stenosis Congenital monorchidism Congenital multiplex arthrogryposis Congenital muscle absence Congenital musculoskeletal anomaly


Date: Version: Status: 03 July 2019 | **Novo Nordisk** 

Status: Final 

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Rare Congenital myopathy Congenital myopia Congenital nail disorder Congenital nephrogenic diabetes insipidus Congenital nephrotic syndrome Congenital neurological degeneration Congenital neurological disorder Congenital neuropathy Congenital night blindness Congenital nipple anomaly Congenital nipple inversion Congenital nose malformation Congenital nystagmus Congenital oculomotor apraxia Congenital oesophageal anomaly Congenital oesophageal stenosis Congenital oesophageal web Congenital optic nerve anomaly Congenital oral malformation Congenital osteodystrophy Congenital ovarian anomaly Congenital oxalosis Congenital pancreatic anomaly Congenital perforated nasal septum Congenital pharyngeal anomaly Congenital pigmentation disorder Congenital pneumonia Congenital poikiloderma Congenital pseudarthrosis Congenital pulmonary artery anomaly Congenital pulmonary hypertension Congenital pulmonary valve atresia Congenital pulmonary valve disorder Congenital pyelocaliectasis Congenital renal disorder Congenital rubella infection Congenital salivary gland anomaly Congenital scleral disorder Congenital scoliosis Congenital scrotal hypertrophy Congenital skin dimples Congenital skin disorder Congenital small intestinal atresia Congenital spinal cord anomaly Congenital spinal fusion Congenital spinal stenosis Congenital spondylolisthesis Congenital spondylolysis Congenital syphilis
Congenital syphilitic encephalitis Congenital syphilitic meningitis Congenital syphilitic osteochondritis Congenital thrombocyte disorder Congenital thrombocytopenia Congenital thymus absence Congenital tongue anomaly Congenital torticollis Congenital toxoplasmosis Congenital tracheomalacia Congenital trichomegaly Congenital tricuspid valve atresia Congenital tricuspid valve incompetence Congenital tricuspid valve stenosis


03 July 2019 Date:

Novo Nordisk

Version: 1.0 Final Status: 

Pre-defined MedDRA search - list of preferred terms

```
Pre-defined MedDRA search
                                              Preferred term
Rare
                                               Congenital tuberculosis
                                               Congenital umbilical hernia
                                               Congenital ureteric anomaly
                                               Congenital ureterocele
                                               Congenital ureterovesical junction anomaly
                                               Congenital urethral anomaly
                                              Congenital urinary tract obstruction
Congenital uterine anomaly
                                               Congenital varicella infection
                                               Congenital varicocele
                                               Congenital vas deferens absence
                                               Congenital vesicoureteric reflux
                                               Congenital visual acuity reduced
                                               Congenital vitreous anomaly
                                               Congenital white blood cell disorder
                                               Conjoined twins
                                              Conjunctivitis gonococcal neonatal Constricted ear deformity
                                               Cor biloculare
                                               Cor triatriatum
                                               Corneal dystrophy
                                               Corneal opacity congenital
                                               Cornelia de Lange syndrome
                                               Corrected transposition of great vessels
                                              Cortical dysplasia
Costello syndrome
                                               Craniofacial deformity
                                               Craniofacial dysostosis
                                               Craniolacunia
                                               Craniorachischisis
                                               Craniosynostosis
                                               Craniotabes
                                               Cri du Chat syndrome
                                               Crigler-Najjar syndrome
                                               Cryopyrin associated periodic syndrome
                                               Cryptophthalmos
                                               Cryptorchism
                                              Currarino syndrome
Cutaneovisceral angiomatosis with thrombocytopenia
                                               Cyclic neutropenia
                                               Cyclopia
                                               Cystathionine beta-synthase deficiency
                                               Cystic fibrosis
                                               Cystic fibrosis carrier
                                              Cystic fibrosis gastrointestinal disease
Cystic fibrosis hepatic disease
                                               Cystic fibrosis lung
                                               Cystic fibrosis pancreatic
                                              Cystic fibrosis related diabetes Cystinosis
                                               Cystinuria
                                              Cytogenetic abnormality
Cytomegalovirus nephritis
                                               Cytopenia
                                               DNA mismatch repair protein gene mutation
                                               DOOR syndrome
                                               Dacryostenosis congenital
                                               Dandy-Walker syndrome
                                               Deaf mutism
                                               Deafness congenital
                                               Deficiency of the interleukin-1 receptor antagonist Deficiency of the interleukin-36 receptor antagonist
                                               Delayed foetal renal development
```


Date: 03 July 2019 Version: 1.0

Novo Nordisk

Status: Final 

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Rare

Delta-beta thalassaemia Dent's disease Dentatorubral-pallidoluysian atrophy Dentinogenesis imperfecta Dentofacial anomaly
Dermatofibrosis lenticularis disseminata
Dermatoglyphic anomaly Developmental glaucoma Developmental hip dysplasia Dextrocardia DiGeorge's syndrome Diabetic foetopathy Diaphragmatic aplasia Diastematomyelia Diastrophic dysplasia Diencephalic syndrome of infancy Diethylstilboestrol syndrome Differential white blood cell count abnormal Dihydropyrimidine dehydrogenase deficiency Dilatation intrahepatic duct congenital Disorder of sex development Distichiasis Diverticulitis Meckel's Diverticulum of pharynx, congenital Dolichocolon Dopa-responsive dystonia Double cortex syndrome Double heterozygous sickling disorders Double outlet left ventricle Double outlet right ventricle Double ureter Dowling-Degos disease Duane's syndrome Dubin-Johnson syndrome Dubowitz syndrome Duchenne muscular dystrophy Duchenne muscular dystrophy gene carrier Ductus arteriosus premature closure Ductus arteriosus stenosis foetal Ductus venosus agenesis Duodenal atresia Duplex appendix Duplication of inferior vena cava Dyke-Davidoff-Masson syndrome Dvschondrosteosis Dyschromatosis Dysgnathia Dysmorphism Dysmyelination Eagle Barrett syndrome Ear malformation Early onset familial Alzheimer's disease Early onset primary dystonia Ebstein's anomaly Ectopia cordis Ectopic kidney Ectopic ovary Ectopic posterior pituitary gland Ectopic ureter Ectrodactyly Ehlers-Danlos syndrome Elliptocytosis hereditary

Ellis-van Creveld syndrome


1.0 Final 136 of 152

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Rare

Emanuel syndrome Emery-Dreifuss muscular dystrophy Encephalocele Encephalocutaneous angiomatosis Enteric duplication Entropion congenital Eosinopenia Eosinophil count abnormal Eosinophil count decreased Eosinophil percentage decreased Epidermal naevus Epilepsy congenital
Epilepsy with myoclonic-atonic seizures Epispadias Erythroblastosis foetalis Erythrokeratodermia variabilis Essential fructosuria Exomphalos Exophthalmos congenital External auditory canal atresia Extrarenal pelvis Eye anterior chamber congenital anomaly Eyelid ptosis congenital Fabry's disease Faciodigitogenital dysplasia Facioscapulohumeral muscular dystrophy Factor I deficiency Factor II deficiency Factor II mutation Factor III deficiency Factor IX deficiency Factor V Leiden carrier Factor V Leiden mutation Factor V deficiency Factor VII deficiency Factor VIII deficiency Factor X deficiency Factor XI deficiency Factor XII deficiency Factor XIII deficiency Fallot's pentalogy Fallot's tetralogy Fallot's terlalogy
Familial amyloidosis
Familial amyotrophic lateral sclerosis
Familial cold autoinflammatory syndrome Familial hemiplegic migraine Familial high density lipoprotein deficiency Familial hypertriglyceridaemia Familial hypocalciuric hypercalcaemia Familial infantile bilateral striatal necrosis Familial isolated hyperparathyroidism Familial mediterranean fever Familial periodic paralysis Familial polycythaemia Familial renal glycosuria Familial scaphocephaly syndrome Familial tremor Fanconi syndrome Fatal familial insomnia Fatty acid oxidation disorder

Febrile bone marrow aplasia Febrile neutropenia


 Date:
 03 July 2019

 Version:
 1.0

 Status:
 Final

Final 137 of 152

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Rare

Femoral anteversion Femoral retroversion Femur-fibula-ulna complex Fibrillary glomerulonephritis Fibrodysplasia ossificans progressiva Fibrous dysplasia of bone Fibrous dysplasia of jaw Fibula agenesis Fissure of tongue, congenital Floating-Harbor syndrome Focal segmental glomerulosclerosis Foetal alcohol syndrome Foetal anticonvulsant syndrome Foetal chromosome abnormality Foetal malformation Foetal megacystis Foetal methotrexate syndrome Foetal retinoid syndrome Foetal warfarin syndrome Foramen magnum stenosis Fragile X carrier Fragile X syndrome Fraser syndrome Freeman-Sheldon syndrome Frenulum breve Friedreich's ataxia Fructose-1,6-bisphosphatase deficiency Fryns syndrome Full blood count abnormal Full blood count decreased GNE myopathy GRACILE syndrome Galactosaemia Gallbladder agenesis Gallbladder anomaly congenital Gastroenteritis clostridial Gastrointestinal arteriovenous malformation Gastrointestinal disorder congenital Gastrointestinal malformation Gastroschisis Gatad2b associated neurodevelopmental disorder Gaucher's disease Gaucher's disease type I Gaucher's disease type II Gaucher's disease type III Gelatinous transformation of the bone marrow Gene mutation Genitalia external ambiguous Gilbert's syndrome Gitelman's syndrome Glomerulonephritis Glomerulonephritis acute Glomerulonephritis chronic Glomerulonephritis membranoproliferative Glomerulonephritis membranous Glomerulonephritis minimal lesion Glomerulonephritis proliferative Glomerulonephritis rapidly progressive Glucose transporter type 1 deficiency syndrome Glucose-6-phosphate dehydrogenase deficiency Glucose-galactose malabsorption Glutathione synthetase deficiency Glycogen storage disease type I

Page:


Date: Version: Status: 03 July 2019 1.0

Novo Nordisk

Status: Final 

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Rare Glycogen storage disease type II Glycogen storage disease type III Glycogen storage disease type IV Glycogen storage disease type V Glycogen storage disease type VI Glycogen storage disease type VII Glycogen storage disease type VIII Glycogen storage disorder Gnathoschisis Gollop-Wolfgang complex Gonadal dysgenesis Granulocyte count decreased Granulocytes abnormal Granulocytes maturation arrest Granulocytopenia Granulocytopenia neonatal Gray matter heterotopia Greig's syndrome Griscelli syndrome HIV associated nephropathy Haematotoxicity Haemochromatosis trait Haemoglobin C disease Haemoglobin C trait Haemoglobin D disease Haemoglobin D trait Haemoglobin E disease Haemoglobin E trait Haemoglobin E-thalassaemia disease Haemoglobinopathy Haemophilia Haemophilia A with anti factor VIII Haemophilia A without inhibitors Haemophilia B with anti factor IX Haemophilia B without inhibitors Haemophilia carrier Haemorrhagic arteriovenous malformation Hand-foot-genital syndrome Harlequin foetus Hartnup disease Heart disease congenital Hemihypertrophy Hemimegalencephaly Hemivertebra Hepatic arteriovenous malformation Hepatitis virus-associated nephropathy Hepato-lenticular degeneration Hereditary angioedema with normal C1 esterase inhibitor Hereditary areflexic dystasia Hereditary cerebral degeneration Hereditary choroidal dystrophy Hereditary disorder Hereditary fructose intolerance Hereditary haemochromatosis Hereditary haemolytic anaemia Hereditary haemorrhagic telangiectasia Hereditary hypophosphataemic rickets
Hereditary motor and sensory neuropathy
Hereditary motor neurone disease
Hereditary neuropathic amyloidosis Hereditary neuropathy with liability to pressure palsies Hereditary optic atrophy Hereditary palmoplantar keratoderma


1.0 Final 139 of 152

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

 ${\tt Pre-defined \ MedDRA \ search}$ 

Preferred term

Rare

Hereditary renal microhaematuria Hereditary retinal dystrophy Hereditary sideroblastic anaemia Hereditary spastic paraplegia Hereditary spherocytosis Hereditary stomatocytosis Hermansky-Pudlak syndrome Hermaphroditism Hernia congenital Heterochromia iridis Heterotaxia Hexokinase deficiency anaemia High arched palate Hollow visceral myopathy Holoprosencephaly Holt-Oram syndrome Homocystinaemia Homocystinuria Hooded prepuce Huntington's disease Hydranencephaly Hydrocele Hydronephrosis Hydroureter
Hydroxyprolinaemia
Hyper IgD syndrome
Hyper IgE syndrome Hyper IgM syndrome Hyperexplexia Hyperglycinaemia Hyperinsulinism syndrome Hyperlysinaemia Hypermethioninaemia Hypermethioniuria Hyperprolinaemia Hypersplenism congenital Hypertelorism of orbit Hyperthermia malignant Hypocalvaria Hypochondroplasia Hypodontia Hypomelanosis of Ito Hypophosphatasia Hypopituitarism foetal Hypoplastic left heart syndrome Hypoplastic nasal cartilage Hypoplastic right heart syndrome Hypospadias Hypotelorism of orbit Hypoxanthine-guanine phosphoribosyl transferase deficiency IPEX syndrome Ichthyosis Idiopathic neutropenia IgA nephropathy IgM nephropathy Ileal atresia Immunodeficiency congenital
Immunotactoid glomerulonephritis Imperforate hymen Imperforate oesophagus Inborn error in primary bile acid synthesis Inborn error of bilirubin metabolism Inborn error of lipid metabolism


1.0 Final 140 of 152

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

 ${\tt Pre-defined \ MedDRA \ search}$ 

Preferred term

Leukodystrophy

Rare

Inborn error of metabolism Infantile cortical hyperostosis Infantile genetic agranulocytosis Inherited cardiac conduction disorder Iniencephaly Interferon gamma receptor deficiency Interruption of aortic arch Intestinal atresia Intestinal malrotation Intestinal neuronal dysplasia Intestinal sepsis
Intestinal transposition Intracranial arterial fenestration Intracranial lipoma Iris coloboma Isodicentric chromosome 15 syndrome Johanson-Blizzard syndrome Joubert syndrome Juvenile Paget's disease Kabuki make-up syndrome Kaufman-McKusick syndrome Kearns-Sayre syndrome Kenny-Caffey syndrome Kenatitis-ichthyosis-deafness syndrome Keratolysis exfoliativa congenital Keratosis follicular Kidney duplex Kidney malformation Kidney malrotation Kimmerle's anomaly Kinematic imbalances due to suboccipital strain Kleefstra syndrome Klinefelter's syndrome Klippel-Feil syndrome Klippel-Trenaunay syndrome Kniest dysplasia Kommerell's diverticulum Kosaki overgrowth syndrome Krabbe's disease Kyphosis congenital LDLR mutation Labial tie Lacrimal punctum agenesis Laevocardia Lafora's myoclonic epilepsy Lamin A C gene mutation Langer-Giedion syndrome Laron syndrome Larsen syndrome Laryngeal cleft Laryngeal web Laryngo-onycho-cutaneous syndrome Laryngocele Laryngomalacia Laurence-Moon-Bardet-Biedl syndrome Leber's congenital amaurosis Lecithin-cholesterol acyltransferase deficiency Left ventricle outflow tract obstruction Left ventricular false tendon Left-to-right cardiac shunt Lens abnormality, congenital


Date: Version: Status:

Page:

03 July 2019 | **Novo Nordisk** 

Final 141 of 152

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Rare

Leukopenia Leukopenia neonatal Li-Fraumeni syndrome Lichen spinulosus Liddle's syndrome Limb hypoplasia congenital Limb malformation Limb reduction defect Lipid proteinosis Lipidosis Lipomeningocele Lissencephaly Loeys-Dietz syndrome Long-chain acyl-coenzyme A dehydrogenase deficiency Low set ears Lowry-Wood syndrome Lumbarisation Lupus nephritis Lymphangiectasia intestinal congenital Lymphocyte count abnormal Lymphocyte count decreased Lymphocyte percentage abnormal Lymphocyte percentage decreased Lymphocytopenia neonatal Lymphopenia Lysinuric protein intolerance Lysosomal acid lipase deficiency MĒLAS syndrome MLASA syndrome MYH9-related disease Macrocephaly Macrocheilia Macrocornea Macrodactyly Macrogenia Macroglossia Macrognathia Macrostomia Macrotia Macular dystrophy congenital Majeed's syndrome Malformation biliary Malformation venous Mandibulofacial dysostosis Maple syrup disease Marcus Gunn syndrome Marfan's syndrome Maxillonasal dysplasia Mayer-Rokitansky-Kuster-Hauser syndrome McLeod neuroacanthocytosis syndrome Medium-chain acyl-coenzyme A dehydrogenase deficiency Megakaryocytes decreased Meier-Gorlin syndrome Melkersson-Rosenthal syndrome Membranous lipodystrophy Meningocele Meningomyelocele Menkes' syndrome

Mesangioproliferative glomerulonephritis Metabolic myopathy Metachromatic leukodystrophy Metamyelocyte count decreased

Metaphyseal dysplasia


 Date:
 03 July 2019

 Version:
 1.0

 Status:
 Final

Page:

Final 142 of 152

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term

Rare

Metatarsus primus varus Methylenetetrahydrofolate reductase deficiency Methylenetetrahydrofolate reductase gene mutation Methylmalonic aciduria Mevalonate kinase deficiency Mevalonic aciduria Microcephaly Microcheilia Microcolon Microcornea Microencephaly Microgenia Microglossia Micrognathia Microorchidism Micropenis Microphthalmos Microstomia Microtia Microvillous inclusion disease Mitochondrial DNA deletion Mitochondrial DNA depletion Mitochondrial DNA duplication Mitochondrial DNA mutation Mitochondrial encephalomyopathy Mitochondrial enzyme deficiency Mitochondrial hepatopathy Mitochondrial myopathy Mitochondrial neurogastrointestinal encephalopathy Mitral valve atresia Mitral valve hypoplasia Mittendorf dot Mobile caecum syndrome Moebius II syndrome Molybdenum cofactor deficiency Monoblast count decreased Monocyte count abnormal Monocyte count decreased Monocyte percentage decreased Monocytopenia Monolid eyes Monopodia Morgagni-Stewart-Morel syndrome Morning glory syndrome Morton's syndrome Mosaicism Mount-Reback syndrome Muckle-Wells syndrome Mucolipidosis Mucolipidosis type I Mucolipidosis type II Mucolipidosis type III Mucolipidosis type IV Mucopolysaccharidosis Mucopolysaccharidosis I Mucopolysaccharidosis II Mucopolysaccharidosis III Mucopolysaccharidosis IV Mucopolysaccharidosis IX Mucopolysaccharidosis V Mucopolysaccharidosis VI

Mucopolysaccharidosis VII Multiple carboxylase deficiency


Date: Version: Status:

Page:

03 July 2019 1.0


Final

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

\_\_\_\_\_

Pre-defined MedDRA search

Preferred term

Multiple cardiac defects

Optic nerve hypoplasia

Rare

Multiple congenital abnormalities Multiple epiphyseal dysplasia Multiple gastrointestinal atresias Multiple lentigines syndrome Muscular dystrophy Mutagenic effect Myeloblast count decreased Myeloblast percentage decreased Myelocyte count decreased Myelocyte percentage decreased Myeloid maturation arrest Myeloperoxidase deficiency Myocardial bridging Myoclonic epilepsy and ragged-red fibres Myotonia congenita Myotonic dystrophy N-acetylglutamate synthase deficiency Naevus anaemicus Naevus flammeus Naevus spider congenital Nail aplasia Nail-patella syndrome Nasopharyngeal atresia Neonatal alloimmune thrombocytopenia Neonatal haemochromatosis Neonatal lupus erythematosus Nephritic syndrome Nephritis haemorrhagic Nephritis radiation Nephrotic syndrome Netherton's syndrome Neural tube defect Neuroacanthocytosis Neuroleptic malignant syndrome Neuronal ceroid lipofuscinosis Neuronal migration disorder Neuropathy, ataxia, retinitis pigmentosa syndrome Neutropenia Neutropenia neonatal Neutropenic infection Neutropenic sepsis Neutrophil count abnormal Neutrophil count decreased Neutrophil count decreased Neutrophil percentage decreased Niemann-Pick disease Nijmegen breakage syndrome Non-compaction cardiomyopathy Noonan syndrome Norrie's disease Ocular albinism Oculocariculovertebral dysplasia Oculocerebrorenal syndrome Oculodentodigital dysplasia Oculopharyngeal dystrophy Oculopharyngeal dystrophy Oesophageal atresia Olfacto genital dysplasia Olfactory nerve agenesis Olmsted syndrome Opitz-G BBB syndrome Optic disc pit


2019 Novo Nordisk 1.0 Final

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Platyspondylia

Rare

Oral-facial-digital syndrome type II Ornithine transcarbamoylase deficiency Oroticaciduria congenital Os trigonum Osteogenesis imperfecta Osteopathia striata Osteopetrosis Osteopoikilosis Osteoporosis-pseudoglioma syndrome Otocephaly Ovarian agenesis Ovarian hypoplasia Oxycephaly PIK3CA related overgrowth spectrum Pachydermoperiostosis Pachygyria Pachyonychia congenita Pallister-Killian syndrome Pancreas divisum Pancytopenia Panmyelopathy Parachute mitral valve Paranasal sinus aplasia Parkes-Weber syndrome Patent ductus arteriosus Pearson's syndrome Pectus carinatum Pectus excavatum Pelizaeus-Merzbacher disease Pelvi-ureteric obstruction Pelvic fibrosis Pelvic kidney Penile torsion Penoscrotal fusion Penoscrotal transposition Perinephritis Periodontal congenital anomaly Perry syndrome Persistent Muellerian duct syndrome Persistent cloaca Persistent foetal circulation Persistent left superior vena cava Persistent pupillary membrane Persistent urogenital sinus Phalangeal agenesis Phalangeal hypoplasia Phenylketonuria Phimosis Phytosterolaemia Pierre Robin syndrome Pilonidal cyst congenital Plagiocephaly Plasma cell disorder Plasma cells absent Plasmablast count decreased Platelet count decreased Platelet glycoprotein gene mutation Platelet maturation arrest Platelet production decreased Platelet toxicity Platonychia Platybasia


Pyloric stenosis

 Date:
 03 July 2019

 Version:
 1.0

 Status:
 Final


Page:

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term

Rare

Poland's syndrome Polycystic liver disease Polydactyly Polymicrogyria Polyorchidism Popliteal pterygium syndrome Porencephaly Porokeratosis Porphyria Porphyria acute Porphyria non-acute Porphyrin metabolism disorder Porphyrinuria Portal venous system anomaly Post infection glomerulonephritis Post streptococcal glomerulonephritis Postauricular fistula Posterior segment of eye anomaly congenital Potter's syndrome Prader-Willi syndrome Preauricular cyst Preduodenal portal vein Preternatural anus Primary cerebellar degeneration Primary ciliary dyskinesia Primary familial hypomagnesaemia Primary hypercholesterolaemia Primary immunodeficiency syndrome Primary insulin like growth factor-1 deficiency Progeria Progressive cerebellar degeneration Progressive external ophthalmoplegia Progressive familial intrahepatic cholestasis Prominent epicanthal folds Promyelocyte count decreased Protein C deficiency Protein S deficiency Proteus syndrome Protuberant ear
Proximal focal femoral deficiency Pseudocholinesterase deficiency Pseudohermaphroditism Pseudohermaphroditism female Pseudohermaphroditism male  ${\tt Pseudohypoaldosteronism}$ Pseudohypoparathyroidism Pseudomembranous colitis Pseudotruncus arteriosus Pseudoxanthoma elasticum Pterygium colli Pulmonary aplasia
Pulmonary arteriovenous fistula
Pulmonary artery atresia
Pulmonary artery stenosis congenital
Pulmonary hypoplasia Pulmonary nypoplasia
Pulmonary lymphangiectasia
Pulmonary malformation
Pulmonary renal syndrome
Pulmonary sequestration
Pulmonary valve stenosis congenital
Pure white cell aplasia


03 July 2019 | **Novo Nordisk** 

Final 146 of 152

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Sickle cell trait

Rare

Pyogenic sterile arthritis pyoderma gangrenosum and acne Pyruvate carboxylase deficiency Pyruvate kinase deficiency anaemia Radiation leukopenia Radioulnar synostosis Rathke's cleft cyst Rectal atresia Red blood cell enzymes abnormal Refsum's disease Renal aplasia Renal arteriovenous malformation Renal dysplasia Renal fusion anomaly Renal hypoplasia Renal malposition Renal vessel congenital anomaly Reproductive tract hypoplasia, male Respiratory tract malformation Retinal anomaly congenital Retinal arteriovenous malformation Retinal coloboma Retinitis pigmentosa Retinopathy congenital Retinoschisis congenital Retroperitonitis Rett syndrome Rhesus haemolytic disease of newborn Rib hypoplasia Rib synostosis Right aortic arch Right ventricular false tendon Right-to-left cardiac shunt Riley-Day syndrome Rippling muscle disease Rotor's syndrome Rubinstein-Taybi syndrome Sacral hypoplasia Sacralisation Sandhoff disease Sarcosinaemia Scaphocephaly Schimke immunoosseous dysplasia Schinzel-Giedion syndrome Schizencephaly Scimitar syndrome Sclerotylosis Sensory neuropathy hereditary Septate hymen Septo-optic dysplasia Septum pellucidum agenesis Serotonin syndrome
Sertoli-cell-only syndrome
Severe myoclonic epilepsy of infancy
Sex chromosome abnormality Shawl scrotum Shigella sepsis Shone complex Short-chain acyl-coenzyme A dehydrogenase deficiency Shwachman-Diamond syndrome Sickle cell anaemia Sickle cell disease


2019 Novo Nordisk 1.0 Final

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Silver-Russell syndrome

Rare

Single umbilical artery Sirenomelia Sjogren-Larsson syndrome Skeletal dysplasia Skin hypoplasia Skin malformation Skull malformation Smith-Lemli-Opitz syndrome Smith-Magenis syndrome
Sotos' syndrome
Special senses congenital anomaly
Spherophakia Spina bifida Spina bifida cystica Spina bifida occulta Spinal muscular atrophy Spine malformation Spinocerebellar ataxia Spleen malformation Spondyloepiphyseal dysplasia Stargardt's disease Stickler's syndrome Sticky platelet syndrome Strabismus congenital Sturge-Weber syndrome Sucrase-isomaltase deficiency Supernumerary nipple Supernumerary vertebra Syndactyly Synostosis Syringomyelia T-lymphocyte count abnormal
T-lymphocyte count decreased Talipes Tangier disease Tay-Sachs disease Telangiectasia congenital Teratogenicity Testicular dysplasia Testotoxicosis Tetrahydrobiopterin deficiency Thalassaemia Thalassaemia alpha Thalassaemia beta Thalassaemia sickle cell Thalidomide embryopathy Thanatophoric dwarfism Thrombocytopenia Thrombocytopenia-absent radius syndrome Thymus hypoplasia Tibial agenesis Tibial torsion Tilted disc syndrome Timothy syndrome Tooth discolouration congenital Tooth hypoplasia Tooth malformation hereditary Tourette's disorder Tracheal atresia Tracheal web Tracheo-oesophageal fistula

Transitional vertebrae


1.0 Final

Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search Preferred term Transposition of the great vessels Rare Trichorhinophalangeal syndrome Trifunctional protein deficiency Trimethylaminuria Triple A syndrome Trisomy 11 Trisomy 13 Trisomy 14 Trisomy 15 Trisomy 17 Trisomy 18 Trisomy 21 Trisomy 22 Trisomy 4p Trisomy 8 Trisomy 9 Truncus arteriosus persistent Tubulointerstitial nephritis and uveitis syndrome Tumour necrosis factor receptor-associated periodic syndrome Turner's syndrome Twin reversed arterial perfusion sequence malformation Type I hyperlipidaemia Type II hyperlipidaemia Type II hyperlipidaemia
Type III hyperlipidaemia
Type IIa hyperlipidaemia
Type IIb hyperlipidaemia
Type IV hyperlipidaemia Type V hyperlipidaemia Tyrosinaemia Uhl's anomaly Umbilical artery hypoplasia Umbilical malformation Unicuspid aortic valve Univentricular heart Urachal abnormality Urea cycle disorder Ureteric atresia Ureteric compression Ureteric dilatation Ureteric obstruction Ureteric stenosis Urethral atresia Urethral valves Urinary tract malformation Urinary tract obstruction Usher's syndrome Uterine aplasia Uterine cervix hypoplasia Uterine hypoplasia Uvula aplasia VACTERL syndrome Vaginal atresia Vaginal hypoplasia Vaginal septum Vascular malformation Velo-cardio-facial syndrome Venolymphatic malformation Ventricular hypoplasia Ventricular septal defect Vertebral artery hypoplasia Vertical talus Very long-chain acyl-coenzyme A dehydrogenase deficiency Vestibulocerebellar syndrome


03 July 2019 Novo Nordisk

1.0 Final 149 of 152

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Rare

Virilism foetal Vitello-intestinal duct remnant

Von Hippel-Lindau disease

Von Willebrand's disease Von Willebrand's disease gene carrier

Waardenburg syndrome Wagner's disease Weill-Marchesani syndrome Welander distal myopathy

Werner's syndrome

White blood cell analysis abnormal White blood cell count abnormal White blood cell count decreased

White blood cell disorder Wildervanck syndrome

Williams syndrome Winchester syndrome Wiskott-Aldrich syndrome Wolf-Hirschhorn syndrome

Wolfram syndrome Wyburn Mason's syndrome

X-linked chromosomal disorder

XXX syndrome

XXXY syndrome XXYY syndrome XYY syndrome Xeroderma pigmentosum

Y-linked chromosomal disorder

Young's syndrome

Zhu-Tokita-Takenouchi-Kim syndrome Zika virus associated birth defect Zika virus associated microencephaly

Zika virus associated ocular birth defect

Suspicion of transmission of infectious disease

Air-borne transmission

Arthropod-borne disease Bacterial disease carrier Community acquired infection

Diphtheria carrier

Direct infection transmission

Faecal-oral transmission of infection

Fungal disease carrier

HIV carrier

HTLV-1 carrier Human immunodeficiency virus transmission

Iatrogenic infection

Indirect infection transmission

Infection transmission via personal contact

Infection via vaccinee Infectious disease carrier Mycobacterial disease carrier Nosocomial infection

Primary transmission Secondary transmission

Sexual transmission of infection Sexually transmitted disease
Sexually transmitted disease carrier

Suspected transmission of an infectious agent via product Transmission of an infectious agent via product Transmission of an infectious agent via transplant

Typhoid carrier

Vaccine virus shedding


03 July 2019

1.0 Final 150 of 152 Novo Nordisk

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Suspicion of transmission of

infectious disease

Vertical infection transmission

Viral disease carrier Viral hepatitis carrier

Vector-borne transmission of infection

Thyroid disorders

Anaplastic thyroid cancer Anti-thyroid antibody

Anti-thyroid antibody positive Antithyroid arthritis syndrome Atrophic thyroiditis

Autoimmune hypothyroidism Autoimmune thyroid disorder Autoimmune thyroiditis

Bannayan-Riley-Ruvalcaba syndrome

Basedow's disease Benign neoplasm of thyroid gland

Biopsy thyroid gland Biopsy thyroid gland abnormal Blood thyroid stimulating hormone abnormal Blood thyroid stimulating hormone decreased Blood thyroid stimulating hormone increased

Butanol-extractable iodine decreased Butanol-extractable iodine increased

Congenital hyperthyroidism Congenital hypothyroidism Congenital thyroid disorder Ectopic thyroid

Endocrine ophthalmopathy Euthyroid sick syndrome

Exophthalmos
Familial medullary thyroid cancer

Follicular thyroid cancer Free thyroxine index abnormal Free thyroxine index decreased Free thyroxine index increased

Gamma radiation therapy to thyroid Generalised resistance to thyroid hormone

Goitre

Goitre congenital

Haemorrhagic thyroid cyst Hashimoto's encephalopathy

Hashitoxicosis

Huerthle cell carcinoma

Hyperthyroidism Hypothyroidic goitre

Hypothyroidism Inappropriate thyroid stimulating hormone secretion

Infectious thyroiditis Iodine uptake abnormal Iodine uptake decreased

Iodine uptake increased Lid lag Malignant exophthalmos

Marine Lenhart syndrome Medullary thyroid cancer Metastases to thyroid

Mvxoedema Myxoedema coma Orbital decompression Papillary thyroid cancer Pendred syndrome

Photon radiation therapy to thyroid

MedDRA version 21.1


Date: Version: Status:

Page:

03 July 2019 | **Novo Nordisk**1.0 |
Final


Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Thyroid disorders

```
Polyglandular autoimmune syndrome type II
Polyglandular autoimmune syndrome type III
Poorly differentiated thyroid carcinoma
Post procedural hypothyroidism
Primary hyperthyroidism
Primary hypothyroidism
Protein bound iodine decreased
Protein bound iodine increased
Radiation thyroiditis
Radioactive iodine therapy
Radiotherapy to thyroid
Reverse tri-iodothyronine decreased
Reverse tri-iodothyronine increased
Secondary hyperthyroidism
Secondary hypothyroidism
Silent thyroiditis
Tertiary hypothyroidism
Thyreostatic therapy
Thyroglobulin absent
Thyroglobulin decreased
Thyroglobulin increased
Thyroglobulin present
Thyroglossal cyst infection
Thyroglossal fistula
Thyroid B-cell lymphoma
Thyroid C-cell hyperplasia
Thyroid adenoma
Thyroid atrophy
Thyroid calcification
Thyroid cancer
Thyroid cancer metastatic
Thyroid cancer recurrent
Thyroid cancer stage 0
Thyroid cancer stage
Thyroid cancer stage II
Thyroid cancer stage III
Thyroid cancer stage IV
Thyroid cyst
Thyroid dermatopathy
Thyroid disorder
Thyroid dysfunction in pregnancy
Thyroid echinococciasis
Thyroid electron radiation therapy
Thyroid fibrosis
Thyroid function test abnormal
Thyroid gland abscess
Thyroid gland injury
Thyroid gland scan abnormal
Thyroid haemorrhage
Thyroid hemiagenesis
Thyroid hormone replacement therapy
Thyroid hormones increased
Thyroid infarction
Thyroid malformation
Thyroid mass
Thyroid neoplasm
Thyroid operation
Thyroid pain
Thyroid releasing hormone challenge test abnormal
Thyroid size decreased
Thyroid steatosis
Thyroid stimulating hormone deficiency
Thyroid stimulating immunoglobulin increased
```


03 July 2019 | Novo Nordisk 1.0

Final 152 of 152

Pre-defined MedDRA search - list of preferred terms

Pre-defined MedDRA search

Preferred term

Thyroid disorders

Thyroid therapy Thyroid tuberculosis Thyroidectomy Thyroiditis Thyroiditis acute Thyroiditis chronic Thyroiditis fibrous chronic Thyroiditis subacute Thyrotoxic cardiomyopathy Thyrotoxic crisis

Thyrotoxic myopathy
Thyrotoxic periodic paralysis
Thyroxin binding globulin abnormal
Thyroxin binding globulin decreased
Thyroxin binding globulin increased

Thyroxine abnormal Thyroxine decreased Thyroxine free abnormal Thyroxine free decreased Thyroxine free increased Thyroxine increased Thyroxine therapy Toxic goitre

Toxic nodular goitre

Transient hypothyroxinaemia of prematurity Tri-iodothyronine abnormal Tri-iodothyronine decreased Tri-iodothyronine free abnormal Tri-iodothyronine free decreased Tri-iodothyronine free increased Tri-iodothyronine free normal Tri-iodothyronine increased Tri-iodothyronine uptake abnormal

Tri-iodothyronine uptake decreased Tri-iodothyronine uptake increased Ultrasound thyroid abnormal X-ray therapy to thyroid

MedDRA version 21.1

nn9535/nn9535-4114/20190704\_rm\_er 02JUL2019:18:22:33 - l\_meddra.sas/l\_meddra.txt